## **Statistical Analysis Plan Amendment 1**

**Study ID:** 213199

**Official Title of Study:** A Phase IIIb, Open-label, Hybrid Type III Trial Evaluating Implementation Strategies for Long-acting Cabotegravir Plus Longacting Rilpivirine Every Two Months in HIV-1 Infected, Virologically Suppressed Adults in Select European Healthcare Settings

**NCTID:** NCT04399551

**Date of Document:** 12 December 2022

#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|---|---|---|
| Information Type | : | Reporting and Analysis Plan (RAP) |
| Title | : | Reporting and Analysis Plan for A Phase IIIb, open-<br>label, hybrid type III trial evaluating implementation<br>strategies for long-acting cabotegravir plus long-acting<br>rilpivirine every two months in HIV-1 infected,<br>virologically suppressed adults in select European<br>healthcare settings. |
| <b>Compound Number</b> | : | GSK1265744 |
| Clinical Study<br>Identifier | : | 213199 |
| Effective Date | : | 30 Nov 2022 |

## **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 213199, specifically for clinical efficacy and safety data. Any implementation science/health outcome analysis non-clinical data will be detailed in the Evidera SAP.
- This RAP will be provided to the study team members to convey the content of pertaining to clinical data for the interim, Month 12, and End of Study (EOS) analyses.

#### RAP Author(s):

| Author | Date |
|--------------------------------------------------|-------------------------|
| PPD | 10-NOV-2022 |
| Principal Statistician (GSK Clinical Statistics) | |
| Co-Author | |
| PPD | Electronic (NOV - 2022) |
| Principal Programmer (GSK Clinical Programming) | |

Copyright 2022 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

#### **RAP Team Reviews:**

# **RAP Team Review Confirmations**

(Method: E-mail)

| Reviewer | Date |
|---|---|
| PPD | 16-NOV-2022 |
| Clinical Science Lead (ViiV Healthcare) | |
| PPD | 18- NOV -2022 |
| Innovation & Implementation Science (ViiV Innovation & Implementation Science) | |
| PPD | 18- NOV -2022 |
| SERM Manager (Pharma Safety SERM) | |
| PPD | 11- NOV -2022 |
| PPD (ViiV Healthcare) | |
| PPD | 18- NOV -2022 |
| Data Management Quality Lead (GSK Data Management) | |
| PPD | 16- NOV -2022 |
| Global Implementation Research (ViiV Innovation & Implementation Science) | |
| PPD | 18- NOV -2022 |
| Clinical Study Manager (Global Clinical Sciences & Delivery, GSK) | |
| PPD | 18- NOV -2022 |
| PPD , Research & Development (Clinical Development Lead, ViiV Physicians) | |
| PPD | 16- NOV -2022 |
| Clinical Development Manager, Virology (ViiV Healthcare) | |

## **Clinical Statistics and Clinical Programming Line Approvals:**

# Clinical Statistics & Clinical Programming Line Approvals (Method: Pharma TMF eSignature)

| Approver | | Date |
|----------|----------------------------------------|-------------------|
| PPD | | Electronic (NOV - |
| PPD | , Statistics (GSK Clinical Statistics) | 2022) |
| PPD | | Electronic (NOV - |
| PPD | Programming (GSK Clinical Programming) | 2022) |

## **TABLE OF CONTENTS**

| | | PAGE |
|----|-----------------------------------------------------------------|------|
| 1. | INTRODUCTION | 6 |
| | 1.1. RAP Amendments | 6 |
| 2. | SUMMARY OF KEY PROTOCOL INFORMATION | 7 |
| | 2.1. Changes to the Protocol Defined Statistical Analysis Plan | 7 |
| | 2.1.1. Changes to Protocol Defined Analysis Plan | |
| | 2.2. Study Objective(s) and Estimand(s) / Endpoint(s) | 8 |
| | 2.3. Study Design | 11 |
| | 2.4. Statistical Hypotheses / Statistical Analyses | 13 |
| | 2.4.1. Sample Size Determination | 13 |
| 3. | PLANNED ANALYSES | 18 |
| | 3.1. Interim Analyses | |
| | 3.2. Final Analyses | 18 |
| 4. | | |
| | 4.1. Protocol Deviations | 19 |
| 5. | | 20 |
| | CONVENTIONS5.1. Study Treatment & Sub-group Display Descriptors | 20 |
| | 5.2. Baseline Definitions | |
| | 5.3. Multicentre Studies | |
| | 5.4. Examination of Covariates, Other Strata and Subgroups | |
| | 5.4.1. Covariates and Other Strata | 20 |
| | 5.4.2. Examination of Subgroups | |
| | 5.5. Other Considerations for Data Analyses and Data Handling | |
| | Conventions | 21 |
| 6. | | |
| | 6.1. Overview of Planned Study Population Analyses | 22 |
| 7. | | |
| | 7.1. Secondary Efficacy Analyses | |
| | 7.1.1. Endpoint / Variables | |
| | 7.1.2. Population of Interest | |
| | 7.1.3. Strategy for Intercurrent (Post-Randomization) Events . | |
| | 7.1.4. Statistical Analyses / Methods | 24 |
| 8. | SAFETY ANALYSES | |
| | 8.1. Safety Endpoints | |
| | 8.2. Adverse Events Analyses | 25 |
| | 8.3. Adverse Events of Special Interest Analyses | |
| | 8.4. Clinical Laboratory Analyses | |
| | 8.5. Other Safety Analyses | 26 |
| 9. | | |
| | 9.1. Endpoint / Variables | 27 |


| | | 9.1.1. | Drug Concentration Measures | 27 |
|---|---|---|---|---|
| 10. | VIROL | OGY | | 28 |
| | | | ic and Phenotypic Data | |
| 11. | OTHE | R ANALY: | SES | 29 |
| | 11.1. | | : / Variables | |
| | | 11.1.1. | | |
| | | 11.1.2. | Pregnancy | |
| 12. | REFE | RENCES. | | 30 |
| 13. | APPE | NDICES | | 31 |
| | 13.1. | Appendix | x 1: Schedule of Activities | 31 |
| | | 13.1.1. | Protocol Defined Schedule of Events: Schedule of Activities for Patient Study Participants | 21 |
| | 13.2. | Annondi | x 2: Assessment Windows | 31<br>27 |
| | 13.2. | 13.2.1. | | |
| | | 13.2.1. | • | |
| | | 13.2.2. | Assessment Windows for Pregnancy Data | |
| | 13.3. | | x 3: Study Phases | 41<br>12 |
| | 13.3. | 13.3.1. | Study Phases | |
| | | 13.3.1. | Treatment State | |
| | | 13.3.3. | Oral Lead-in Period | |
| | 13.4. | | x 4: Data Display Standards & Handling Conventions | |
| | 10.4. | 13.4.1. | Reporting Process | |
| | | 13.4.2. | Reporting Standards | |
| | | 13.4.3. | Reporting Standards for Pharmacokinetic Data | |
| | 13.5. | | x 5: Derived and Transformed Data | |
| | 10.0. | 13.5.1. | General | |
| | | 13.5.2. | Study Population | |
| | | 13.5.3. | Efficacy | |
| | | 13.5.4. | Safety | |
| | | 13.5.5. | Virology | |
| | | 13.5.6. | Other Assessments | |
| | 13.6. | | x 6: Reporting Standards for Missing Data | |
| | | | Premature Withdrawals | |
| | | 13.6.2. | Handling of Missing Data | |
| | 13.7. | Appendix | x 7: Values of Potential Clinical Importance | |
| | | 13.7.1. | Hepatobiliary Abnormality Criteria | |
| | 13.8. | Appendix | x 8: Snapshot Algorithm Details | |
| | 13.9. | | x 9: Identification of Adverse Events of Special Interest | |
| | | 13.9.1. | Hepatic Safety Profile | |
| | | 13.9.2. | Hyperglycaemia | 69 |
| | | 13.9.3. | Hypersensitivity Reactions | 71 |
| | | 13.9.4. | Rash including severe cutaneous adverse reactions | 72 |
| | | 13.9.5. | Prolongation of the Corrected QT Interval of the ECG in Supra Therapeutic Doses | 7/ |
| | | 13.9.6. | Suicidal Ideation/Behaviour | |
| | | 13.9.0. | Depression | |
| | | 13.9.8. | Bipolar Disorder | |
| | | 13.9.9. | Psychosis | |
| | | 10.0.0. | . 5,5,5,5,6 | 1 0 |


| | 13.9.11. | Mood Disorders Anxiety Sleep Disorders | 83 |
|--------|----------|-------------------------------------------------|-----|
| | CCI | | |
| | 13.9.14. | Seizures | 91 |
| | 13.9.15. | Weight Gain | 96 |
| | 13.9.16. | Rhabdomyolysis | 97 |
| | | Pancreatitis | |
| | 13.9.18. | Impact on Creatinine | 99 |
| | 13.9.19. | Safety During Pregnancy | 101 |
| 13.10. | Appendix | ( 10: Identification of COVID-19 Adverse Events | 102 |
| 13.11. | Appendix | < 11: Abbreviations & Trade Marks | 104 |
| | | Abbreviations | |
| | 13.11.2. | Trademarks | 105 |
| 13.12. | Appendix | < 12: List of Data Displays | 106 |
| | | Data Display Numbering | |
| | 13.12.2. | Mock Example Shell Referencing | 106 |
| | | Deliverables | |
| | | Study Population Tables | |
| | | Efficacy Tables | |
| | 13.12.6. | Efficacy Figures | 114 |
| | 13.12.7. | Safety Tables | 116 |
| | | Safety Figures | |
| | 13.12.9. | Other Tables | 127 |
| | 13.12.10 | .ICH Listings | 128 |
| | 13.12.11 | .Non-ICH Listings | 131 |
| 13.13. | | ( 13: Example Mock Shells for Data Displays | |

#### 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol 213199. This RAP is based on the original protocol (Dated 06-MAY-2020) of study GSK1265744/213199 (GSK Document Number 2019N420690\_01) and its protocol amendments 01 (Dated 02-DEC-2020, GSK Document Number 2019N420690\_02) and 02 (Dated 24-MAY-2021, GSK Document No. TMF-13794092).

| GlaxoSmithKline<br>Document Number | Date | Version |
|------------------------------------|-------------|-----------------|
| TMF-11899418 | 12-MAR-2021 | Original |
| TMF-15213711 | 30 Nov 2022 | Amendment No. 1 |

The reasons for this amendment were to: plan specific outputs related to participant pregnancy in line with protocol amendment 02; add clarity on the Covid PD impact on exposure formula; Adjust on treatment definition to add 63 days post injection instead of 35; Additional categories added to summarize oral exposure to Oral Bridging (Covid and Non-Covid related); if SOC ART started immediately after missed injection, then injection would not be count as missed. Clarity added around entry into LTFU and transition to commercial product. List of displays for EOS updated to account for pregnancy and RAPIDO Data Viewer.

#### 1.1. RAP Amendments

Revision chronology:

| RAP Section | Amendment Details | |
|---|---|---|
| Reporting and Analysis Pl | Reporting and Analysis Plan (RAP) CARISEL_213199_Final [12-MAR-2021] | |
| Reporting and Analysis Pl | an (RAP) CARISEL_213 | 3199_Amendment_1 [30 Nov 2022] |
| Inclusion of additional pregnancy based output | | Protocol amendment 02 allows pregnant participants to continue on study. Listings have been added to address pregnancy specific events. |
| Data Handling | | <ul> <li>Pregnancy data accommodations have been added.</li> <li>Exposure formulas were adjusted to account for Q8W dosing, protocol deviation impact, transition to commercial product, and various scenarios related to Oral Bridging or missed injections.</li> </ul> |
| Data Displays | | Display status for EOS was updated to<br>consider use of the RAPIDO Data Viewer. The<br>following displays were added for pregnancy<br>summarization: Listings 49-57 |

#### 2. SUMMARY OF KEY PROTOCOL INFORMATION

Cabotegravir long-acting + rilpivirine long-acting (CAB LA + RPV LA) is an HIV-1 treatment regimen administered as two individual intramuscular injections monthly or every two months (following an optional oral lead-in [OLI] period). The overall objective of the CAB LA + RPV LA clinical development program was to develop a highly effective, well-tolerated, two-drug, long-acting injectable regimen which has the potential to offer improved treatment convenience, compliance and improved quality of life for people living with HIV (PLHIV) compared to current standard of care.

This new HIV treatment will require changes to the current standard of prescribing oral antiretroviral therapies to prescribing and delivering a complete antiretroviral long acting injectable regimen. As this is a new treatment modality, it is important to understand how to optimize the delivery of CAB LA + RPV LA from a patient, healthcare provider and healthcare system perspective in order to implement into routine care with fewer obstacles. Each country's healthcare system has its own challenges and nuanced differences in the delivery of HIV care. Strategies to support the unique and dynamic contexts for CAB LA + RPV LA implementation is key. As a result, this research study will examine different implementation strategies in different clinics settings across European countries to identify which strategies best meet the needs in each local context. The research in this study will involve both patients receiving the study treatment CAB LA + RPV LA (patient study participants, PSP) as well as the healthcare providers at the investigator site level (staff study participants, SSP).

For PSPs, the study is single-arm, unblinded and interventional, where all patients who fulfil eligibility requirements will be assigned to receive CAB LA + RPV LA and complete assessments as per the study protocol.

For SSPs, the study is two-arm, unblinded, non-interventional and cluster-randomized at the country level. Sites within a given country will be randomized to either the Standard (Arm-s) or the Enhanced (Arm-e) implementation arm. The two arms will involve the provision of overlapping but distinct types of implementation components that are designed to assist in the local implementation of the study drug at each site. Arm-s represents the traditional provider support by a medical science lead and product materials. Arm-e models a higher level of provider support with added face to face meeting, trainings, and additional touchpoints for administration of CAB LA + RPV LA. The study will evaluate both qualitative and quantitative measures across arm, clinic type, provider type, and country to determine the most effective implementation strategies and to identify barriers and facilitators (including solutions). Clinical data will be collected to monitor safety and efficacy.

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

A change to the originally planned statistical analysis specified in the 213199 protocol [Dated: 06MAY2020] consists of dropping the ITT-E population and introducing the Enrolled population. This is being done as the ITT-E carries the same definition as the Safety population so both populations are not needed. Efficacy is also a secondary endpoint so it would add unnecessary programming work to include an identical

population. The Safety population will serve as the primary population for both safety and efficacy analyses. The Enrolled population is being added in order to adhere to EudraCT standards.

# 2.1.1. Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | Rationale |
|---|---|---|
| An ITT-E population is listed to be used in statistical analysis. | This population is being dropped and the Safety population will be used for efficacy analysis. An Enrolled population is also being added. | The ITT-E and Safety populations carry the same definition so only one is needed for analysis. The Enrolled population is added to adhere to EudraCT standards. |

# 2.2. Study Objective(s) and Estimand(s) / Endpoint(s)

| Objectives | Endpoints/Estimands |
|---|---|
| Primary | |
| Staff Study Participants (SSP): To evaluate | Quantitative Change of Acceptability of Implementation Measure (AIM) Score, Implementation Appropriateness Measure (IAM) Score, Feasibility of Implementation Measure (FIM) Score over time assessed quantitatively via questionnaires through Month 12.a Qualitative Semi-structured interviews (SSI) assessed qualitatively through Month 12. |
| Secondary | |
| <ul> <li>Staff Study Participants: To evaluate</li> <li>Facilitators to implementation</li> <li>Barriers to implementation</li> <li>Adaptations/Modifications to address barriers and facilitators</li> </ul> | Quantitative: Change of Implementation Leadership Scale (ILS), Change and Implementation Climate Scale (ICS) over time assessed quantitatively via questionnaires through Month 12. <sup>a</sup> Summarize components from Enhanced Implementation & Standard Implementation: • FRAME-IS outcome Months 2 – 12 (monthly) |
| | Summarize components from Enhanced Implementation: • CQI 1-hour calls/PDSAs minimum of Months 2-7 (monthly) |

| Objectives | Endpoints/Estimands |
|---|---|
| Patient Study Participants (PSP) To evaluate • Facilitators to implementation • Barriers to Implementation | Qualitative SSIs assessed qualitatively through Month 12. Quantitative: Questionnaires assessed quantitatively through Dose 7.b Length of patient study participant visit from arrival until departure from clinic assessed at Dose 1, Dose 2, Dose 4, and Dose 5. Qualitative SSIs assessed qualitatively through Dose 7. |
| To evaluate Patient Study Participants experience for delivering CAB LA + RPV LA, including • Acceptability • Appropriateness • Feasibility | Quantitative Change in Acceptability of Intervention Measure (AIM) Score, Intervention Appropriateness Measure (IAM) Score, and Feasibility of Intervention Measure (FIM) Score over time. Assessed via questionnaires at Dose 7. b Qualitative SSIs assessed qualitatively through Dose 7. |
| To evaluate sustainability of CAB<br>LA + RPV LA with <b>Study Staff</b><br><b>Participants</b> each clinic | Total score of the Clinical Sustainability Assessment Tool (CSAT) at Month 12. |
| To assess fidelity to CAB LA + RPV LA injection dosing windows | Percentage of injections occurring within target window from the target date. |
| Evaluate efficacy and safety measures of CAB LA + RPV LA | Proportion of participants with plasma HIV-1 RNA <50 c/mL over time. Proportion of participants with confirmed virologic failure (CVF) over time Incidence of treatment-emergent genotypic and phenotypic resistance to CAB and RPV in patient study participants with CVF |

| Objectives | Endpoints/Estimands |
|---|---|
| | Incidence and severity of AEs, SAEs and proportion of participants who discontinue treatment due to AEs over time |
| To assess preference between CAB LA + RPV LA and oral ART medication received prior to entering the study | Preference between CAB + RPV LA and daily oral ART medication (received prior to entering the study) at quantitatively assessed via preference questionnaire at Dose 7 |



## 2.3. Study Design

Study 213199 (Cabotegravir And Rilpivirine Implementation Study in European Locations -CARISEL) is a cluster randomized, two-arm, open-label, hybrid effectiveness-implementation study designed to evaluate two implementation strategy conditions (Enhanced [Arm-e] vs Standard [Arm-s]) in various clinical settings across five European countries.

This study is an evaluation of implementation strategies on the degree of acceptability, appropriateness, feasibility, fidelity, and sustainability of clinic practices to deliver the CAB LA + RPV LA regimen. The study will use an implementation science approach to understand the barriers and facilitators for both patients and providers, including best practices for delivering CAB LA + RPV LA within an interventional clinical trial where the CAB LA + RPV LA regimen is delivered to HIV-1-infected, virologically-suppressed adult patients. This design allows for a simultaneous focus on both implementation and effectiveness, which allows for maximizing our understanding of how-to best support translation of CAB LA + RPV LA into routine care while continuing to collect effectiveness and safety data. The hybrid type III focuses primarily on the impact of the implementation to get the intervention (CAB LA + RPV LA) into routine care. As a result, the primary focus of this study is implementation. The secondary focus is on the clinical effectiveness.

All patients who fulfill eligibility requirements will receive the study treatment of CAB LA + RPV LA and will begin oral therapy with CAB 30 mg + RPV 25 mg once daily for approximately one month to determine individual safety and tolerability prior to receiving CAB LA + RPV LA for an additional 11 months. Total patient study participant duration in the study is approximately 13 months including screening.

Patient participants in CARISEL who successfully complete the study (Dose 7), without meeting study-defined withdrawal criteria, will be given the option to continue to receive CAB LA + RPV LA, administered Q2M in the Extension Phase until the study treatment is either locally approved and commercially available (including through local public/government health sectors), the participant no longer derives clinical benefit, the participant meets a protocol-defined reason for discontinuation or until development of either CAB LA + RPV LA Q2M is terminated. Alternatively, participants can choose to complete study participation and enter the 52-week LTFU Phase of the study.

Any participant who receives at least one dose of CAB LA and/or RPV LA and discontinues the CAB LA + RPV LA regimen for any reason will enter a 52-week LTFU Phase. Those participants must remain on suppressive highly active antiretroviral therapy (HAART) for at least 52 weeks after the last dose of CAB LA and/or RPV LA.

There are two arms for the providers (arm-e and arm-s) which contain different levels and type of support for the implementation of the HIV Regimen. Cluster randomization will be used to randomize sites in each country to either arm-e or arm-s.



## 2.4. Statistical Hypotheses / Statistical Analyses

The hypotheses on the quantitative aspects of this study is that enhanced implementation strategy is superior than the standard implementation strategy in terms of mean staff study participant (SSP) AIM/IAM/FIM scores. i.e.,

•  $H_0$ :  $\mu$ (enhanced) =  $\mu$ (standard) vs.  $H_1$ :  $\mu$ (enhanced) >  $\mu$ (standard)

Further analysis details for this hypothesis will be covered in the Evidera SAP.

### 2.4.1. Sample Size Determination

The study size is based on practical considerations in terms of feasibility of enrolling an adequate number of sites on each implementation strategy balanced with the desire to have interventions tested across several types of investigative sites; as well as enrolling an adequate number of patient study participants in each site.

Approximately 24 sites (from feasibility process) will be selected from the feasibility process to achieve 18 sites randomly assigned to study implementation strategies and approximately 54 evaluable staff study participants for an estimated total of 27 evaluable study staff participants per implementation strategy group.

Assuming 10% screen failures, it is estimated that with 18 sites approximately 527 patient study participants will be screened to achieve 474 subjects enrolled and 450 evaluable patient study participants completing the study (assumes 5% of patient study participants would be non-evaluable) for an estimated total of 225 evaluable patient study participants per implementation strategy group.

#### 2.4.1.1. Power to Show Superiority in mean SSP AIM/IAM/FIM scores

Table A shows preliminary AIM/IAM/FIM data from the ongoing U.S. implementation study CUSTOMIZE (209493).

Table A Staff Study Participants Scores at Month 4 in CUSTOMIZE (209493)

| | N | Mean | SD | Median | Observed<br>Range<br>(min-max) | Floor<br>n (%) | Ceiling<br>n (%) | Skewness | Kurtosis |
|---|---|---|---|---|---|---|---|---|---|
| AIM<br>Scale<br>(Total<br>Sample) | 24 | 4.39 | 0.61 | 4.13 | 3.25-5.00 | 0 (0.0%) | 11<br>(45.8%) | -0.16 | -1.58 |
| IAM<br>Scale<br>(Total<br>Sample) | 24 | 4.45 | 0.59 | 4.50 | 3.25-5.00 | 0 (0.0%) | 12<br>(50.0%) | -0.34 | -1.39 |
| FIM<br>Scale<br>(Total<br>Sample) | 24 | 4.32 | 0.71 | 4.25 | 3.00-5.00 | 0 (0.0%) | 11<br>(45.8%) | -0.47 | -1.09 |

Based on these preliminary data from CUSTOMIZE study, and the given sample size (the number of study participants), the power to detect a difference of 0.5 between the implementation arms in terms of AIM, IAM and FIM in line with our primary hypothesis are shown in Table B.

Table B Power to Detect a 0.5 Difference in AIM/IAM/FIM

| Endpoint | ARM-<br>S | ARM-<br>E | Delta | SD | Alpha | N(S) | N(E) | Power* |
|---|---|---|---|---|---|---|---|---|
| AIM | 4.39 | 4.89 | 0.5 | 0.61 | 0.05 | 27 | 27 | 84% |
| | | | | | | 36 | 36 | 93% |
| IAM | 4.45 | 4.95 | 0.5 | 0.59 | 0.05 | 27 | 27 | 86% |
| | | | | | | 36 | 36 | 94% |
| FIM | 4.32 | 4.82 | 0.5 | 0.71 | 0.05 | 27 | 27 | 72% |
| | | | | | | 36 | 36 | 84% |

<sup>\*</sup>Power calculation using two-sided T-test assuming equal variance.

As shown in Table B, with 27 study staff participants (3 per site) surveyed on each arm, the study would have 72%-86% power to detect a 0.5 difference in FIM, AIM and IAM endpoints between ARM-E (Enhanced implementation strategy arm) and ARM-S (Standard implementation arm) assuming data from Table A (CUSTOMIZE study) for ARM-S.

And with 36 study staff participants (4 per site) surveyed on each arm, the study would have 84% - 94% power to detect a 0.5 difference in FIM, AIM and IAM endpoints between ARM-E and ARM-S.

#### 2.4.1.2. Sample Size for Provider Population

An overall average number of 9 sites, per arm (18 sites), would produces a two-sided 95% confidence interval with a distance from the mean paired difference (e.g. site level mean change from baseline in AIM, IAM or FIM score) to the limits (half-width) that is equal to 0.497 when the estimated standard deviation of the paired differences is 1.0, across sites.

Table C Sensitivity Analysis for Sample Size versus Half-Width (Precision)-Two-Sided 95% Confidence Interval (For Number of Sites)

| Sample Size | Actual Distance from Mean | |
|-------------|---------------------------------|--------|
| | Difference to Limits (Precision | |
| | SD=0.5 | SD=1.0 |
| 10 | 0.358 | 0.715 |
| 11 | 0.336 | 0.672 |
| 12 | 0.318 | 0.635 |
| 13 | 0.302 | 0.604 |
| 14 | 0.289 | 0.577 |
| 15 | 0.277 | 0.554 |
| 16 | 0.266 | 0.533 |
| 17 | 0.257 | 0.514 |
| 18 | 0.249 | 0.497 |
| 19 | 0.241 | 0.482 |
| 20 | 0.234 | 0.468 |

A sample size of 27 providers, per arm, produces a two-sided 95% confidence interval with a distance from the mean paired difference to the limits (half-width) that is equal to 0.396 when the estimated standard deviation of the paired differences is 1.0.

Table D Sensitivity Analysis for Sample Size versus Half-Width (Precision)-Two-Sided 95% Confidence Interval (for Number of Providers)

| Sample Size | Actual Distance from Mean Difference to Limits (Precision) | |
|---|---|---|
| | SD=0.5 | SD=1.0 |
| 21 | 0.228 | 0.455 |
| 22 | 0.222 | 0.443 |
| 23 | 0.216 | 0.432 |
| 24 | 0.211 | 0.422 |
| 25 | 0.206 | 0.413 |
| 26 | 0.202 | 0.404 |
| 27 | 0.198 | 0.396 |
| 28 | 0.194 | 0.388 |
| 29 | 0.190 | 0.380 |
| 30 | 0.187 | 0.373 |



Figure A Sensitivity Analysis for Sample Size versus Half-Width (Precision)-Two-Sided 95% Confidence Interval (for Sites and Providers)

#### 2.4.1.3. Sample Size for Patient Population

A sample size of 225 patient subjects per implementation strategy group produces a two-sided 95% confidence interval with a distance from the mean paired difference to the limits that is equal to 0.131 when the estimated standard deviation of the paired difference is 1.

Table E Sensitivity Analysis for Sample Size versus Half-Width (Precision)-Two-Sided 95% Confidence Interval (for Patients)

| Sample Size | Actual Distance from Mean Difference to Limits (Precision) SD=0.5 SD=1.0 | |
|---|---|---|
| 400 | 0.000 | 0.400 |
| 100 | 0.099 | 0.198 |
| 125 | 0.089 | 0.177 |
| 150 | 0.081 | 0.161 |
| 175 | 0.075 | 0.149 |
| 200 | 0.070 | 0.139 |
| 225 | 0.066 | 0.131 |
| 250 | 0.062 | 0.125 |



Figure B Sensitivity Analysis for Sample Size versus Half-Width (Mean Diff to Limit) versus Sample Size - Patients (Multiple Confidence Levels)

As explained in the protocol, launching CAB LA + RPV LA in the real world may present challenges that were not observed in a clinical trial setting. Therefore, in addition to the primary analyses which focuses on study staff participants data, statistical analyses of patient outcome endpoints will be performed to evaluate changes in study patients' satisfaction score results, to allow an informal comparison between the two implementation strategies.



#### 3. PLANNED ANALYSES

This RAP describes standard analyses that will be applied to descriptively summarize clinical adverse events, laboratory evaluations, virologic parameters and other clinical safety and efficacy outcomes.

Details pertaining to reporting of survey/interview data and health outcomes/effectiveness analyses will be described in a separate analysis plan provided by Evidera or other CRO partner under GSK's oversight.

At least three analyses will be conducted to evaluate primary and secondary objectives of the protocol; an interim analysis after 50% of subjects have received their 3<sup>rd</sup> injection, and interim analysis after 100% of subjects have received their 3<sup>rd</sup> injection, and finally the primary analysis at Month 12. Further data cuts and analyses may be conducted as necessary, in order to support for internal use and publications.

A final end-of-study (EOS) analysis will be conducted when all subjects have completed the study.

## 3.1. Interim Analyses

As mentioned previously, interim analyses will be performed when 50% and 100% of subjects have received their 3<sup>rd</sup> injection. No formal criteria for stopping or amending the study based on the interim analysis are envisioned. Further interim analyses may be planned for publication data.

## 3.2. Final Analyses

The planned Month 12 primary analysis will be performed after the completion of the following sequential steps:

- All participants have completed Month 12 of the study as defined in the protocol, including any required re-tests.
- All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.

#### 4. ANALYSIS POPULATIONS

This RAP defines patient study participants in detail. Analysis populations that pertain to implementation science deliverables are documented in the Evidera SAP.

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Subjects Screened Population | All participants who were screened for eligibility and inclusion in the study | Patient Study Population |
| Enrolled Population | All patient study participants who passed screening and entered the study. | <ul><li>Patient Study<br/>Population</li></ul> |
| Safety | All enrolled participants who received at least one dose of CAB + RPV Oral or CAB LA + RPV LA. | <ul> <li>Patient Study Population, Safety, Efficacy, Virology, Other Assessments </li> </ul> |
| Long Term<br>Follow-up<br>Population | All subjects receiving at least one dose of CAB LA and/or RPV LA who have discontinued CAB LA +RPV LA regimen and have at least one Long Term Follow-up phase clinic visit | Efficacy, Safety |

Refer to Appendix 12: List of Data Displays which details the population used for each display.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan [25NOV2020 v2.0].

- o Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

Protocol deviations related to the implementation process, and not the clinical conduct of the study will be reported separately. The identification and categorization of PDs as important may be different for implementation PDs vs those associated with the clinical conduct of the study.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | |
|---|---|---|
| Data Displays for Reporting | | |
| Description Order in TLF Analysis | | |
| CAB Oral +RPV Oral | 1 | OLI Safety |
| CAB LA +RPV LA (includes both QM and Q2M dosing) 1 Study Population, Efficacy, Safety | | |

#### 5.2. Baseline Definitions

For all endpoints the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

#### 5.3. Multicentre Studies

In this multicentre, European-based study, enrolment and demographics will be presented by investigator site.

Exploratory analyses will be considered only if applicable.

## 5.4. Examination of Covariates, Other Strata and Subgroups

#### 5.4.1. Covariates and Other Strata

The list of covariates and other strata may be used in descriptive summaries and statistical analyses, some of which may also be used for subgroup analyses. Additional covariates and other strata of clinical interest may also be considered.

| Category | Details |
|---|---|
| Covariates | Implementation strategy, Site, Country, Gender, Age Group, Race, CD4 Count |

## 5.4.2. Examination of Subgroups

The list of subgroups may be used in descriptive summaries and statistical analyses. Additional subgroups of clinical interest may also be considered.

If the percentage of subjects is small within a particular subgroup, then the subgroup categories may be combined.

| Subgroup | Categories |
|-------------------------|-------------------|
| Implementation Strategy | Standard |
| | Enhanced |
| Site | 18 European sites |
| Country | As collected |
| Gender | Male |
| | Female |
| Age | • ≥50 |
| | • <50 |
| Race | White |
| | African Heritage |
| | Asian |
| | Other |
| CD4 Count | • <350 |
| | • ≥350 |

# 5.5. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|-----------------------------------------------------------|
| 13.1 | Appendix 1: Schedule of Activities |
| 13.2 | Appendix 2: Assessment Windows |
| 13.3 | Appendix 3: Study Phases |
| 13.4 | Appendix 4: Data Display Standards & Handling Conventions |
| 13.5 | Appendix 5: Derived and Transformed Data |
| 13.6 | Appendix 6: Reporting Standards for Missing Data |
| 13.7 | Appendix 7: Values of Potential Clinical Importance |

## 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the Safety population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in <a href="Appendix 12">Appendix 12</a>: List of Data Displays. Enrollment and demographics will be displayed by Implementation strategy, site, country, and overall.

For the two interim analyses based on subjects' 3<sup>rd</sup> injection data, study population tables and listings will be produced by GSK. Details of these Interim Analysis deliverables can be found in Appendix 12: List of Data Displays.

#### 7. EFFICACY ANALYSES

Implementation Science/Health Outcomes endpoints will form the basis for the overall primary analysis of the study, and details of implementation science/health outcomes analyses are documented in a separate Evidera SAP. Clinical efficacy endpoints are evaluated as secondary objectives for this study.

Efficacy analyses will be performed at Month 12 and EOS. There will be no efficacy reported at the interim analyses.

## 7.1. Secondary Efficacy Analyses

## 7.1.1. Endpoint / Variables

- Proportion of participants with Plasma HIV-RNA < 50 copies/mL and plasma HIV-1 RNA ≥ 50 copies/mL as per Food and Drug Administration (FDA) Snapshot algorithm at Month 12 (Safety Population). See <u>Appendix 8</u> for Snapshot Algorithm details.
- Participants with protocol-defined confirmed virologic failure (CVF) over time (Safety population)
- Incidence of treatment-emergent genotypic and phenotypic resistance to CAB and RPV in patient study participants with CVF (Safety population)

#### 7.1.2. Population of Interest

The primary efficacy analyses will be based on the Safety population, unless otherwise specified. HIV-1 RNA summaries will also be reported for the Long-Term Follow-up Population.

## 7.1.3. Strategy for Intercurrent (Post-Randomization) Events

Participants with last available HIV-1 RNA measurement less than 50 copies/mL while the participant is on treatment within the analysis visit window of interest are classified as HIV-1 RNA < 50 c/mL. Participants without evaluable HIV-RNA data for the visit of interest or who change treatment not permitted per protocol before the analysis window are considered non-responders.

Participants with last available HIV-1 RNA measurement greater or equal to 50 copies/mL while the participant is on treatment within the analysis visit window of interest are classified as HIV-1 RNA  $\geq$  50 c/mL. Participants without evaluable HIV-RNA data for the visit of interest and who discontinue treatment for reasons not related to adverse event while having HIV-1 RNA  $\geq$ 50 copies/mL at time of discontinuation or who change study treatment not permitted per protocol before the analysis window are also classified as having HIV-RNA  $\geq$ 50 copies/mL.

Missing viral load values for reasons related to COVID-19 issues (e.g. participant is unable to have viral load assessed due to barriers in attending the clinic during the pandemic or COVID-19 related adverse events leading to treatment discontinuation) will

be considered as random missingness and classified the same as all other missingness for the primary efficacy Snapshot analysis. A sensitivity analysis using a modified Snapshot which includes subcategories for Covid-19 related and Non-Covid-19 related missingness will also be performed to display the impact of Covid-19 intercurrent events on the study. See <u>Appendix 8</u> for Modified Snapshot Algorithm details.

### 7.1.4. Statistical Analyses / Methods

Details of the planned displays are provided in <u>Appendix 12</u>: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in <u>Section 7.1.1</u> will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 7.1.4.1. Statistical Methodology Specification

#### **Endpoint / Variables**

- Proportion of participants with plasma HIV-1 RNA < 50 c/mL at Month 12 using the FDA Snapshot algorithm (Safety population)
- Proportion of participants with plasma HIV-1 RNA ≥50 c/mL at Month 12 using the FDA Snapshot algorithm (Safety population)
- Proportion of participants with protocol-defined confirmed virologic failure (CVF) over time (Safety population)
- Incidence of treatment-emergent genotypic and phenotypic resistance to CAB and RPV in patient study participants with CVF (Safety population)

#### **Results Presentation**

- The proportion of participants with HIV-1 RNA <50 c/mL, HIV-1 RNA ≥ 50c/mL, and with recorded CVF at each planned visit with corresponding 95% confidence intervals calculated using the Clopper-Pearson exact method.
- Proportion of subjects with incidence of treatment-emergent genotypic and phenotypic resistance to CAB and RPV in patient study participants with CVF at each visit with corresponding 95% confidence intervals calculated using the Clopper-Pearson exact method.
- Descriptive statistics for the nominal values and change from baseline values in CD4+ cell counts and the CD4/CD8 ratio.

#### **Subgroup Analyses**

- Summary of study outcomes will be repeated for subgroups of interest as specified in Section 5.4.2: Implementation strategy, Participant sex, age group (<50 vs ≥50), race (White, African Heritage, Asian, Other), and CD4 count (<350, ≥350).
- The proportion of participants in each Snapshot study outcome category and sub-category will be summarized in which default sub-categories have been expanded to present Covid-19 vs. Non-Covid-19 related impact (as described in Appendix 8).

#### 8. SAFETY ANALYSES

The safety analyses will be based on the Safety and Long Term Follow-up (LTFU) populations, unless otherwise specified.

For the interim analyses, adherence to dosing will be reported for the Safety population. For the Month 12 primary analysis, outputs will be presented for the Safety population in the Intervention Phase unless otherwise specified. For the EOS analysis, outputs will be presented for the Safety population in the Intervention and Extension phases as well as for the LTFU population in the LTFU phase.

For the Month 12 analysis, a set of separate outputs will also be presented for the oral lead-in period, including a summary of adverse events, SAEs, AEs leading to withdrawal, post-baseline emergent chemistry/haematology abnormalities, and subjects with hepatobiliary abnormality criteria.

## 8.1. Safety Endpoints

Secondary and tertiary safety endpoints for this study include:

- Percentage of injections occurring within target window from the target date.
- Incidence and severity of AEs and SAEs over time



## 8.2. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs), Drug-related AEs, AEs leading to withdrawal, AEs by maximum severity, COVID-19 AEs, and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in <u>Appendix 12</u>: List of Data Displays.





## 8.3. Adverse Events of Special Interest Analyses

A comprehensive list of MedDRA terms based on clinical review will be used to identify Adverse Events of Special Interest (AESI). Changes to the MedDRA dictionary may occur between the start of the study and the time of reporting and/or emerging data from on-going studies may highlight additional adverse events of special interest, therefore the list of terms to be used for each event of interest and the specific events of interest will be based on the safety review team (SRT) agreements in place at the time of reporting. The details of the current planned grouping, including Standardized MedDRA Query (SMQ) values (as applicable), and planned displays are provided in <u>Appendix 9</u>: AESI identification and <u>Appendix 12</u>: List of Data Displays.

## 8.4. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests and Hematology laboratory tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 12: List of Data Displays.

# 8.5. Other Safety Analyses

The analyses of injections in the target window as well as non-laboratory safety test results including vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in <u>Appendix 12</u>: List of Data Displays.

## 9. PHARMACOKINETIC ANALYSES

# 9.1. Endpoint / Variables

## 9.1.1. Drug Concentration Measures

Available concentration-time data for CAB and RPV will be presented in listings as specified in <a href="Appendix 12">Appendix 12</a>: List of Data Displays and will be based on GSK Data Standards and statistical principles

# 10. VIROLOGY

# 10.1. Genotypic and Phenotypic Data

Available genotypic and phenotypic data at all collection timepoints will be presented by subject (separately for CVF and Non-CVF subjects), as specified in <u>Appendix 12</u>: List of Data Displays.

## 11. OTHER ANALYSES

## 11.1. Endpoint / Variables

#### 11.1.1. Study Visit length

Study Visit Length will be reported for all analyses including interim analyses, Month 12, and EOS. Details of the planned displays for study visit length data are provided in <a href="Appendix 12">Appendix 12</a> List of Data Displays and will be based on GSK Data Standard and statistical principle.

#### 11.1.2. Pregnancy

Protocol amendment 02 allows for pregnant participants to remain on study and continue the use of study drug. Should any participants become pregnant while on study drug, pregnancy specific listings will be produced. Listings will include any adverse events, clinical lab results including HIV-1 RNA and plasma CAB & RPV concentrations, exposure to study drug during pregnancy, and pregnancy details including duration and outcomes reported by the participants including birth outcomes. Details of the planned displays are provided in Appendix 12

## 12. REFERENCES

GSK document number 2019N420690\_01. A Phase IIIb, open-label, hybrid type III trial evaluating implementation strategies for long-acting cabotegravir plus long-acting rilpivirine every two months in HIV-1 infected, virologically suppressed adults in select European healthcare settings.

GSK document number 2019N420690\_02. A Phase IIIb, open-label, hybrid type III trial evaluating implementation strategies for long-acting cabotegravir plus long-acting rilpivirine every two months in HIV-1 infected, virologically suppressed adults in select European healthcare settings.

Wensing AM, et al. 2019 update of the drug resistance mutations in HIV-1. *Topics in antiviral medicine*. 2019;27:111-121.

# 13. APPENDICES

# 13.1. Appendix 1: Schedule of Activities

The protocol also lists a schedule of activities for staff study participants (not listed here)

## 13.1.1. Protocol Defined Schedule of Events: Schedule of Activities for Patient Study Participants

| | | | | | Interven | tion Period | (Month) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screening <sup>a</sup><br>up to 35d | Day 1 | Month<br>1 | Month 2 | Month<br>4 | Month<br>6 | Month<br>8 | Month 10 <sup>b</sup> | Month 12 b | Withdrawal <sup>m</sup> | Long Term<br>Follow-up <sup>n</sup> |
| | ng <sup>a</sup><br>5d | Oral<br>Lead-<br>in | Dose 1<br>(D1) | Dose 2<br>(D2) | Dose 3 (D3) | Dose 4<br>(D4) | Dose 5<br>(D5) | Dose 6<br>(D6) | Dose 7<br>(D7) | ıwal <sup>m</sup> | Term<br>w-up <sup>n</sup> |
| Written Informed consent | X | | | | | | | | | | |
| Eligibility Verification | X | | | | | | | | | | |
| Demography | X | | | | | | | | | | |
| Physical Exam | X | | | | | | | | | | |
| Medical history | X | | | | | | | | | | |
| Current medical conditions | X | | | | | | | | | | |
| Center for Disease Control and<br>Prevention (CDC) HIV-1<br>Classification | X | | | | | | | | | | |

| | Procedure | Screening <sup>a</sup><br>up to 35d | Intervention Period (Month) | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Day 1 | Month<br>1 | Month 2 | Month 4 | Month<br>6 | Month<br>8 | Month 10 b | Month 12 b | Withdrawalm | Long Term<br>Follow-up <sup>n</sup> |
| | | | Oral<br>Lead-<br>in | Dose 1<br>(D1) | Dose 2<br>(D2) | Dose 3<br>(D3) | Dose 4<br>(D4) | Dose 5<br>(D5) | Dose 6<br>(D6) | Dose 7<br>(D7) | walm | rm<br>Ip" |
| | Syphilis serology + reflex<br>Rapid Plasma Reagin (RPR) | X | | | | | | | | | | |
| CI | | | | | | | | | | | | |
| | Symptom Directed Physical<br>Exam and Medical<br>Assessment | | X | X | | X | | X | | X | X | X |
| | HIV-associated Conditions,<br>AE and serious adverse event<br>(SAE) Assessments <sup>d</sup> , Con<br>Meds | X | X | X | | X | | X | | Х | X | X |
| | Vital Signs<br>(blood pressure [BP], heart<br>rate [HR]) <sup>e</sup> | X | X | X | | x | | X | | X | X | |
| | Weight, Height & body mass index (BMI) <sup>f</sup> | X | X | X | | x | | X | | X | X | |
| | Clinical Chemistry,<br>Hematology and other Tests° | X | X | X | X | X | | X | | X | X | X |

| | | Intervention Period (Month) | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screening <sup>a</sup> up to 35d | Day 1 | Month<br>1 | Month 2 | Month<br>4 | Month<br>6 | Month<br>8 | Month 10 b | Month 12 b | Withdrawalm | Long Term<br>Follow-up <sup>n</sup> |
| | <u> </u> | Oral<br>Lead-<br>in | Dose 1<br>(D1) | Dose 2<br>(D2) | Dose 3 (D3) | Dose 4<br>(D4) | Dose 5 (D5) | Dose 6<br>(D6) | Dose 7<br>(D7) | | |
| HIV-1 RNA and plasma sample for storage <sup>h</sup> | X | X | X | X | X | | X | | X | X | X |
| CD4+ count | X | X | X | X | X | | X | | X | X | X |
| CD8+ cell count (will be reported at Baseline and Month 12) | | X | | | | | | | X | | |
| Urinalysis | X | | | | | | | | | X | X |
| Hepatitis Serology <sup>q</sup> | X | | | | | | | | | | |
| Whole Blood PBMC <sup>p</sup> | | X | | | | | | | | X | |
| Prothrombin time (PT)/ partial thromboplastin time (PTT)/international normalized ratio (INR) | X | | | | | | | | | X | X |
| Pregnancy Testing<br>Urine (U) or Serum <sup>g</sup> | U | U | U | U | U | U | U | U | U | U | U |
| Notification of Interview <sup>t</sup> | | X | | | | | | | | | |

| | Screening <sup>a</sup><br>up to 35d | Intervention Period (Month) | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | | Day 1 | Month<br>1 | Month 2 | Month<br>4 | Month<br>6 | Month<br>8 | Month 10 <sup>b</sup> | Month 12 b | Withdrawal <sup>m</sup> | Long Term<br>Follow-up <sup>n</sup> |
| | | Oral<br>Lead-<br>in | Dose 1<br>(D1) | Dose 2<br>(D2) | Dose 3 (D3) | Dose 4<br>(D4) | Dose 5 (D5) | Dose 6<br>(D6) | Dose 7 (D7) | | |
| Oral CAB + RPV Medication<br>Dispensation | | X | | | | | | | | | |
| CAB LA + RPV LA IM<br>Treatment Administration <sup>i</sup> | | | X | X | X | X | X | X | X | | |
| Participant Visit Reminder<br>Contact | X | X | X | X | X | X | X | X | | | |
| Participant Contact Detail<br>Confirmation | X | X | X | X | X | X | X | X | | | |
| Patient Toolkits | | X | X | X | X | | | X | | | |
| Record Visit Length <sup>j</sup> | | | X | X | | X | X | | | | |
| Contraception Counseling <sup>u</sup> | | | | | | | | | | X | X |
| HAART dispensation <sup>v</sup> | | | | | | | | | | X | X |
| Patient Questionnaires <sup>k</sup> | | | X | | X | | | | X | | |
| Selected Patient Interviews <sup>1</sup> | | X | | | | | | | X | | |

| | | Intervention Period (Month) | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screening <sup>a</sup> up to 35d | Day 1 | Month<br>1 | Month 2 | Month<br>4 | Month<br>6 | Month<br>8 | Month 10 b | Month 12 b | Withdra | Long Term<br>Follow-up <sup>n</sup> |
| | 3d 3g | Oral<br>Lead-<br>in | Dose 1<br>(D1) | Dose 2<br>(D2) | Dose 3<br>(D3) | Dose 4<br>(D4) | Dose 5<br>(D5) | Dose 6<br>(D6) | Dose 7<br>(D7) | walm | -ip" |
| HIV and patient satisfaction (HIVTSQs) | | Xr | X | | X | | | | X | | |
| HIVTSQc | | | | | | | | | X | | |
| Preference Question | | | | | | | | | X | | |

- a) A screening visit will be conducted within 35 days of Day 1. However, it is preferred for Day 1 to be conducted as soon as practical after all screening results are available.
- b) Continue this pattern for visits for the remainder of the study if needed, until CAB LA + RPV LA is locally approved and available. For example, Dose 8 will be conducted as per Dose 6, Dose 9 will be conducted as per Dose 6 and so on. The exception to this pattern is that no questionnaires, study visit length collection, or patient interviews will be conducted after Dose 7 visit. See protocol Section 6.8.
- c) Physical exams should be conducted as part of normal routine clinical care but data will not be collected in the electronic case report form (eCRF) unless abnormalities are observed. Medical assessments include any decisions the study staff must make for participant management.
- d) AE and SAEs will not be proactively assessed at M 2, M 6 and M 10. However, all AEs and SAEs reported by study participants **must** be recorded in eCRF at all visits and reported within required timelines as per protocol Section 8.5.1.
- e) Measure vital signs after about 5 minutes of rest in a semi-supine position.
- f) Height is collected at screening only.
- g) A (-) urine pregnancy test is required prior to oral lead-in at day 1 and prior to any injection and as required by Medical Monitor after a treatment interruption. A (+) urine test should be confirmed with a stat serum test. If (+), participant will need to be withdrawn. A Serum pregnancy test should be performed at any time pregnancy is suspected by the Investigator. Pregnant participants who remain in the study do not need pregnancy testing for the duration of the pregnancy See Protocol Appendix 15: Information and Guidance for Managing Pregnant Participants.
- h) Plasma for storage samples are collected for possible future analyses. Can be used for back-up in cases of loss/damage in transit, geno/pheno analyses for virologic failures. Only for women becoming pregnant and continuing on CAB LA+RPV LA as if pregnant a plasma HIV-1 RNA test and plasma for storage samples at Month 6 and Month 10 visits are required.
- i) All injections are 1 x CAB LA 600 mg IM + 1 x RPV LA 900 mg IM. Doses 1 and 2 are one month apart. Subsequent injections beginning at Dose 3 are every two months. The injections should be spaced approximately 2 cm from one another and from the site of any previous injection and/or any injection site
reaction. Bring RPV LA to approximately room temperature prior to injecting. Time and location of injection (right or left) as well as needle length used will be collected in the eCRF. IM dosing is expected to occur on the same date of the month as determined by IM Dose 1 visit date, this is the Target Date; where possible, this first injection should be performed within 2 hours of taking the last oral regimen dose. For Dose 2, a dosing window of +0 / -7 days from the target visit date is stipulated. A (+ or -) 7-day window from the target date visit is stipulated for IM dosing beginning at Dose 3. All decisions regarding dose interruption/ resumption must be discussed with the Medical Monitor in advance.

- j) Length of study visit from arrival until departure from clinic will be evaluated. Participant's time of arrival, actual start time of the appointment, and actual end time of the appointment will be collected in the eCRF.
- **k)** Questionnaires should be completed before receiving the injections.
- Interviews should be conducted before the PSP receives Dose 1 and within 4 weeks of receiving Dose 7. Interviews may be done in person, virtually, or by phone. A minimum of 6 patients per site will be selected for interviews.
- m) Withdrawal Visit Conduct ~4 weeks after the last dose of investigational product (IP) if not entering Long-Term Follow Up and only if the participant has ongoing AEs or lab abnormalities at the last on-study visit. May be conducted by telephone.
- n) Participants receiving one or more injections with CAB LA and/or RPV LA will be assessed with clinic visits at months 3, 6, 9 and 12 during the Long-Term Follow-Up phase. The start of the 52-week follow-up period begins the day of the last CAB LA and/or RPV LA dose.
- o) See protocol Section 8.4.4 for list of tests
- p) Whole blood/PBMC collection samples may be used for virologic analyses. PBMCs will be collected at baseline Dayl and at Withdrawal.
- q) Hepatitis B (HBsAg), Anti-HBc, Anti-HBsAg, Hepatitis C (anti-HCVAb). A (+) anti-HCVAb will be followed by a confirmatory nucleic acid test for HCV RNA. HBV DNA will only be performed for participants with a (+) anti-HBc and (-) HBsAg and (-) anti-HBs (past and/or current evidence).
- r) Administer HIVTSQs in Day 1 before OLI initiation.
- s) At a minimum the study toolkit will be offered at the time pointed noted in the protocol Table 6. However, the toolkit items are intended to be used throughout the study.
- t) Notification of interviews may occur between Day 1 or during the 7 days after Day 1.
- women of childbearing potential should continue to receive counselling on the need to use adequate contraception for the entirety of the Long-Term Follow-Up period.
- v) Investigators must discuss choice of HAART regimen and timing of initiation with the Medical Monitor before initiating.

# 13.2. Appendix 2: Assessment Windows

# 13.2.1. Definitions of Assessment Windows for Analyses

Laboratory data, vital signs, adverse events, and genotypic/phenotypic data will be assigned to assessment windows according to actual dates rather than the nominal visit labels as recorded on the eCRF or in the laboratory database.

Prior to visit slotting, assessments are first assigned to a study phase (Screening, Intervention Phase, Extension, or Long Term Follow Up) as defined in <u>Appendix 3</u>.

According to the protocol, the nominal target study visit date will be based on the first injection, the Month 1 date. For instance, if Month 1 occurred on July 7th, all subsequent visits are expected to occur on the 7th of each month such that subsequent visits will be August 7th, September 7th, October 7th, etc. Since there are not >28 days in every month of the year, if the Month 1 injection occurred on the 29th, 30th, or 31st of the month, then the target study visit date for the remainder of the visits will be the 28th of the month.

The nominal target study visit day is derived as

- M1 Target Day = Date of Actual M1 Injection Visit Date Date of First Oral lead-in Dose + 1, if subject receives M1 injection; else M1 Target Day = 30.
- Mx Target Day = Mx Nominal Target Study Visit Date Date of First Oral lead-in Dose + 1, for x=2,3, ...

Assessment windows will be derived based on the midpoint between two consecutive planned target study visit dates. For the Snapshot efficacy data, the same approach will be used, except for Month 12, which will use a +/- 6-week window around the projected target study visit date at Month 12.

For parameters which are not scheduled to be assessed at visits, the all-inclusive assessment windows will still be used; however, data summaries will only report scheduled visits. Assessments at unscheduled visits will be included in summaries of worst-case values across visit (e.g. during the intervention phase) and in data listings, as well any algorithms that make use of additional data (e.g., Snapshot).

For participants transitioning to commercial product at EOS, the safety follow-up visit date will be the last date referenced and serve as the ending timepoint for the final visit window.

Table 1 Assessment Windows for Screening, Intervention and Extension Phase Data (Excluding HIV-1 RNA)

| Target | Analysis Window | | Analysis |
|---|---|---|---|
| (Study<br>Day) | Beginning Timepoint | Ending Timepoint | Timepoint |
| Day of earliest record | Assessment Stud | dy Day ≤1 | Screening |
| | For subjects discontinuing prior t | o receiving first injection: | |
| 30 | Assessment Study Day = 2 | Study Day of Last CAB/RPV<br>Oral Dose+1 | Month 1 |
| | Assessment Stu<br>(Study Day of Last CAB/RPV | • • | Follow-up |
| | For subjects receiving | ı first injection: | |
| Day of First<br>Injection | Study Day = 2 | M1 target day + floor [(M2 target day – M1 target day)/2] | Month 1 |
| M2<br>Target Day | M1 target day + floor [(M2 target day - M1 target day)/2] + 1 | M2 target day + floor [(M4 target day – M2 target day)/2] | Month 2 |
| M4<br>Target Day | M2 target day + floor [(M4 target day – M2 target day)/2] + 1 | M4 target day + floor [(M6 target day – M4 target day)/2] | Month 4 |
| M6<br>Target Day | M4 target day + floor [(M6 target day<br>– M4 target day)/2] + 1 | M6 target day + floor [(M8 target day – M6 target day)/2] | Month 6 |
| M8<br>Target Day | M6 target day + floor [(M8 target day – M6 target day)/2] + 1 | M8 target day + floor [(M12 target day – M8 target day)/2] | Month 8 |
| M10<br>Target Day | M8 target day + floor [(M10 target day – M8 target day)/2] + 1 | M10 target day + floor [(M12<br>target day – M10 target<br>day)/2] | Month 10 |
| M12<br>Target Day | M10 target day + <i>floor</i> [(M12 target day – M10 target day)/2] + 1 | M12 target day + floor [(M14<br>target day – M12 target<br>day)/2] | Month 12 |
| M <b>x</b><br>Target Day | M(x-2) target day - floor [(Mx target day - M(x-2) target day)/2] + 1 | M <b>x</b> target day + floor<br>[(M( <b>x+2</b> ) target day – M <b>x</b><br>target day)/2] | Month <b>x</b> For <b>x</b> = 14, 16, etc. |
| For subjects who permanently discontinue study treatment: | | | |
| | Assessment Study Day > Min (LTFU ART Start Date, Max (Study Day of Last Dose of Oral Study Treatment (CAB+RPV or SOC Bridging) + 1, Study Day of Last CAB + RPV Injection + 63)) | | |

Table 2 Assessment Windows for Screening and Intervention Phase HIV-1 RNA Data

| Target | Analysis Window | | |
|---|---|---|---|
| (Study Day) | Beginning Timepoint Ending Timepoint | | Timepoint |
| Day of earliest record | Assessment Study Day ≤1 | | Screening |
| | For subjects discontinu | uing prior to receiving first injection | n: |
| 28 | Assessment Study Day = 2 | Study Day of Last Oral Lead-<br>in Dose +1 | Month 1 |
| | Assessment<br>(Study Day of Last CAB/F | Study Day ><br>RPV Oral Lead-in Dose +1) | Follow-up |
| | For subjects | s receiving first injection: | |
| Date of First<br>Injection | Study Day = 2 | M1 target day + floor [(M2 target day – M1 target day)/2] | Month 1 |
| M2 Target Day | M1 target day + floor [(M2<br>target day – M1 target day)/2]<br>+1 | M2 target day + floor [(M4 target day – M2 target day)/2] | Month 2 |
| M4 Target Day | M2 target day + floor [(M4<br>target day – M2 target day)/2] +<br>1 | M4 target day + <i>floor</i> [(M6 target day – M4 target day)/2] | Month 4 |
| M6 Target Day | M4 target day + floor [(M6 target day - M4 target day + 1 | M6 target day + floor [(M8 target day – M6 target day)/2] | Month 6 |
| M8 Target Day | M6 target day + floor [(M8 target day – M6 target day)/2] + | M8 target day + floor [(M10 target day – M8 target day)/2] | Month 8 |
| M10 Target<br>Day | M8 target day + floor [(M10 target day – M8 target day)/2] + | M12 target day – 43 | Month 10 |
| M12 Target<br>Day | M12 target day - 42 | M12 target day + 42 | Month 12 |
| M14 Target<br>Day | Assessment Study Day > M12 target day + 42 | | Month 14 |
| For subjects who permanently discontinue study treatment during the Intervention Phase: | | | |
| | Assessment Study Day > Min (LTFU ART Start Date, Max (Study Day of Last Dose of Oral Study Treatment (CAB+RPV or SOC Bridging) +1, Study Day of Last CAB + RPV Injection + 63)) | | Follow-up |

Table 3 Assessment Windows for Extension Phase HIV-1 RNA Data

| Target | Analysis | Analysis | |
|---|---|---|---|
| (Study Day) | Beginning Timepoint | Ending Timepoint | Timepoint |
| M14 Target | Study Day of Nominal Week 14 | M14 target day - floor [(M16 | Month 14 |
| Day | Visit | target day – M14 target day)/2] | |
| M16 Target | M14 target day - <i>floor</i> [(M16 | M16 target day + <i>floor</i> [(M18 | Month 16 |
| Day | target day – M14 target day)/2] | target day – M16 target day)/2] | |
| | + 1 | | |
| M <b>x</b> Target Day | M( <b>x-2)</b> target day - floor [(M <b>x</b> | Mx target day + floor [(M(x+2) | Month x |
| | target day – M( <b>x-2</b> ) target | target day – M <b>x</b> target day)/2] | For <b>x</b> =18, |
| | day)/2] + 1 | | 20 etc. |
| For subjects who permanently discontinue study treatment during the Extension Phase: | | | |
| | Assessment Study Day > | | Follow-up |
| | Min (LTFU ART Start Date, Max (Study Day of Last Dose of Oral | | |
| | Study Treatment (CAB+RPV or SOC Bridging) +1, Study Day of | | |
| | Last CAB + RPV Injection + 63)) | | |

Table 4 Assessment Windows for Study Visit Length Data (Intervention and Extension Phase)

| Target | Analysis Window | | Analysis |
|---|---|---|---|
| (Study Day) | Beginning<br>Timepoint | Ending Timepoint | Timepoint |
| Study Day of Actual M1 Injection | Study Day of Ad | ctual M1 Injection | Month 1 |
| Study Day of Actual M2<br>Injection | Study Day of Actual M2 Injection | | Month 2 |
| Study Day of Actual M6<br>Injection | Study Day of Actual M6 Injection | | Month 6 |
| Study Day of Actual M8<br>Injection | Study Day of Actual M8 Injection | | Month 8 |
| Study Day of Actual M <b>x</b> Injection | Study Day of Actual Mx Injection | | Month <b>x</b> For <b>x</b> =17, 20, etc. |
| | If none of the above, then Analysis Timepoint = Other | | |

Table 5 Assessment Windows for Summaries of Long-Term Follow-up
Phase Data from Subjects who Received at Least One Injection of
CAB+RPV and Permanently Discontinued from the Study

| Day of Assessment | Assessment Window | Target LTFU Study Day of Window |
|---|---|---|
| 1 ≤ LTFU Study Day ≤ 135 | LTFU Month 3 | 90 |
| 136≤ LTFU Study Day ≤ 225 | LTFU Month 6 | 180 |
| 226 ≤ LTFU Study Day ≤ 315 | LTFU Month 9 | 270 |
| 316 ≤ LTFU Study Day ≤ 405 | LTFU Month 12 | 360 |
| (30*m-44) ≤ LTFU Study Day ≤ | LTFU Month m | 30*m |
| (30*m+45) | M = 15, 18, 21 | |

<sup>•</sup> LTFU Study Day is defined in 13.5.1

# 13.2.2. Assessment Windows for PK Concentration Data

PK data will be presented in data listings according to planned nominal visits (i.e. as collected in the eCRF), without additional assignment to assessment windows.

# 13.2.3. Assessment Windows for Pregnancy Data

Pregnancy visits will be assigned in accordance with the derivations listed in Table 1 to Table 5 as appropriate for the relevant data. Post-partum visit data will be labelled based on the nominal timepoint

# 13.3. Appendix 3: Study Phases

# 13.3.1. Study Phases

Participants are considered to have entered the Extension phase if they have a Month 14 visit. They are considered to enter the LTFU period if they have a post-treatment, non-bridging ART start date or LTFU visit entered in the CRF, including LTFU withdrawal.

Participants are considered to have completed the Intervention Phase upon successful completion of the Month 12 visit without discontinuing from study treatment. Extension Phase completion is defined as successful transition to commercial product whenever it becomes available by attending a Safety Follow-up visit and not discontinuing treatment.

Table 6 Participant Phase Entry and Conclusion Windows

| Phase | Qualifying Entry<br>Timepoint | Qualifying Conclusion Timepoint |
|---|---|---|
| Intervention<br>Phase | First CAB + RPV dose date | Month 14 visit date; or Safety Follow-up visit date (if transitioned to commercial product); or LTFU ART start date (if discontinued from treatment after receiving at least one dose of CAB/RPV LA) |
| Extension Phase | Month 14 visit date | Safety Follow-up visit date (if transitioned to commercial product); or LTFU ART start date (if discontinued from treatment after receiving at least one dose of CAB/RPV LA) |
| LTFU Phase | LTFU ART start date or LTFU Visit date existence | LTFU Month 12 visit date |

AEs will be assigned to study phases as defined in Table 7. Laboratory data (efficacy, safety, and virology), HIV associated Conditions, health outcomes assessments, and vital signs will be assigned to study phases as defined in Table 8.

Assessments/events are assigned to study phases sequentially, starting from the top of each table.

Table 7 Study Phases for AEs

| Study Phase | Definition |
|---|---|
| Screen | Date < Intervention Phase Treatment Start Date |
| Intervention Phase | For subjects continuing into the Extension Phase: Intervention Phase Treatment Start Date ≤ Date < Date of Nominal Month 14 Visit |
| | For subjects not continuing into the Extension Phase: Intervention Phase Treatment Start Date ≤ Date < LTFU ART Start Date[a] |

| Study Phase | Definition |
|---|---|
| | For subjects transitioning to commercial product without discontinuing or entering Extension: |
| | Intervention Phase Treatment Start Date ≤ Date ≤ Safety Follow-up visit date |
| | For AEs leading to treatment withdrawal with start date equal to the LTFU ART Start Date, Intervention Phase instead of Long-term Follow-up Phase will be assigned. |
| Extension Phase | For subjects transitioning to commercial product: |
| | Date of Nominal Month 14 Injection ≤ Date ≤ Safety Follow-up visit date |
| | For subjects not transitioning to commercial product: |
| | Date of Nominal Month 14 Injection ≤ Date < LTFU ART Start Date [a] |
| | For AEs leading to treatment withdrawal with start date equal to the LTFU ART Start Date, Extension Phase instead of Long-Term Follow-up Phase will be assigned. |
| Long Term Follow- | For subjects who receive at least one CAB/RPV injection and permanently |
| Up | discontinue study treatment: |
| | AE Start Date ≥ LTFU ART Start Date |
| AEs with completely | missing start date: |

- If AE end date is ≤ Intervention Phase Treatment Start Date, then assign to Screening Phase;
- Else if AE end date is completely missing or Intervention Phase Treatment Start Date < AE end date 

  Date of Nominal Month 14 Injection, then assign to Intervention Phase;
- Else if AE end date > Date of Nominal Month 14 Injection, then assign to Extension Phase.
- Date=AE Start Date
- [a] If participants have missing LFTU ART start date, only the lower bound will be considered in the derivation.

Study Phases for Laboratory, Vital Signs, HIV-1 Associated Table 8 **Conditions, and Protocol Deviation Data** 

| Study Phase | Definition |
|---|---|
| Screen | Date ≤ Study Treatment Start Date |
| Intervention Phase | For subjects continuing into the Extension Phase: |
| | Intervention Phase Treatment Start Date < Date < Date of Nominal Month 14 Visit |
| | For subjects not continuing into the Extension Phase: |
| | Intervention Phase Treatment Start Date < Date ≤ LTFU ART Start Date [a] |
| | For subjects transitioning to commercial product without discontinuing or entering Extension: |
| | Intervention Phase Treatment Start Date < Date ≤ Safety Follow-up visit date |
| Extension Phase | For subjects continuing into Extension Phase: |
| | Date of Nominal Month 14 Visit ≤ Date ≤ LTFU ART Start Date [a] or Safety Follow-<br>up visit date |
| Long Term Follow- | For subjects who receive at least one CAB/RPV injection and permanently |
| Up | discontinue study treatment: |
| | Assessment Date > LTFU ART Start Date |

- Date = start or assessment date
- [a] If participants have missing LFTU ART start date, only the lower bound will be considered in the derivation.

Study phase of discontinuation will be determined according to Table 9.

Table 9 Study Phases for Study Conclusion/IP Discontinuation

| Study Phase | Definition |
|---|---|
| Intervention Phase | Discontinuation Date is not missing, and no assessments collected at any extension phase nominal visits (i.e. Month 14, Month 16, Month 18 etc.). |
| Extension Phase | Discontinuation Date is not missing, and assessments collected at any extension phase nominal visits (i.e. Month 14, Month 16, Month 18 etc.). |

<sup>•</sup> Discontinuation Date = date of failure to complete study/date of IP discontinuation

Medication use will be classified as prior and concomitant with study treatment according to Table 10, noting that a medication can be assigned as "taken" during more than one study phase.

Table 10 Study Phases for Non-ART Medications/ART Medications

| | Definition |
|---|---|
| Prior | Medication Taken < Intervention Treatment Start Date |
| Concomitant during | For subjects continuing into Extension Phase: |
| Intervention Phase | Intervention Treatment Start Date <sup>[a]</sup> ≤ Medication Taken < Date of Nominal Month 14 Visit |
| | For subjects not continuing into Extension Phase <sup>[b]</sup> : |
| | Intervention Treatment Start Date[a] ≤ Medication Taken < LTFU ART Start Date |
| | For subjects transitioning to commercial product without discontinuing or entering Extension: |
| | Intervention Phase Treatment Start Date ≤ Medication Taken ≤ Safety Follow-up visit date |
| Concomitant during | For subjects transitioning to commercial product: |
| Extension Phase | Date of Nominal Month 14 Injection ≤ Medication Taken ≤ Safety Follow-up visit date |
| | For subjects not transitioning to commercial product: |
| | Date of Nominal Month 14 Injection ≤ Medication Taken < LTFU ART Start Date |
| Received during | For subjects who received at least one CAB and/or RPV injection and have |
| Long-term Follow-up | started LTFU ART: |
| | Medication Taken ≥ LTFU ART Start Date |

#### NOTES:

- Please refer to <u>Appendix 6</u>: Reporting Standards for Missing Data for handling of missing and partial dates for medications. Use the rules in this table if medication date is completely missing.
- a. The ART medication stopped on start date of Intervention treatment will be considered a prior medication and will not be considered concomitant during the Intervention phase. If the stop date of ART medication is completely missing and this medication is recorded in eCRF as prior, it will be considered a prior medication and will not be considered concomitant during the intervention phase.
- b. If subjects have missing LFTU ART start date, only the lower bound will be considered in the derivation.

#### 13.3.2. Treatment State

Within each study phase (based on assignment of study phase described in <u>Section 13.3.1</u>), only those events/assessments which occur within the ranges shown in Table 11 will be considered 'on-treatment' for the given phase. No treatment states will be assigned to medications.

For adverse events, partial AE start date will use imputation as described in 13.6.2.1.

Table 11 Treatment State within Study Phases

| Study Phase | State | Definition |
|---|---|---|
| Screen | Pre-Treatment | All assessments/events within phase |
| Intervention/Extension | On-treatment | Date ≤ max (Date of Last CAB LA +RPV LA IM Dose + 63, Date of Last Dose of Oral Study Treatment (CAB+RPV or SOC Bridging) +1) |
| | Post-Treatment | Date > max (Date of Last CAB LA +RPV LA IM Dose + 63, Date of Last Dose of Oral Study Treatment (CAB+RPV or SOC Bridging) +1) |
| Long Term Follow-Up | Post-Treatment | All assessments/events within phase |

#### NOTES:

- Date = Assessment/Start Date
- a. Treatment State is determined after data has been assigned to the study phases as defined in Section 13.3.1.
- b. Last injection and/or last dose of oral study treatment (CAB+RPV or SOC bridging) are only applied to participants who permanently discontinued the study treatment. The assessments for participants who did not permanently discontinue the study treatment will be considered 'On-treatment'. For participants continuing into extension phase, all data assigned to intervention phase per Section 13.3.1 will be considered 'On-treatment'.

#### 13.3.3. Oral Lead-in Period

Certain displays will be produced for data collected or events occurring during the oral-lead-in period as defined in Table 12 and Table 13.

Table 12 Oral Lead-in Period for AEs

| Study Period | Date Range |
|---|---|
| Oral Lead-in | For participants receiving at least one Injection: |
| | Intervention Treatment Start Date ≤ Date [a] < Date of First IM Injection |
| | For participants withdrawing prior to first Injection: Date ≥ Intervention Treatment Start Date |
| | Note that the oral lead-in period is only applicable to the participants who received at least one dose of study treatment during the oral lead-in period in the study. Oral lead-in period is within the intervention phase. |
| | tely missing start date which have been assigned to the Intervention Phase based on Table 7 to the Oral Lead-in Period. |

#### NOTES:

Date = AE Start date

Table 13 Oral Lead-in Period for Laboratory Data

| Period | Date Range |
|---|---|
| Oral Lead-in | For participants receiving at least one Injection: Intervention Treatment Start Date < Date ≤ Date of First IM Injection |
| | For participants withdrawing prior to first Injection: Date > Intervention Treatment Start Date |
| | Note that the oral lead-in period is only applicable to the participants who received at least one dose of study treatment during the oral lead-in period in the study. Oral lead-in period is within the intervention phase. |

# NOTES:

• Date = Date of assessment

# 13.4. Appendix 4: Data Display Standards & Handling Conventions

# 13.4.1. Reporting Process

| Software | |
|---|---|
| The currently sup- | The currently supported versions of SAS software will be used. |
| Reporting Area | |
| HARP Server | us1salx00259 |
| HARP Compound | \ARPROD\GSK1265744\mid213199\interim_01 |
| | \ARPROD\GSK1265744\mid213199\interim_02 |
| | \ARPROD\GSK1265744\mid213199\primary_01 |
| Analysis Datasets | |

- Analysis datasets will be created for the interim analyses according to SI data standards.
- Analysis datasets will be created for the Month 12 reporting effort according to CDISC standards (SDTM IG Version 3.2 & ADaM IG Version 1.1).

#### Generation of RTF Files

RTF files will be generated for all reporting efforts described in the RAP.

## 13.4.2. Reporting Standards

#### General

- The current GSK Statistical Display Standards in the GSK Standards Library (IDSL) will be applied for reporting, unless otherwise stated (Library Location:
  - https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- GSK Statistical Display Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the GSK Standard Statistical Display Principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to GSK Standard Statistical Display Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the participant's listings.

#### **Unscheduled Visits**

- Unscheduled visits will be assigned to an analysis visit using the all-inclusive windows defined in <u>Section 13.2</u>.
- However, data summaries will only report visits that are planned assessment time points for each parameter (according to the Schedule of Activities in <u>Section 13.1.1</u>).
- Evaluable assessments at unscheduled visits will be used when categorizing values across
  visits, such as 'maximum grade during the intervention phase' or 'at any time postbaseline', and for any algorithm that has specific rules for which observation to use (e.g.
  snapshot algorithm or CVF identification).

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data | Refer to GSK Standard Statistical Display Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| Refer to GSK Standard Statistical Display Principals 7.01 to 7.13. | |

# 13.4.3. Reporting Standards for Pharmacokinetic Data

| Pharmacokinetic Concentration Data | |
|---|---|
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to the GSK Standard PK Display Standard. Refer to the GSK Standard Statistical Display Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive |
| | summary statistics/analysis and summarized graphical displays only. |

# 13.5. Appendix 5: Derived and Transformed Data

#### 13.5.1. General

#### **Multiple Measurements at One Analysis Time Point**

- If there are two values within a time window (as per <u>Section 13.2.1</u>) the value closest to the target day for that window will be used. If values are the same distance from the target, then the mean (geometric mean for HIV-1 RNA, arithmetic mean for all other measurement) will be taken.
- Assessments not chosen for use in summary statistics by this algorithm will still appear in the associated listings.
- All applicable valid assessments, irrespective of proximity to the target study day, will be used when
  categorizing values across visits, such as 'maximum grade during the intervention phase' or 'at any
  time post-baseline', and for any algorithm that has specific rules for which observation to use (e.g.
  snapshot algorithm, LOCF or CVF identification).
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### **Treatment Start Date**

 Intervention Phase Treatment Start Date = Earliest date of CAB + RPV oral lead-in entered in the IP exposure eCRF form

#### **Nominal Month 14 Visit Date**

- For participants who received Month 14 injection, the nominal Month 14 visit date is defined by the Month 14 injection date.
- Otherwise, nominal Month 14 visit date is defined by the date of latest Month 14 assessment.
- For participants who continued into Extension Phase but missed the Month 14 visit, the nominal Month 14 visit date is defined by the last contact date prior to the date of the first nominal extension phase visit (i.e. Month 16, Month 18, etc.).

#### Study Day

- The Study Day of an event (e.g., lab assessment, vital sign, ECG, start date of AE or HIV associated condition) will be derived as the number of days between the date of the event and the Intervention Phase treatment start date as follows:
  - If date of event ≥ start date of study treatment, then
    - Study Day = Date of Event Intervention Phase Treatment Start Date +1
  - If date of event < start date of study treatment, then</li>
    - Study Day = Date of Event Intervention Phase Treatment Start Date
- Note that the start date of intervention phase study treatment is on Study Day 1 and the day before this is Study Day -1; i.e., there is no Study Day 0.

#### Long Term Follow-up Study Day

- Participants are considered to have entered LTFU if they have a post-treatment, non-bridging ART medication start date or a LTFU visit entered in the CRF.
- The Long-Term Follow Up (LTFU) Study Day of an event (e.g., lab assessment, start date of AE or HIV associated condition) will be derived as the number of days between the date of the event and the end of IP treatment [i.e. min(LTFU ART Start Date, max(Last IM Injection Date, Last Oral Bridging End Date)] as follows:
  - If the date of event falls in Long-term Follow up phase, then
    - LTFU Study Day = Date of event min(LTFU ART Start Date, max(Last IM Injection Date, Last Oral Bridging End Date)) + 1

#### **Study Treatment**

Refers to CAB+RPV oral lead-in, CAB + RPV oral bridging, SOC bridging, CAB LA + RPV LA

## Change from Baseline

- Post-Dose Visit Value Baseline
  - Unless otherwise specified, the baseline definitions specified in <u>Section 5.2</u> will be used for derivations for endpoints / parameters.

## 13.5.2. Study Population

#### **Demographics**

#### Age

- Age, in whole years, will be calculated with respect to the subject's Screening visit.
- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.
- Completely missing dates of birth will remain as missing, with no imputation applied. Consequently, the age of the subject will not be calculated and will remain missing.

#### **Body Mass Index**

Calculated as Weight (kg)/Height (m)<sup>2</sup>

#### **Hepatitis Status**

- Hepatitis C status will be determined using antibody and/or hepatitis C virus (HCV) RNA assessments performed during screening or during the conduct of the study.
- If both antibody and virus RNA assessments are available, then the latter will take precedence and
  positive/negative status will be based on whether HCV RNA is detectable (i.e., ≥ limit of
  quantification) or not.
- A participant will be considered positive for hepatitis B virus (HBV) if they have a positive surface antigen or detectable HBV DNA result. "HBV DNA DETECTED" in the lab comment takes precedence over HBV DNA test result for positive hepatitis B status; for example, if a participant has HBV DNA test result below level of detection and the lab comment shows that HBV DNA detected, this participant will be considered positive for hepatitis B. If HBV DNA result is available, it will be used to qualify hepatitis B status as positive or negative (positive if ≥ limit of quantification); otherwise Hepatitis B status will be determined using the surface antigen result.
- Hepatitis status at entry will be based on the assessments prior to/on the start of the study treatment.

#### Adherence to CAB/RPV Injection Schedule

 Timeliness of Injections relative to Date of Projected Dosing Visits are assessed by using "actual injection visit date - projected visit date from first injection". The injections of interest in adherence

#### **Demographics**

analysis are those after first injection at Month 1. (. Each injection visit is counted only once. Individual CAB and RPV injections administered at the same visit are not counted twice. "Extra" unscheduled injections are excluded from all derivations. For example, if during a scheduled visit a participant receives 1 ml of injection instead of 2 ml due to a dosing error, but this participant returns one week later for the remaining 1 ml injection, then the additional visit is excluded. If a participant receives an extra injection at an unscheduled visit by mistake, this visit will also be excluded.

- The categories of Timeliness of Injections relative to Date of Projected Dosing Visits are listed below:
  - < -14 days</li>
  - -14 to -8 days
  - -7 to 1
  - (
  - 1 to 7 days
  - 8 to 14 days
  - >14 days
  - Missed Injection without Oral Bridging (COVID-19 related)
  - Missed Injection without Oral Bridging (Non COVID-19 related)
  - Missed Injection with Oral Bridging (COVID-19 related)
  - Missed Injection with Oral Bridging (non COVID-19 related)
  - Missed Injection with subsequent SOC ART Initiation
- The following categories surrounding out of window (OOW) visits will also be calculated separately for participants at each visit.
  - Oral Bridging without a Missed Injection
  - OOW Injection with Oral Bridging (non-Covid-19 related)
  - OOW Injection with Oral Bridging (Covid-19 related)
  - OOW Injection without Oral Bridging (Covid-19 related)
- Injection visits are expected bi-monthly after an initial Month 1 Q4W injection from Month 2 until the nominal month of a participant's last injection visit during the phase(s) of interest. For example:
  - If a participant discontinues study treatment with last injection visit occurring at nominal visit Month 6, then injection visits are expected at Month 1, Month 2, Month 4, and Month 6.
- Expected injection visits will include all treatment visits (not LTFU) where an assessment was recorded regardless of whether the injection took place, including visits where treatment was discontinued.
- Missed injections with subsequent LTFU SOC ART Initiation are not counted in 'Missed Injection without Oral Bridging' categories. Missed injections will be slotted to this category if LTFU SOC ART is initiated within 30 days of the missed injection.
- Out of Window injections are determined based on criteria listed in protocol Section 4.3.3.
- Covid-19 relatedness is determined as follows:
  - As labelled in concomitant medication or exposure as Oral Bridging due to Covid-19
  - As indicated by Covid-19 protocol deviations that occur on the impacted visit date

# 13.5.3. **Efficacy**

#### **Efficacy**

## Snapshot

- The Snapshot algorithm is intended to be primarily a virologic assessment of the endpoint, and as such follows a "virology first" hierarchy.
- 'HIV-1 RNA < 50 c/mL' or 'HIV-1 RNA ≥ 50 c/mL' within an analysis window (see Table 2 and Table 3) is typically determined by the last available HIV-1 RNA measurement in that window while the participant is On-treatment in the Intervention Phase (as assigned based on Section 13.3).
- When no HIV-1 RNA data is available within a window, a participant cannot be assigned to the category of 'HIV-1 RNA < 50 c/mL'. Depending on the reason for lack of data, the participant will be classified as 'HIV-1 RNA ≥ 50 c/mL' or reported as 'No Virologic Data at Week X'; in the latter case, the algorithm further classifies the nature of the missing data. Typically, a participant withdrawn (i) due to AE or, (ii) for another reason yet was suppressed at the time, will be counted as 'No Virologic Data at Week X'. Should a participant withdraw for reasons other than AE and was not suppressed at the time, they will be categorized as 'HIV-1 RNA ≥ 50 c/mL'.</p>
- Full details of the algorithm, including the handling of special cases, are included in <a href="Appendix 8">Appendix 8</a>: Snapshot Algorithm Details.

#### Plasma HIV-1 RNA

HIV-1 RNA results may be provided as censored values, such as <40 or >9,999,999 c/mL. For the
purposes of summary statistics, such values will be replaced by the next value beyond the limit of
detection, e.g., 39 or 10,000,000 c/mL, respectively, for the given examples. Data listings will show
the censored values as provided.

# Confirmed Virologic Failure (CVF)

- For the purposes of clinical management in this study, CVF is defined as:
  - o Rebound as indicated by two consecutive plasma HIV-1 RNA levels ≥ 200 c/mL.
- The CVF definition is provided in the protocol Section 7.1.7
- Only plasma HIV-1 RNA values determined by the central laboratory will be used to assess virologic failure.

#### CDC Classification for HIV-1 Infection (2014)

 CDC HIV-1 Classification at Baseline is collected in eCRF and no derivation with be performed programmatically for analysis purposes. Please refer to study protocol for detail description of CDC HIV-1 Classification.

# 13.5.4. Safety

#### **Adverse Events**

# **DAIDS Grading**

- Clinical adverse events will be graded based on the Division of AIDS Table for Grading the Severity
  of Adult and Pediatric Adverse Events Version 2.1, March 2017, as specified in the protocol
  Appendix 10.2.
- If a grade value is expected per DAIDS but is missing in the eCRF, then the missing grade will be given an ordinal grade value of -1 for determining the maximum grade within and across preferred terms. For example:

#### **Adverse Events**

- if a participant has two separate instances of the same preferred term, one with grade 2 and one with missing grade, then the maximum grade for the preferred term will be set to grade 2.
- if a participant reports two different AE preferred terms overall, one with grade 1 and one with missing grade (where a DAIDS grade is expected), then the maximum grade across preferred terms (i.e. in the ANY EVENT row) will be set to grade 1.
- If a participant reports only one AE overall and this has a missing grade (where a DAIDS grade is expected), then this will be presented under a grade = missing category

#### **Days since First Dose (Days)**

AE Start Date – Intervention Phase Treatment Start Date + 1

#### Days since Last Dose (Days)

 AE Start Date – Date of Last Dose of Study Treatment (Oral CAB+RPV, SOC bridging, CAB/RPV IM Injection) prior to/on the Start Date of AE + 1

# **Days since Phase Start**

- For AEs in Intervention/Extension Phase:
  - AE Start Date Intervention Treatment Start Date + 1
- For AEs in Long-term Follow-up Phase:
  - AE Start Date LTFU ART Start Date

## **Duration (Days)**

• AE Resolution Date – AE Start Date + 1

#### **Drug-related**

- If relationship is marked 'YES' on Inform/eCRF
- Injection site reactions will be considered as drug-related if the relationship to study drug value is missing in the eCRF.

# **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value. If a character value starting with "<=x", then the numeric value will be x.
  - Example 1: 2 Significant Digits = '< x 'becomes x 0.01
  - Example 2: 1 Significant Digit = '> x' or '>=x' becomes x + 0.1
  - Example 3: 0 Significant Digits = '< x' becomes x 1

#### Lab Toxicities – DAIDS Grading

- Toxicities will be based on the Division of AIDS (DAIDS) grading system, Version 2.1, March 2017, as specified in the protocol of Appendix 10.2
- Toxicity grades provided by the central laboratory do not distinguish between abnormally high or low criteria, when both are relevant for a particular parameter.

#### **Other Safety Endpoints**

#### **Extent of Exposure**

 Exposure to CAB+RPV (oral lead-in or oral bridging) and CAB LA+RPV LA will be calculated from the IP eCRF pages.

#### For Intervention Phase:

- Exposure to CAB+RPV Oral Lead-in = IP (oral lead-in) stop date IP (oral lead-in) start date +1
- Exposure to CAB LA + RPV LA = Number of IP injection visits received during the Intervention Phase (up to but not including injections administered at Month 14)
- **Exposure to SOC oral bridging**: Duration of the SOC ART medication taken as oral bridging during the Intervention Phase. If the SOC oral bridging is taken in different periods during the Intervention Phase, the duration will be calculated by the sum of non-overlapped periods.
- Exposure to CAB+RPV Oral Bridging (COVID-19 Related): Duration of the CAB+RPV taken as
  oral bridging for reasons related to COVID-19 during the Intervention Phase. If COVID-19 related
  CAB+RPV oral bridging is taken in different periods during the Intervention Phase, the duration will
  be calculated by the sum of the non-overlapped periods.
- Exposure to CAB+RPV Oral Bridging (Non COVID-19 Related): Duration of the CAB+RPV taken
  as oral bridging for reasons not related to COVID-19 during the Intervention Phase. If non COVID-19
  related CAB+RPV oral bridging is taken in different periods during the Intervention Phase, the
  duration will be calculated by the sum of the non-overlapped periods.
- Overall Exposure to Study Treatment: min [Date of Latest Intervention Phase Visit up to and including Month 12, max (Date of Last Injection + 63, Date of Last Dose of Oral CAB+RPV, Date of Last Dose of SOC Oral Bridging)] min (Start Date for Oral lead-in CAB+RPV, Date of First CAB/RPV Injection) + 1
- Overall Exposure to CAB + RPV = Overall Exposure to Study Treatment Exposure to SOC Oral Bridging

#### For Intervention + Extension Phase:

- Exposure to CAB LA + RPV LA = Number of IP injection visits received during Intervention Phase and Extension Phase
- Exposure to SOC or CAB+RPV Oral Bridging during the Intervention and Extension Phase will be
  calculated similarly to that during the Intervention Phase except that the exposure includes both
  Intervention and Extension Phase.
- Overall Exposure to Study Treatment: min [LTFU ART start date, Commercial product Safety Follow-up Visit date, max (Date of Last Injection + 63, Date of Last Dose of Oral CAB+RPV, Date of Last Dose of SOC Oral Bridging)] min (Start Date for Oral lead-in CAB+RPV, Date of First Study Injection) + 1
- Overall Exposure to IP = Overall Exposure to Study Treatment Exposure to SOC Oral Bridging
- Duration of dosing in participant years will be calculated as the sum of participant duration of dosing in days (across all participants)/365.25

# 13.5.5. Virology

#### Genotype

## **Amino Acid Changes**

- A mutation is considered present whenever the encoded amino acid residue differs from the amino acid that would have been encoded by the wild-type (e.g., HXB2, NL43) comparator gene; e.g., Q148K.
- If the encoded amino acid is seen as a mixture of wild-type and mutant amino acid, e.g., Q148Q/K, the mutated amino acid is considered present at the codon of interest.
- If the encoded amino acid is seen as a mixture of two or more amino acids, which may or may not
  include wild type, e.g., Q184K/H or Q184K/H/Q, etc., for the purposes of calculating the number of
  mutated amino acids, only one mutation is considered to be present at the codon of interest.

## **Representation of Amino Acid Changes**

| Mutations | Amino Acid Change |
|---|---|
| T69S | Single mutation from amino acid 'T' (vendor reference) to 'S' (sample) at codon '69 |
| Q148H/K/R | Mixture of amino acid mutations 'H', 'K' and 'R' (sample) from amino acid 'Q (vendor reference) at codon '148' |
| _69_1T | First insertion of amino acid 'T' (sample) at codon '69' |
| _69_2S | Second insertion of amino acid 'S' (sample) at codon '69' |
| _69_3S/A | Third insertion of a mixture of amino acids 'S' and 'A' (sample) at codon '69' |
| L74L/- | Mixture of amino acid 'L' (sample) and a deletion at codon '74' |
| V75- | Single deletion of amino acid (sample) at codon '75' |

#### **Resistance Associated mutations**

Known INI mutations associated with the development of resistance to Integrase Strand Transfer Inhibitors:

| | H51Y, <b>T66</b> A/ <b>I</b> /K, L68V/I, L74I/M, <b>E92Q</b> /V/G, Q95K, T97A, <b>G118R</b> , <b>F121Y</b> , E138A/D/K/T, <b>G140</b> A/C/ <b>R</b> /S, <b>Y143</b> C/ <b>H</b> / <b>R</b> /K/S/G/A, P145S, Q146P, <b>S147G</b> , |
|---|---|
| Analysis | <b>Q148H/K/R</b> /N, V151/IL/A, S153F/Y, <b>N155H</b> /S/T, E157Q, G163R/K, G193E, S230R, <b>R263K</b> |

- Draft listing; may be modified in case of additional substantive data availability.
- Based on the IAS-USA list of mutations associated with resistance to Bictegravir, Cabotegravir, Dolutegravir, Elvitegravir, or Raltegravir (IAS-USA 2019 resistance mutations update volume 27 issue 3, 2019): T66A/I/K, L74M, E92Q/G, T97A, G118R, F121Y, E138A/K/T, G140A/C/R/S, Y143C/H/R, S147G, Q148H/K/R, S153F/Y, N155H, R263K) and observed mutations during in vitro passage of DTG or seen in a previous DTG study in INI-experienced subjects (study ING112574): H51Y, L74I, L68V/I, E92V, Q95K, E138D, Y143K/S/G/A, P145S, Q146P, V151I/L/A, N155S/T, E157Q, G163R/K, G193E, S230R.
- Major USA-IAS mutations associated with resistance to INSTI are bolded.
- Major resistance mutations to other classes (i.e., NRTI, NNRTI, PI) as defined by the International Antiviral Society-USA (IAS-USA). The most up to date IAS-USA guidelines available at the time of DBF will be used in the analysis [Wensing, 2019].

| Class | Mutations |
|---|---|
| NRTIs | M41L, A62V, K65R/E/N, D67N, 69 insert, K70E/R, L74V, V75I, F77L, Y115F, F116Y, |
| | Q151M, M184V/I, L210W, T215Y/F, K219Q/E |
| NNRTIs | L100I, K101E/P, K103N/S, V106A/M, V108I, E138/A/G/K/Q/R, V179L, |
| | Y181C/I/V, Y188C/L/H, G190S/A, H221Y, P225H, F227C, M230I/L |

| Genotype | |
|---|---|
| Pls | D30N, V32I, M46I/L, I47A/V, G48V, I50V/L, I54V/M/L, Q58E, T74P, L76V, |
| | V82A/T/F/L/S, N83D, I84V, N88S, L90M |
| Draft listing: may be modified in case of additional substantive data availability. | |

# 13.5.6. Other Assessments

# Study Visit Length

- Lead Time = Actual Start Time of Appointment Arrival Time
- Process Time = Actual End Time of Appointment Actual Start Time of Appointment
- Total Time = Actual End Time of Appointment Arrival Time

# 13.6. Appendix 6: Reporting Standards for Missing Data

# 13.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Withdrawn participants were not replaced in the study. |
| | <ul> <li>All available data from participants who were withdrawn from the study will be listed<br/>and all available planned data will be included in summary tables and figures, unless<br/>otherwise specified.</li> </ul> |
| | Withdrawal visits will be slotted according to <u>Appendix 2</u> : Assessment Windows (excluding PK data) |

# 13.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in participant listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 13.6.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Partial dates will be displayed as captured in participant listing displays.</li> <li>Where necessary, display macros may impute dates as temporary variables for sorting data in listings only. In addition, partial dates may be imputed for 'slotting' data to study phases or for specific analysis purposes as outlined below.</li> <li>Imputed partial dates will not be used to derive study day, time to onset or duration (e.g., time to onset or duration of adverse events), or elapsed time variables (e.g., time since diagnosis). In addition, imputed dates are not used for deriving the last contact date in overall survival analysis dataset.</li> </ul> |
| Adverse<br>Events | <ul> <li>Imputations in the adverse events dataset are used for slotting events to the appropriate study time periods and for sorting in data listings.</li> <li>Partial dates for AEs recorded in the CRF will be imputed using the following conventions:</li> </ul> |
| | Missing start day If study treatment start date is missing (i.e. participant did not start study treatment), then set start date = 1st of month. Else if study treatment start date is not missing: |

| Element | Reporting Detail | |
|---|---|---|
| | Missing start day and month | <ul> <li>If stop date contains a full date and stop date is earlier than study treatment start date, then set start date= 1st of month.</li> <li>Else set start date = study treatment start date.</li> <li>Else <ul> <li>For Non-ISR AEs: set start date = 1st of month</li> <li>For ISR AEs: if oral bridging taken during the month and year, set start date = min(last day of the month, day of AE stop date if available, day of study treatment discontinuation if occurring during the month and year); else set start date = 1st of month.</li> </ul> </li> <li>If study treatment start date is missing (i.e. participant did not start study treatment), then set start date = January 1.</li> <li>Else if study treatment start date is not missing: <ul> <li>If year of start date = year of study treatment start date, then</li> <li>If stop date contains a full date and stop date is earlier than study treatment start date, then set start date = January 1.</li> </ul> </li> </ul> |
| | Missing stop day Missing stop day | <ul> <li>Else set start date = study treatment start date.</li> <li>Else set start date = January 1.</li> <li>Last day of the month will be used.</li> <li>No Imputation</li> </ul> |
| | and month Completely missing start/end date | No imputation |
| | Completely missing start or end dates will remain missing, with no imputation applied. | |
| Non-ART<br>Medications<br>(including<br>Oral<br>Bridging<br>CAB + RPV) | Partial dates for a using the following | any concomitant medications recorded in the CRF will be imputed ng convention: |
| | Missing start day | <ul> <li>If study treatment start date is missing (i.e. participant did not start study treatment), then set start date = 1st of month.</li> <li>Else if study treatment start date is not missing: <ul> <li>If month and year of start date = month and year of study treatment start date, then</li> <li>If stop date contains a full date and stop date is earlier than study treatment start date, then set start date= 1st of month.</li> <li>Else set start date = study treatment start date.</li> <li>Else set start date = 1st of month.</li> </ul> </li> </ul> |
| | Missing start day and month | <ul> <li>If study treatment start date is missing (i.e. participant did not start study treatment), then set start date = January 1.</li> <li>Else if study treatment start date is not missing: <ul> <li>If year of start date = year of study treatment start date, then</li> <li>If stop date contains a full date and stop date is earlier than study treatment start date, then set start date = January 1.</li> <li>Else set start date = study treatment start date.</li> <li>Else set start date = January 1.</li> </ul> </li> </ul> |

| Element | Reporting Detail | |
|---|---|---|
| | Missing end day | A '28/29/30/31' will be used for the day (dependent on the month and year) |
| | Missing end day and month | A '31' will be used for the day and 'Dec' will be used for the month. |
| | Completely missing start/end date | No imputation |
| | The recorded par | tial date will be displayed in listings. |
| ART<br>Medications | Partial dates recorded in the eCRF will be imputed using the following convention: | |

# 13.6.2.2. Handling of Missing Data for Statistical Analysis

| Element | Reporting Detail |
|---|---|
| Snapshot | <ul> <li>In the Snapshot dataset, subjects without HIV – 1 RNA data in the assessment window for the visit of interest (due to missing data or discontinuation of IP prior to the visit window) do not belong to 'HIV-1</li> <li>50 c/mL (or 200 c/mL) The nature of this missing data will be further classified in Snapshot summaries as either 'HIV-1 RNA≥50' or 'No Virologic Data at Week X';</li> </ul> |
| | See <u>Appendix 8</u> : Snapshot Algorithm Details |
| | <ul> <li>Note: The primary snapshot analysis will not impute any missing<br/>data due to Covid-19 and will consider Covid-19 related missing<br/>data in accordance with all other missing data.</li> </ul> |

# 13.7. Appendix 7: Values of Potential Clinical Importance

Values of clinical importance will be summarized for hepatobiliary abnormalities. Abnormal laboratory value grades will be assigned as specified by protocol Section 10.2. Liver chemistry stopping criteria can be found in the protocol Section 10.3.1.

# 13.7.1. Hepatobiliary Abnormality Criteria

| Element | Reporting Detail |
|---|---|
| General | To include ALT, ALP, Bilirubin, & INR parameters |
| ALT >=3xULN and BIL >=2xULN | <ul> <li>If direct bilirubin is available (on the same date as Total Bilirubin), then direct bilirubin as a portion of total bilirubin must be &gt;=35% when total bilirubin is &gt;=2xULN, in order to satisfy the criteria.</li> <li>Bilirubin value is on or up to 28 days after ALT value.</li> </ul> |
| ALT >=3xULN and INR >1.5 | INR value is on or up to 28 days after ALT value. |
| ALT >=3xULN and BIL >=2xULN and ALP 2 (<1%) <2xULN | If direct bilirubin is available (on the same date as Total Bilirubin), then direct bilirubin as a portion of total bilirubin must be >=35% when total bilirubin is >=2xULN, in order to satisfy the criteria. |
| | <ul> <li>Bilirubin value is on or up to 28 days after ALT value.</li> <li>The ALP value must occur on or up to 28 days after the ALT value.</li> </ul> |
| Hepatocellular injury | Hepatocellular injury is defined as ((ALT/ALT ULN)/(ALP/ALP ULN)) >= 5 and ALT >= 3xULN. ALT and ALP values must occur on the same day. |
| Hepatocellular injury and BIL >=2xULN | <ul> <li>Hepatocellular injury is defined as ((ALT/ALT ULN)/(ALP/ALP ULN)) &gt;=5 and ALT &gt;=3xULN. ALT and ALP values must occur on the same day.</li> <li>If direct bilirubin is available (on the same date as Total Bilirubin), then direct bilirubin as a portion of total bilirubin must be &gt;=35% when total bilirubin is &gt;=2xULN, in order to satisfy the criteria.</li> <li>Bilirubin value is on or up to 28 days after ALT value.</li> </ul> |
| BIL >=2xULN | If direct bilirubin is available (on the same date as Total Bilirubin), then direct bilirubin as a portion of total bilirubin must be >=35% when total bilirubin is >=2xULN, in order to satisfy the criteria. |
| AST >3xULN and ALP <2xULN and BIL >=2xULN ALT>=X ULN and AST>=X ULN | <ul> <li>ALP and BIL values must occur on or up to 28 days after AST value.</li> <li>If direct bilirubin is available (on the same date as Total Bilirubin), then direct bilirubin as a portion of total bilirubin must be &gt;=35% when total bilirubin is &gt;=2xULN, in order to satisfy the criteria.</li> <li>AST and ALT values must occur on the same day</li> </ul> |

# 13.8. Appendix 8: Snapshot Algorithm Details

# **Detailed Algorithm Steps**

- Consider an analysis visit window for Month X as defined in Table 2.
- The HIV-1 RNA threshold of 50 will be analysed in this study
- The COVID-19 pandemic presents significant logistical challenges for many clinical sites around the world, with variable restrictions being placed on site resources and operations, and on an individual participants ability to attend clinic visits. The snapshot algorithm is modified to allow for the presentation of full scope of COVID-19 relatedness. The analysis window for 'Month 12' and HIV-1 RNA threshold of '50 c/mL' are used for the purpose of illustration. A participant's Snapshot response and reason at Month 12 are categorized as below.

```
o HIV-1 RNA < 50 c/mL
o HIV-1 RNA \geq 50 c/mL
  Data in window not below 50
    Non-COVID-19 related
         Discontinued for lack of efficacy
         Discontinued for other reason while not below 50
    COVID-19 related
         Discontinued for lack of efficacy
         Discontinued for other reason while not below 50
 No Virologic Data at Month 12 Window
    Non-COVID-19 related
         Discontinued study due to AE or death
         Discontinued study for other reasons
         On study but missing data in window
  COVID-19 related
         Discontinued study due to AE or death
         Discontinued study for other reasons
         On study but missing data in window
 Change in background therapy*
```

- \* Note: Use of CAB + RPV oral bridging and SOC oral bridging medication, where the latter is due to unavailability of CAB/RPV IM injections or oral CAB+RPV during the pandemic, will not be considered a "Change in background therapy" in the Snapshot algorithm. All other permanent changes in ART are not permitted in this protocol.
- The steps in determining response and reasons are indicated in the table below, in the order stated.
- Background therapy is not given to participants while on study. The "change in background therapy" in detailed steps below refers to the "change in ART" in this study.

## **Detailed steps**

 Please note that the following scenarios will NOT be penalized in the Snapshot algorithm Oral bridging (CAB+RPV or SOC, where SOC oral bridging medication is permitted during COVID-19 pandemic due to the unavailability of the CAB/RPV IM injections and oral CAB+RPV)

| Detailed Algorithm Steps | | |
|---|---|---|
| Condition ('Month 12' indicates Month 12 window) | Response | Reasons |
| If non-permitted change in background therapy prior to Month 12 | HIV-1 RNA ≥ 50 | Change in background therapy |
| If non-permitted change in background therapy during Month 12 | | |
| <ul> <li>Last on-treatment VL during Month 12 prior to/on<br/>the date of change ≥ 50 c/mL</li> </ul> | HIV-1 RNA ≥ 50 | Data in window not below 50 |
| <ul> <li>Last on-treatment VL during Month 12 prior to/on<br/>the date of change &lt; 50 c/mL</li> </ul> | HIV-1 RNA < 50 | |
| No VL during Month 12 prior to/on the date of change | HIV-1 RNA ≥ 50 | Change in background therapy |
| 3. If none of the above conditions met | | |
| 3.1. On-treatment VL available during Month 12 | | |
| <ul> <li>Last on-treatment VL during Month 12 ≥ 50<br/>c/mL</li> </ul> | HIV-1 RNA ≥ 50 | Data in window not below 50 |
| Last on-treatment VL during Month 12 < 50 c/mL | HIV-1 RNA < 50 | |
| 3.2. No on-treatment VL during Month 12 | | |
| <ul> <li>3.2.1. If participants are still on study, i.e. a participant has not permanently discontinued the study treatment yet, or if a participant permanently discontinued the study treatment and the upper bound of analysis snapshot window is prior to the following date: <ul> <li>Min[max(Date of last injection + 35, Date of Last Dose of Oral Study Treatment (CAB+RPV, SOC Bridging) + 1), LTFU ART Start Date]</li> </ul> </li> </ul> | | |
| 3.2.1.1. If no on-treatment VL during Month<br>12 is not due to COVID-19 | No virologic<br>data at Month<br>12 Window | On study but missing data in window (Non-COVID-19 related) |
| 3.2.1.2. If no on-treatment VL during Month 12 is due to COVID-19 | No virologic<br>data at Month<br>12 Window | On study but missing data in window (COVID-19 related) |
| 3.2.2. If participants withdraw before/during Month 12 due to | | |
| 3.2.2.1. Non-COVID-19 related safety reasons (e.g. AE/death, liver chemistry stopping criteria, renal toxicity withdrawal criteria, QTc withdrawal criteria etc., as recorded in eCRF Conclusion form) | No virologic<br>data at Month<br>12 Window | Disc due to AE/death<br>(Non-COVID-19<br>related) |

| Detailed Algorithm Steps | | |
|---|---|---|
| 3.2.2.2. COVID-19 related safety reasons (e.g. AE/death, liver chemistry stopping criteria, renal toxicity withdrawal criteria, QTc withdrawal criteria etc., as recorded in eCRF Conclusion form) | No virologic<br>data at Month<br>12 Window | Disc due to AE/death<br>(COVID-19 related) |
| 3.2.2.3. Non-safety and Non-COVID-19 related reasons (e.g. Lack of efficacy, protocol deviation, withdrew consent, loss to follow-up, study closed/terminated, investigator discretion etc., as recorded in eCRF Treatment Discontinuation Form) | | |
| <ul> <li>Last on-treatment VL &lt;50 c/mL</li> <li>OR no on-treatment VL</li> <li>available during study</li> <li>Last on-treatment VL ≥ 50</li> <li>c/mL AND withdrawal due to</li> </ul> | No virologic Data at Month 12 Window HIV-1 RNA ≥ 50 | Disc for other<br>reasons (Non-<br>COVID-19 related)<br>Disc. for lack of<br>efficacy (Non- |
| Lack of efficacy o Last on-treatment VL ≥ 50 c/mL AND withdrawal due to all other non-safety related reasons | HIV-1 RNA ≥ 50 | Disc. for other reason while not below 50 (Non-COVID-19 related) |
| 3.2.2.4. Non-safety and COVID-19 related reasons (e.g. protocol deviation, withdrew consent, loss to follow-up, study closed/terminated, investigator discretion etc., as recorded in eCRF Conclusion Form) | | |
| <ul> <li>Last on-treatment VL &lt;50 c/mL</li> <li>OR no on-treatment VL</li> <li>available during study</li> </ul> | No virologic Data at Month 12 Window | Disc for other<br>reasons (COVID-19<br>related) |
| <ul> <li>Last on-treatment VL ≥ 50</li> <li>c/mL AND withdrawal due to</li> <li>Lack of efficacy</li> </ul> | HIV-1 RNA ≥ 50 | Disc. for lack of efficacy (COVID-19 related) |
| <ul> <li>Last on-treatment VL ≥ 50</li> <li>c/mL AND withdrawal due to all other non-safety related reasons</li> </ul> | HIV-1 RNA ≥ 50 | Disc. for other<br>reason while not<br>below 50 (COVID-19<br>related) |

a. Excluding permitted change in background therapy where change or decision to change is made prior to/on the first on-treatment viral result

# **Examples from FDA guidance**

# Data in Window

Virologic outcome should be determined by the last available measurement while the patient is on treatment and continued on trial within the time window:

 HIV-1 RNA = 580 c/mL at Day 336, HIV-1 RNA below 50 c/mL on Day 350. This should be categorized as HIV-1 RNA below 50 c/mL.

#### No Data in Window

## **Detailed Algorithm Steps**

## Discontinued study due to Adverse Event or Death:

- Any patient who discontinues because of an AE or death before the window should be classified as
   Discontinued due to AE or Death (as appropriate), regardless of the HIV-1 RNA result, even if the HIV-1
   RNA is below 50 c/mL at the time of discontinuation.
- However, if a patient has an HIV-1 RNA value in the time window and also discontinues in the time window, the viral load data should be used to classify the patient's response. This is the Virology First hierarchy:
  - a. HIV-1 RNA below 50 c/mL at Day 336 and discontinues because of AE or even dies on Day 360 this person is categorized as having HIV-1 RNA below 50 c/mL.
  - b. HIV-1 RNA is 552 c/mL on Day 336 and the patient discontinues on Day 360, the patient is categorized as having HIV-1 RNA ≥ 50 c/mL.

#### Discontinued for Other Reasons:

- Only patients who have achieved virologic suppression can be counted as Discontinued for Other Reasons.
- If a patient discontinues the study before the time window because of lack of efficacy, then the patient should be included in the HIV-1 RNA ≥ 50 row and not in the Discontinued for Other Reasons row.
- If a patient discontinues because *participant withdrew consent* and his or her HIV-1 RNA result at the time of discontinuation was equal to or above 50 c/mL, then he or she should be categorized as HIV-1 RNA ≥ 50 and NOT as Discontinued for Other Reasons.
- If a patient discontinued because of *Lost to Follow-Up* and the last HIV-1 RNA result was 49 c/mL, then the patient can be categorized as Discontinued for Other Reasons.
- If patients changed background treatment *not permitted by protocol* they should be considered an efficacy failure and captured in the HIV-1 RNA ≥ 50 c/mL row.

# On study but missing data in window:

- If there are no data during Days 294 to 377, but there is an HIV-1 RNA below 50 c/mL on Day 380, this patient should be considered *On Study but Missing Data in Window.*
- If there are no data during Days 294 to 377, but there is an HIV-1 RNA equal to or above 50 c/mL on Day 280, this patient also should be classified as On Study but Missing Data in Window.

# 13.9. Appendix 9: Identification of Adverse Events of Special Interest

SMQ and PT codes based on MedDRA dictionary version 23.1 for the Month 12 analysis.

# 13.9.1. Hepatic Safety Profile

Medical concept of hepatic failure and hepatitis. Sub- SMQs (1) 'Hepatic failure, fibrosis and cirrhosis and other liver damage-related conditions' and (2) 'Hepatitis, non-infectious', both of parent SMQ 'Hepatic Disorders (SMQ code 20000005)'; only narrow terms selected from sub-SMQs. Some preferred terms, e.g. PT 'hepatitis fulminant' are duplicated.

| SMQ: 'Hepatic Disorders'; SMQ Code: 20000005 | |
|---|---|
| Sub-SMQ: 'Hepatic failure, fibrosis and cirrhosis and other liver damage-related | |
| conditions' | |
| Category: A | |
| Scope: Narrow | |
| Preferred Term | PT Code |
| Acquired hepatocerebral degeneration | 10080860 |
| Acute hepatic failure | 10000804 |
| Acute on chronic liver failure | 10077305 |
| Acute yellow liver atrophy | 10070815 |
| Ascites | 10003445 |
| Asterixis | 10003547 |
| Bacterascites | 10068547 |
| Biliary cirrhosis | 10004659 |
| Biliary fibrosis | 10004664 |
| Cardiohepatic syndrome | 10082480 |
| Cholestatic liver injury | 10067969 |
| Chronic hepatic failure | 10057573 |
| Coma hepatic | 10010075 |
| Cryptogenic cirrhosis | 10063075 |
| Diabetic hepatopathy | 10071265 |
| Drug-induced liver injury | 10072268 |

| SMQ: 'Hepatic Disorders'; SMQ Code: 20000005 | |
|----------------------------------------------------|----------|
| Duodenal varices | 10051010 |
| Gallbladder varices | 10072319 |
| Gastric variceal injection | 10076237 |
| Gastric variceal ligation | 10076238 |
| Gastric varices | 10051012 |
| Gastric varices haemorrhage | 10057572 |
| Gastrooesophageal variceal haemorrhage prophylaxis | 10066597 |
| Flood Syndrome | 10084797 |
| Hepatectomy | 10061997 |
| Hepatic atrophy | 10019637 |
| Hepatic calcification | 10065274 |
| Hepatic cirrhosis | 10019641 |
| Hepatic encephalopathy | 10019660 |
| Hepatic encephalopathy prophylaxis | 10066599 |
| Hepatic failure | 10019663 |
| Hepatic fibrosis | 10019668 |
| Hepatic hydrothorax | 10067365 |
| Hepatic infiltration eosinophilic | 10064668 |
| Hepatic lesion | 10061998 |
| Hepatic necrosis | 10019692 |
| Hepatic steato-fibrosis | 10077215 |
| Hepatic steatosis | 10019708 |
| Hepatitis fulminant | 10019772 |
| Hepatobiliary disease | 10062000 |
| Hepatocellular foamy cell syndrome | 10053244 |
| Hepatocellular injury | 10019837 |
| Hepatopulmonary syndrome | 10052274 |
| Hepatorenal failure | 10019845 |

| Hepatotoxicity 1 Immune-mediated cholangitis 1 Immune-mediated hepatic disorder 1 Intestinal varices 1 Intestinal varices haemorrhage 1 Liver dialysis 1 Liver disorder 1 | 10019846<br>10019851<br>10083406<br>10083521<br>10071502<br>10078058<br>10076640<br>10024670<br>10067125 |
|---|---|
| Immune-mediated cholangitis1Immune-mediated hepatic disorder1Intestinal varices1Intestinal varices haemorrhage1Liver dialysis1Liver disorder1 | 10083406<br>10083521<br>10071502<br>10078058<br>10076640<br>10024670<br>10067125 |
| Immune-mediated hepatic disorder 1 Intestinal varices 1 Intestinal varices haemorrhage 1 Liver dialysis 1 Liver disorder 1 | 10083521<br>10071502<br>10078058<br>10076640<br>10024670<br>10067125 |
| Intestinal varices 1 Intestinal varices haemorrhage 1 Liver dialysis 1 Liver disorder 1 | 10071502<br>10078058<br>10076640<br>10024670<br>10067125 |
| Intestinal varices haemorrhage 1 Liver dialysis 1 Liver disorder 1 | 10078058<br>10076640<br>10024670<br>10067125 |
| Liver dialysis 1 Liver disorder 1 | 10076640<br>10024670<br>10067125 |
| Liver disorder 1 | 10024670<br>10067125 |
| | 10067125 |
| Liver injury 1 | |
| Liver operation 1 | 10062040 |
| Liver transplant 1 | 10024714 |
| Lupoid hepatic cirrhosis 1 | 10025129 |
| Minimal hepatic encephalopathy | 10076204 |
| Mixed liver injury 1 | 10066758 |
| Nodular regenerative hyperplasia 1 | 10051081 |
| Nonalcoholic fatty liver disease | 10082249 |
| Non-alcoholic steatohepatitis 1 | 10053219 |
| Non-cirrhotic portal hypertension | 10077259 |
| Oedema due to hepatic disease | 10049631 |
| Oesophageal varices haemorrhage | 10030210 |
| Peripancreatic varices 1 | 10073215 |
| Portal fibrosis 1 | 10074726 |
| Portal hypertension 1 | 10036200 |
| Portal hypertensive colopathy 1 | 10079446 |
| Portal hypertensive enteropathy 1 | 10068923 |
| Portal hypertensive gastropathy 1 | 10050897 |
| Portal vein cavernous transformation 1 | 10073979 |
| Portal vein dilatation 1 | 10073209 |

| SMQ: 'Hepatic Disorders'; SMQ Code: 20000005 | |
|---|---|
| Portopulmonary hypertension | 10067281 |
| Primary biliary cholangitis | 10080429 |
| Regenerative siderotic hepatic nodule | 10080679 |
| Renal and liver transplant | 10052279 |
| Retrograde portal vein flow | 10067338 |
| Reye's syndrome | 10039012 |
| Reynold's syndrome | 10070953 |
| Splenic varices | 10067823 |
| Splenic varices haemorrhage | 10068662 |
| Steatohepatitis | 10076331 |
| Subacute hepatic failure | 10056956 |
| Sugiura procedure | 10083010 |
| Varices oesophageal | 10056091 |
| Varicose veins of abdominal wall | 10072284 |
| White nipple sign | 10078438 |
| SMQ: 'Hepatic Disorders'; SMQ Code: 20000005 Sub-SMQ: 'Hepatitis, non-infectious' Category: A Scope: Narrow | |
| Preferred Term | PT Code |
| Acute graft versus host disease in liver | 10066263 |
| Allergic hepatitis | 10071198 |
| Alloimmune hepatitis | 10080576 |
| Autoimmune hepatitis | 10003827 |
| Chronic graft versus host disease in liver | 10072160 |
| Chronic hepatitis | 10008909 |
| Graft versus host disease in liver | 10064676 |
| Hepatitis | 10019717 |
| Hepatitis acute | 10019727 |
| Hepatitis cholestatic | 10019754 |

| SMQ: 'Hepatic Disorders'; SMQ Code: 20000005 | |
|----------------------------------------------|----------|
| Hepatitis chronic active | 10019755 |
| Hepatitis chronic persistent | 10019759 |
| Hepatitis fulminant | 10019772 |
| Hepatitis toxic | 10019795 |
| Immune-mediated hepatitis | 10078962 |
| Ischaemic hepatitis | 10023025 |
| Lupus hepatitis | 10067737 |
| Non-alcoholic steatohepatitis | 10053219 |
| Radiation hepatitis | 10051015 |
| Steatohepatitis | 10076331 |

# 13.9.2. Hyperglycaemia

Medical concept of Hyperglycaemia/new onset diabetes mellitus - SMQs (1) 'Hyperglycaemia/new onset diabetes mellitus (SMQ) Narrow SMQ code 20000041.

| SMQ: 'Hyperglycaemia/new onset diabetes mellitus '; SMQ Code: 20000041 | |
|---|---|
| Sub-SMQ: 'Hepatic failure, fibrosis and cirrhosis and other liver damage-related | |
| Category: A | |
| Scope: Narrow | |
| Preferred Term | PT Code |
| Acquired lipoatrophic diabetes | 10073667 |
| Blood 1,5-anhydroglucitol decreased | 10065367 |
| Blood glucose increased | 10005557 |
| Diabetes complicating pregnancy | 10012596 |
| Diabetes mellitus | 10012601 |
| Diabetes mellitus inadequate control | 10012607 |
| Diabetes with hyperosmolarity | 10012631 |
| Diabetic arteritis | 10077357 |
| Diabetic coma | 10012650 |
| Diabetic coronary microangiopathy | 10080788 |
| Diabetic hepatopathy | 10071265 |

| Diabetic hyperglycaemic coma Diabetic hyperosmolar coma Diabetic ketoacidosis Diabetic ketoacidosis Diabetic ketoacidotic hyperglycaemic coma Diabetic ketosis Diabetic ketosis Diabetic ketosis Diabetic metabolic decompensation Diabetic wound Diabetic ketoacidosis Diabetic ketoac | SMQ: 'Hyperglycaemia/new onset diabetes mellitus '; SMQ Code: 20000041 | |
|---|---|---|
| Diabetic ketoacidosis Diabetic ketoacidotic hyperglycaemic coma Diabetic ketoacidotic hyperglycaemic coma Diabetic ketosis Diabetic metabolic decompensation Diabetic wound Diabetic wound Diabetic wound Diabetic ketoacidosis Euglycaemic diabetic ketoacidosis Fructosamine increased Diapetic wound Diapetic w | Diabetic hyperglycaemic coma | 10012668 |
| Diabetic ketoacidotic hyperglycaemic coma Diabetic ketosis 10012673 Diabetic metabolic decompensation Diabetic wound Diabetic wound Diabetic ketoacidosis Euglycaemic diabetic ketoacidosis Fructosamine increased 10017395 Fulminant type I diabetes mellitus Gestational diabetes Glucose tolerance impaired Glucose tolerance impaired Glucose tolerance impaired in pregnancy Glucose urine present Glycated albumin increased Glycosuria Glycosuria Glycosuria during pregnancy Glycosylated haemoglobin abnormal Glycosylated haemoglobin increased Hyperglycaemia Hyperglycaemic hyperosmolar nonketotic syndrome Hyperglycaemic unconsciousness Inountable Insulin resistance Inountable 10022489 Insulin resistant diabetes 10022491 Insulin-requiring type 2 diabetes mellitus 10074309 | Diabetic hyperosmolar coma | 10012669 |
| Diabetic ketosis Diabetic metabolic decompensation Diabetic wound Diabetic wound Diabetic wound Diabetic wound Diabetic wound Diabetic ketoacidosis Euglycaemic diabetic ketoacidosis Fructosamine increased Fructosamine increased Fructosamine increased Diabetic wound Diabete Diabetes wound Diabete Diabetes Diabetes wound Diabete Diabetes wound Diabete Diabetes Wound Diab | Diabetic ketoacidosis | 10012671 |
| Diabetic metabolic decompensation Diabetic wound Diabetes Diabetes wellitus Diabetes wound | Diabetic ketoacidotic hyperglycaemic coma | 10012672 |
| Diabetic wound 10081558 Euglycaemic diabetic ketoacidosis 10080061 Fructosamine increased 10017395 Fulminant type 1 diabetes mellitus 10072628 Gestational diabetes 10018209 Glucose tolerance impaired 10018429 Glucose tolerance impaired 10018430 Glucose urine present 10018478 Glycated albumin increased 10082836 Glycosuria 10018473 Glycosuria during pregnancy 10018475 Glycosylated haemoglobin abnormal 10018481 Glycosylated haemoglobin increased 10082836 Hyperglycaemia 10020635 Hyperglycaemic hyperosmolar nonketotic syndrome 10063554 Hyperglycaemic seizure 10071394 Hyperglycaemic unconsciousness 10071286 Impaired fasting glucose 10022489 Insulin resistant diabetes 10022491 Insulin-requiring type 2 diabetes mellitus 10053247 | Diabetic ketosis | 10012673 |
| Euglycaemic diabetic ketoacidosis Fructosamine increased 10017395 Fulminant type 1 diabetes mellitus Gestational diabetes 10018209 Glucose tolerance impaired 10018429 Glucose tolerance impaired in pregnancy 10018430 Glucose urine present 10018478 Glycated albumin increased 10082836 Glycosuria 10018473 Glycosuria during pregnancy 10018475 Glycosylated haemoglobin abnormal 10018481 Glycosylated haemoglobin increased 10020635 Hyperglycaemic hyperosmolar nonketotic syndrome 10071394 Hyperglycaemic unconsciousness 10071286 Impaired fasting glucose 10022489 Insulin resistance 10023247 | Diabetic metabolic decompensation | 10074309 |
| Fructosamine increased Fulminant type 1 diabetes mellitus Gestational diabetes Glucose tolerance impaired Glucose tolerance impaired in pregnancy Glucose urine present Glycated albumin increased Glycosuria Glycosuria Glycosuria during pregnancy Glycosylated haemoglobin abnormal Glycosylated haemoglobin increased Hyperglycaemia Hyperglycaemia Hyperglycaemic seizure Hyperglycaemic seizure Ino071286 Impaired fasting glucose Insulin resistance 10022491 Insulin-requiring type 2 diabetes mellitus 10018209 10018429 10018430 10018478 10018478 10018473 10018473 10018475 10018484 10018484 10018484 10022491 Insulin-requiring type 2 diabetes mellitus | Diabetic wound | 10081558 |
| Fulminant type 1 diabetes mellitus Gestational diabetes Glucose tolerance impaired Glucose tolerance impaired in pregnancy Glucose urine present Glycated albumin increased Glycosuria Glycosuria Glycosuria during pregnancy Glycosylated haemoglobin abnormal Glycosylated haemoglobin increased Hyperglycaemia Hyperglycaemic hyperosmolar nonketotic syndrome Hyperglycaemic seizure Hyperglycaemic unconsciousness Inou71286 Impaired fasting glucose Insulin resistance 10022491 Insulin-requiring type 2 diabetes mellitus | Euglycaemic diabetic ketoacidosis | 10080061 |
| Gestational diabetes 10018209 Glucose tolerance impaired 10018429 Glucose tolerance impaired 10018430 Glucose urine present 10018478 Glycated albumin increased 10082836 Glycosuria 10018473 Glycosuria during pregnancy 10018475 Glycosylated haemoglobin abnormal 10018481 Glycosylated haemoglobin increased 10018484 Hyperglycaemia 10020635 Hyperglycaemic hyperosmolar nonketotic syndrome 10063554 Hyperglycaemic seizure 10071394 Hyperglycaemic unconsciousness 10071286 Impaired fasting glucose 10022489 Insulin resistance 10022491 Insulin-requiring type 2 diabetes mellitus 10053247 | Fructosamine increased | 10017395 |
| Glucose tolerance impaired 10018429 Glucose tolerance impaired in pregnancy 10018430 Glucose urine present 10018478 Glycated albumin increased 10082836 Glycosuria 10018473 Glycosuria during pregnancy 10018475 Glycosylated haemoglobin abnormal 10018481 Glycosylated haemoglobin increased 10018484 Hyperglycaemia 10020635 Hyperglycaemic hyperosmolar nonketotic syndrome 10063554 Hyperglycaemic seizure 10071394 Hyperglycaemic unconsciousness 10071286 Impaired fasting glucose 10056997 Insulin resistance 10022489 Insulin resistant diabetes 10022491 Insulin-requiring type 2 diabetes mellitus 10053247 | Fulminant type 1 diabetes mellitus | 10072628 |
| Glucose tolerance impaired in pregnancy Glucose urine present Glycated albumin increased Glycosuria Glycosuria Glycosuria during pregnancy Glycosylated haemoglobin abnormal Glycosylated haemoglobin increased Hyperglycaemia Hyperglycaemic hyperosmolar nonketotic syndrome Hyperglycaemic seizure Hyperglycaemic unconsciousness Inou71286 Impaired fasting glucose Insulin resistance Inou22489 Insulin-requiring type 2 diabetes mellitus | Gestational diabetes | 10018209 |
| Glucose urine present 10018478 Glycated albumin increased 10082836 Glycosuria 10018473 Glycosuria during pregnancy 10018475 Glycosylated haemoglobin abnormal 10018481 Glycosylated haemoglobin increased 10018484 Hyperglycaemia 10020635 Hyperglycaemic hyperosmolar nonketotic syndrome 10063554 Hyperglycaemic seizure 10071394 Hyperglycaemic unconsciousness 10071286 Impaired fasting glucose 10022489 Insulin resistant diabetes 10022491 Insulin-requiring type 2 diabetes mellitus 10053247 | Glucose tolerance impaired | 10018429 |
| Glycosuria 10082836 Glycosuria 10018473 Glycosuria during pregnancy 10018475 Glycosylated haemoglobin abnormal 10018481 Glycosylated haemoglobin increased 10018484 Hyperglycaemia 10020635 Hyperglycaemic hyperosmolar nonketotic syndrome 10063554 Hyperglycaemic seizure 10071394 Hyperglycaemic unconsciousness 10071286 Impaired fasting glucose 10056997 Insulin resistance 10022489 Insulin-requiring type 2 diabetes mellitus 10053247 | Glucose tolerance impaired in pregnancy | 10018430 |
| Glycosuria 10018473 Glycosuria during pregnancy 10018475 Glycosylated haemoglobin abnormal 10018481 Glycosylated haemoglobin increased 10018484 Hyperglycaemia 10020635 Hyperglycaemic hyperosmolar nonketotic syndrome 10063554 Hyperglycaemic seizure 10071394 Hyperglycaemic unconsciousness 10071286 Impaired fasting glucose 10056997 Insulin resistance 10022489 Insulin-requiring type 2 diabetes mellitus 10053247 | Glucose urine present | 10018478 |
| Glycosuria during pregnancy Glycosylated haemoglobin abnormal Glycosylated haemoglobin increased Hyperglycaemia Hyperglycaemic hyperosmolar nonketotic syndrome 10063554 Hyperglycaemic seizure 10071394 Hyperglycaemic unconsciousness 10071286 Impaired fasting glucose 10022489 Insulin resistant diabetes 10023247 Insulin-requiring type 2 diabetes mellitus | Glycated albumin increased | 10082836 |
| Glycosylated haemoglobin abnormal Glycosylated haemoglobin increased Hyperglycaemia Hyperglycaemic hyperosmolar nonketotic syndrome 10063554 Hyperglycaemic seizure 10071394 Hyperglycaemic unconsciousness 10071286 Impaired fasting glucose 10056997 Insulin resistance 10022489 Insulin resistant diabetes 10053247 | Glycosuria | 10018473 |
| Glycosylated haemoglobin increased 10018484 Hyperglycaemia 10020635 Hyperglycaemic hyperosmolar nonketotic syndrome 10063554 Hyperglycaemic seizure 10071394 Hyperglycaemic unconsciousness 10071286 Impaired fasting glucose 10056997 Insulin resistance 10022489 Insulin resistant diabetes 10022491 Insulin-requiring type 2 diabetes mellitus 10053247 | Glycosuria during pregnancy | 10018475 |
| Hyperglycaemia 10020635 Hyperglycaemic hyperosmolar nonketotic syndrome 10063554 Hyperglycaemic seizure 10071394 Hyperglycaemic unconsciousness 10071286 Impaired fasting glucose 10056997 Insulin resistance 10022489 Insulin resistant diabetes 10022491 Insulin-requiring type 2 diabetes mellitus 10053247 | Glycosylated haemoglobin abnormal | 10018481 |
| Hyperglycaemic hyperosmolar nonketotic syndrome 10063554 Hyperglycaemic seizure 10071394 Hyperglycaemic unconsciousness 10071286 Impaired fasting glucose 10056997 Insulin resistance 10022489 Insulin resistant diabetes 10022491 Insulin-requiring type 2 diabetes mellitus | Glycosylated haemoglobin increased | 10018484 |
| Hyperglycaemic seizure 10071394 Hyperglycaemic unconsciousness 10071286 Impaired fasting glucose 10056997 Insulin resistance 10022489 Insulin resistant diabetes 10022491 Insulin-requiring type 2 diabetes mellitus 10053247 | Hyperglycaemia | 10020635 |
| Hyperglycaemic unconsciousness 10071286 Impaired fasting glucose 10056997 Insulin resistance 10022489 Insulin resistant diabetes 10022491 Insulin-requiring type 2 diabetes mellitus 10053247 | Hyperglycaemic hyperosmolar nonketotic syndrome | 10063554 |
| Impaired fasting glucose10056997Insulin resistance10022489Insulin resistant diabetes10022491Insulin-requiring type 2 diabetes mellitus10053247 | Hyperglycaemic seizure | 10071394 |
| Insulin resistance 10022489 Insulin resistant diabetes 10022491 Insulin-requiring type 2 diabetes mellitus 10053247 | Hyperglycaemic unconsciousness | 10071286 |
| Insulin resistant diabetes 10022491 Insulin-requiring type 2 diabetes mellitus 10053247 | Impaired fasting glucose | 10056997 |
| Insulin-requiring type 2 diabetes mellitus 10053247 | Insulin resistance | 10022489 |
| | Insulin resistant diabetes | 10022491 |
| Ketoacidosis 10023379 | Insulin-requiring type 2 diabetes mellitus | 10053247 |
| | Ketoacidosis | 10023379 |

| SMQ: 'Hyperglycaemia/new onset diabetes mellitus '; SMQ Code: 20000041 | |
|---|---|
| Ketonuria | 10023388 |
| Ketosis | 10023391 |
| Ketosis-prone diabetes mellitus | 10023392 |
| Latent autoimmune diabetes in adults | 10066389 |
| Monogenic diabetes | 10075980 |
| Neonatal diabetes mellitus | 10028933 |
| New onset diabetes after transplantation | 10082630 |
| Pancreatogenous diabetes | 10033660 |
| Steroid diabetes | 10081755 |
| Type 1 diabetes mellitus | 10067584 |
| Type 2 diabetes mellitus | 10067585 |
| Type 3 diabetes mellitus | 10072659 |
| Urine ketone body present | 10057597 |

# 13.9.3. Hypersensitivity Reactions

Notes: Medical concept of hypersensitivity reactions/DRESS. Only narrow terms selected from Category A of SMQ 'Drug reaction with eosinophilia and systemic symptoms syndrome'. Algorithmic approach for this SMQ not used due to complexity in applying and poor specificity of remaining categories. Category A selected as PTs because more specific for concept (only narrow terms) and a pre-requisite for any combination in algorithmic search. Overlap of some preferred terms with SMQ 'Severe Cutaneous Adverse Reactions'. Plus additional preferred terms selected from HGLT 'Allergic conditions' under SOC 'Immune system disorders'.

| SMQ: Drug reaction with eosinophilia and systemic symptoms syndrome SMQ Code: 20000225 Category: A Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Drug reaction with eosinophilia and systemic symptoms | 10073508 |
| Pseudolymphoma | 10037127 |
| Additional preferred terms selected from HLGT 'Allergic conditions' under SOC 'Immune system disorders'; HLGT code 10001708 | |
| Preferred Term | PT Code |
| SMQ: Drug reaction with eosinophilia and systemic symptoms syndrome | |
|---|---|
| SMQ Code: 20000225 | |
| Category: A | |
| Scope: Narrow | |
| Drug hypersensitivity | 10013700 |
| Hypersensitivity | 10020751 |
| Type IV Hypersensitivity reaction | 10053613 |
| Eosinophillia | 10014950 |
| Eye swelling | 10015967 |
| Eyelid oedema | 10015993 |
| Lip swelling | 10024570 |
| Angioedema | 10002424 |
| Circumoral oedema | 10052250 |
| Face oedema | 10016029 |
| Idiopathic angioedema | 10073257 |
| Lip oedema | 10024558 |
| Mouth swelling | 10075203 |
| Oedema mouth | 10030110 |
| Periorbital oedema | 10034545 |
| Swelling face | 10042682 |
| Periorbital swelling | 10056647 |
| Swelling of eyelid | 10042690 |
| Granulomatous T-cell pseudolymphoma | 10084214 |

# 13.9.4. Rash including severe cutaneous adverse reactions

Medical concept of rash including severe cutaneous adverse reactions. Only narrow terms from SMQ 'Severe cutaneous adverse reactions' selected. Plus several additional preferred terms selected from HLTs 'Rashes, eruptions and exanthems NEC', 'Pruritus NEC', 'Pustular conditions', 'Dermatitis ascribed to specific agent' all under SOC 'Skin and subcutaneous tissue disorders'.

| SMQ: Severe Cutaneous Adverse Reactions SMQ Code: 20000020 Category: A Scope: Narrow | |
|---|---|
| SMQ | PT Code |
| Acute generalised exanthematous pustulosis | 10048799 |
| Bullous haemorrhagic dermatosis | 10083809 |
| Cutaneous vasculitis | 10011686 |
| Dermatitis bullous | 10012441 |
| Dermatitis exfoliative | 10012455 |
| Dermatitis exfoliative generalised | 10012456 |
| Drug reaction with eosinophilia and systemic symptoms | 10073508 |
| Epidermal necrosis | 10059284 |
| Erythema multiforme | 10015218 |
| Erythrodermic atopic dermatitis | 10082985 |
| Exfoliative rash | 10064579 |
| Oculomucocutaneous syndrome | 10030081 |
| SJS-TEN overlap | 10083164 |
| Skin necrosis | 10040893 |
| Stevens-Johnson syndrome | 10042033 |
| Target skin lesion | 10081998 |
| Toxic epidermal necrolysis | 10044223 |
| Toxic skin eruption | 10057970 |
| Addition selected preferred terms from HLTs 'Rashes, eruptions and exanthems NEC', HLT Code 1005266; 'Pruritus NEC', HLT Code 10049293, 'Pustular conditions', HLT Code 10037573; 'Dermatitis ascribed to specific agent', HLT Code 10012437. | |
| Preferred Term | PT Code |
| Eyelid rash | 10074620 |
| Genital rash | 10018175 |
| Mucocutaneous rash | 10056671 |

| SMQ: Severe Cutaneous Adverse Reactions<br>SMQ Code: 20000020<br>Category: A<br>Scope: Narrow | |
|---|---|
| Nodular rash | 10075807 |
| Perineal rash | 10075364 |
| Rash | 10037844 |
| Rash erythematous | 10037855 |
| Rash generalised | 10037858 |
| Rash macular | 10037867 |
| Rash maculo-papular | 10037868 |
| Rash maculovesicular | 10050004 |
| Rash morbilliform | 10037870 |
| Rash papular | 10037876 |
| Rash rubelliform | 10057984 |
| Rash scarlatiniform | 10037890 |
| Rash vesicular | 10037898 |
| Rash pruritic | 10037884 |
| Rash follicular | 10037857 |
| Rash pustular | 10037888 |
| Drug eruption | 10013687 |

# 13.9.5. Prolongation of the Corrected QT Interval of the ECG in Supra Therapeutic Doses

Medical concept of QT prolongation and complications. Only narrow terms from SMQ 'Torsade de pointes/QT prolongation' selected plus one additional PT under HLT 'ECG investigations'.

| SMQ: Torsade de pointes/QT prolongation<br>SMQ Code: 20000001<br>Category: A<br>Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Electrocardiogram QT interval abnormal | 10063748 |

| SMQ: Torsade de pointes/QT prolongation<br>SMQ Code: 20000001<br>Category: A<br>Scope: Narrow | |
|---|---|
| Electrocardiogram QT prolonged | 10014387 |
| Long QT syndrome | 10024803 |
| Long QT syndrome congenital | 10057926 |
| Torsade de pointes | 10044066 |
| Ventricular tachycardia | 10047302 |
| Additional selected preferred terms from HLT 'ECG investigations', HLT Code 10053104. | |
| Preferred Term | PT Code |
| Electrocardiogram repolarisation abnormality | 10052464 |

# 13.9.6. Suicidal Ideation/Behaviour

Medical concept of suicidal ideation and behaviour. Sub-SMQ 'Suicide/self-injury' (SMQ) from parent SMQ of 'Depression and Suicide/Self Injury (SMQ Code 20000035)'. Only narrow terms from the sub-SMQ selected.

| SMQ: 'Depression and Suicide/Self Injury' SMQ Code: 20000035 Sub-SMQ: 'Suicide/self-injury' Category: A Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Assisted suicide | 10079105 |
| Columbia suicide severity rating scale abnormal | 10075616 |
| Completed suicide | 10010144 |
| Depression suicidal | 10012397 |
| Intentional overdose | 10022523 |
| Intentional self-injury | 10022524 |
| Poisoning deliberate | 10036000 |
| Self-injurious ideation | 10051154 |
| Suicidal behaviour | 10065604 |

| SMQ: 'Depression and Suicide/Self Injury' SMQ Code: 20000035 Sub-SMQ: 'Suicide/self-injury' Category: A Scope: Narrow | |
|---|---|
| Suicidal ideation | 10042458 |
| Suicide attempt | 10042464 |
| Suicide threat | 10077417 |
| Suspected suicide | 10082458 |
| Suspected suicide attempt | 10081704 |

# 13.9.7. Depression

Medical concept of Depression. Sub-SMQ 'Depression (excl suicide and self-injury)' (SMQ) from parent SMQ of 'Depression and Suicide/Self Injury'. Only narrow terms from the sub-SMQ selected.

| SMQ: ''Depression and Suicide/Self Injury' SMQ Code: 20000035 Sub-SMQ: 'Depression (excl suicide and self-injury)' Category: A Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Activation syndrome | 10066817 |
| Adjustment disorder with depressed mood | 10001297 |
| Adjustment disorder with mixed anxiety and depressed mood | 10001299 |
| Agitated depression | 10001496 |
| Anhedonia | 10002511 |
| Antidepressant therapy | 10054976 |
| Childhood depression | 10068631 |
| Decreased interest | 10011971 |
| Depressed mood | 10012374 |
| Depression | 10012378 |
| Depression rating scale score increased | 10084390 |
| Discouragement | 10084257 |
| Depression postoperative | 10012390 |
| Depressive symptom | 10054089 |
| Dysphoria | 10013954 |
| Electroconvulsive therapy | 10014404 |
| Feeling guilty | 10049708 |
| Feeling of despair | 10016344 |
| Feelings of worthlessness | 10016374 |
| Helplessness | 10077169 |

| SMQ: ''Depression and Suicide/Self Injury' SMQ Code: 20000035 Sub-SMQ: 'Depression (excl suicide and self-injury)' Category: A Scope: Narrow | |
|---|---|
| Major depression | 10057840 |
| Menopausal depression | 10067371 |
| Mixed anxiety and depressive disorder | 10080836 |
| Perinatal depression | 10078366 |
| Persistent depressive disorder | 10077804 |
| Post stroke depression | 10070606 |
| Postictal depression | 10071324 |

# 13.9.8. Bipolar Disorder

Medical concept of bipolar disorder. All preferred terms from HLGT 'Manic and Bipolar mood disorders and disturbances' under SOC "Psychiatric disorders"; HLGT Code 10026753.

| Preferred Term | PT Code |
|----------------------|----------|
| Bipolar I disorder | 10004939 |
| Bipolar II disorder | 10004940 |
| Bipolar disorder | 10057667 |
| Cyclothymic disorder | 10011724 |
| Hypomania | 10021030 |
| Mania | 10026749 |
| Manic symptom | 10084119 |

# 13.9.9. Psychosis

Medical concept of psychosis. Only narrow terms from SMQ 'Psychosis and psychotic disorders' selected.

| SMQ: Psychosis and psychotic disorders' SMQ Code: 20000117 Preferred Code: 20000117 Category: A Scope: Narrow PT Code Preferred Term PT Code Acute psychosis 10001022 Alcoholic psychosis 10001632 Alice in wonderland syndrome 10001666 Brief psychotic disorder with marked stressors 10056395 Brief psychotic disorder, with postpartum onset 1006362 Charles Bonnet syndrome 1006334 Childhood psychosis 10061040 Clang associations 10061040 Clang associations 10012032 Cotard's syndrome 1001223 Delusion 10012239 Delusion of grandeur 10012241 Delusion of parasitosis 10012241 Delusion of reference 10012242 Delusion of replacement 10012245 Delusion of theft 10012245 Delusional disorder, grandiose type 10012250 Delusional disorder, jealous type 10012250 Delusional disorder, persecutory type 10012252 Delusional disorder, somatic type 10012255 <th></th> <th></th> | | |
|---|---|---|
| Acute psychosis 10001022 Alcoholic psychosis 10001632 Alice in wonderland syndrome 10001666 Brief psychotic disorder with marked stressors 10048549 Brief psychotic disorder without marked stressors 10056395 Brief psychotic disorder, with postpartum onset 10006362 Charles Bonnet syndrome 10063354 Childhood psychosis 10061040 Clang associations 1009232 Cotard's syndrome 10059591 Delusion 10012239 Delusion of grandeur 10012241 Delusion of parasitosis 10012242 Delusion of reference 10012244 Delusion of replacement 10012245 Delusion of theft 10084030 Delusional disorder, crotomanic type 10012251 Delusional disorder, grandiose type 10012252 Delusional disorder, mixed type 10053195 Delusional disorder, persecutory type 10053195 Delusional disorder, unspecified type 10012255 Delusional perception 10012258 | SMQ Code: 20000117<br>Category: A | |
| Alcoholic psychosis Alice in wonderland syndrome 10001666 Brief psychotic disorder with marked stressors 10048549 Brief psychotic disorder without marked stressors 10056395 Brief psychotic disorder, with postpartum onset 10006362 Charles Bonnet syndrome 10063354 Childhood psychosis 10061040 Clang associations 1009232 Cotard's syndrome 10059591 Delusion 10012239 Delusion of grandeur 10012241 Delusion of parasitosis 10012242 Delusion of reference 10012244 Delusion of replacement 10012245 Delusion of theft 10084030 Delusional disorder, erotomanic type 10012250 Delusional disorder, grandiose type 10012252 Delusional disorder, mixed type 10012252 Delusional disorder, persecutory type 10012254 Delusional disorder, somatic type 10012255 Delusional disorder, unspecified type 10012255 Delusional perception 10012258 | Preferred Term | PT Code |
| Alice in wonderland syndrome Brief psychotic disorder with marked stressors Brief psychotic disorder without marked stressors Brief psychotic disorder, with postpartum onset 1006362 Charles Bonnet syndrome 10063354 Childhood psychosis 10061040 Clang associations 1009232 Cotard's syndrome 10059591 Delusion 10012239 Delusion of grandeur 10012241 Delusion of parasitosis 10012242 Delusion of reference 10012244 Delusion of replacement 10012245 Delusion of theft 10084030 Delusional disorder, erotomanic type 10012250 Delusional disorder, jealous type 10012252 Delusional disorder, mixed type 10012252 Delusional disorder, persecutory type 10053195 Delusional disorder, somatic type 10012254 Delusional disorder, unspecified type 10012255 Delusional perception 10012258 | Acute psychosis | 10001022 |
| Brief psychotic disorder with marked stressors Brief psychotic disorder without marked stressors Brief psychotic disorder, with postpartum onset 1006352 Charles Bonnet syndrome 10063354 Childhood psychosis 10061040 Clang associations 1009232 Cotard's syndrome 10059591 Delusion 10012239 Delusion of grandeur 10012241 Delusion of parasitosis 10012242 Delusion of reference 10012244 Delusion of replacement 10012245 Delusional disorder, erotomanic type 10012250 Delusional disorder, jealous type 10012252 Delusional disorder, persecutory type 10012254 Delusional disorder, persecutory type 10012255 Delusional disorder, unspecified type 10012258 Delusional perception 10012258 | Alcoholic psychosis | 10001632 |
| Brief psychotic disorder without marked stressors Brief psychotic disorder, with postpartum onset 10006362 Charles Bonnet syndrome 10063354 Childhood psychosis 10061040 Clang associations 10009232 Cotard's syndrome 10012239 Delusion Delusion of grandeur Delusion of parasitosis 10012242 Delusion of reference 10012244 Delusion of replacement 10012245 Delusion of theft 10084030 Delusional disorder, erotomanic type Delusional disorder, grandiose type Delusional disorder, mixed type Delusional disorder, persecutory type Delusional disorder, somatic type Delusional disorder, somatic type Delusional disorder, somatic type Delusional disorder, somatic type Delusional disorder, unspecified type Delusional perception 10012258 | Alice in wonderland syndrome | 10001666 |
| Brief psychotic disorder, with postpartum onset Charles Bonnet syndrome 10063354 Childhood psychosis 10061040 Clang associations 10009232 Cotard's syndrome 10012239 Delusion Delusion of grandeur Delusion of parasitosis 10012241 Delusion of reference 10012244 Delusion of replacement 10012245 Delusion of theft 10084030 Delusional disorder, erotomanic type 10012250 Delusional disorder, jealous type 10012251 Delusional disorder, mixed type Delusional disorder, persecutory type Delusional disorder, somatic type 10012254 Delusional disorder, somatic type 10012255 Delusional disorder, unspecified type Delusional perception 10012258 | Brief psychotic disorder with marked stressors | 10048549 |
| Charles Bonnet syndrome 10063354 Childhood psychosis 10061040 Clang associations 10009232 Cotard's syndrome 10059591 Delusion 10012239 Delusion of grandeur 10012241 Delusion of parasitosis 10012242 Delusion of reference 10012244 Delusion of replacement 10012245 Delusion of theft 10084030 Delusional disorder, erotomanic type 10012249 Delusional disorder, grandiose type 10012250 Delusional disorder, mixed type 10012252 Delusional disorder, persecutory type 10053195 Delusional disorder, somatic type 10012254 Delusional disorder, somatic type 10012255 Delusional disorder, unspecified type 10012255 Delusional disorder, unspecified type 10012255 Delusional perception 10012258 | Brief psychotic disorder without marked stressors | 10056395 |
| Childhood psychosis 10061040 Clang associations 10009232 Cotard's syndrome 10012239 Delusion 10012241 Delusion of grandeur 10012241 Delusion of parasitosis 10012242 Delusion of reference 10012244 Delusion of replacement 10012245 Delusion of theft 10084030 Delusional disorder, erotomanic type 10012249 Delusional disorder, grandiose type 10012250 Delusional disorder, mixed type 10012251 Delusional disorder, persecutory type 10053195 Delusional disorder, somatic type 10012254 Delusional disorder, unspecified type 10012255 Delusional perception 10012258 | Brief psychotic disorder, with postpartum onset | 10006362 |
| Clang associations 10009232 Cotard's syndrome 10059591 Delusion 10012239 Delusion of grandeur 10012241 Delusion of parasitosis 10012242 Delusion of reference 10012244 Delusion of replacement 10012245 Delusion of theft 10084030 Delusional disorder, erotomanic type 10012249 Delusional disorder, grandiose type 10012250 Delusional disorder, jealous type 10012251 Delusional disorder, mixed type 10012252 Delusional disorder, persecutory type 10053195 Delusional disorder, somatic type 10012254 Delusional disorder, unspecified type 10012255 Delusional perception 10012258 | Charles Bonnet syndrome | 10063354 |
| Cotard's syndrome 10059591 Delusion 10012239 Delusion of grandeur 10012241 Delusion of parasitosis 10012242 Delusion of reference 10012244 Delusion of replacement 10012245 Delusion of theft 10084030 Delusional disorder, erotomanic type 10012249 Delusional disorder, grandiose type 10012250 Delusional disorder, jealous type 10012251 Delusional disorder, mixed type 10053195 Delusional disorder, somatic type 10012254 Delusional disorder, unspecified type 10012255 Delusional perception 10012255 | Childhood psychosis | 10061040 |
| Delusion 10012239 Delusion of grandeur 10012241 Delusion of parasitosis 10012242 Delusion of reference 10012244 Delusion of replacement 10012245 Delusion of theft 10084030 Delusional disorder, erotomanic type 10012249 Delusional disorder, grandiose type 10012250 Delusional disorder, jealous type 10012251 Delusional disorder, mixed type 10012252 Delusional disorder, persecutory type 10053195 Delusional disorder, somatic type 10012254 Delusional disorder, unspecified type 10012255 Delusional perception 10012258 | Clang associations | 10009232 |
| Delusion of grandeur Delusion of parasitosis 10012242 Delusion of reference 10012244 Delusion of replacement 10012245 Delusion of theft 10084030 Delusional disorder, erotomanic type 10012249 Delusional disorder, grandiose type 10012250 Delusional disorder, jealous type 10012251 Delusional disorder, mixed type 10012252 Delusional disorder, persecutory type 10053195 Delusional disorder, somatic type 10012254 Delusional disorder, unspecified type 10012255 Delusional perception 10012258 | Cotard's syndrome | 10059591 |
| Delusion of parasitosis Delusion of reference 10012244 Delusion of replacement 10012245 Delusion of theft 10084030 Delusional disorder, erotomanic type 10012249 Delusional disorder, grandiose type 10012250 Delusional disorder, jealous type 10012251 Delusional disorder, mixed type 10012252 Delusional disorder, persecutory type 10053195 Delusional disorder, somatic type 10012254 Delusional disorder, unspecified type 10012255 Delusional perception 10012258 | Delusion | 10012239 |
| Delusion of reference 10012244 Delusion of replacement 10012245 Delusion of theft 10084030 Delusional disorder, erotomanic type 10012249 Delusional disorder, grandiose type 10012250 Delusional disorder, jealous type 10012251 Delusional disorder, mixed type 10012252 Delusional disorder, persecutory type 10053195 Delusional disorder, somatic type 10012254 Delusional disorder, unspecified type 10012255 Delusional perception 10012258 | Delusion of grandeur | 10012241 |
| Delusion of replacement 10012245 Delusion of theft 10084030 Delusional disorder, erotomanic type 10012249 Delusional disorder, grandiose type 10012250 Delusional disorder, jealous type 10012251 Delusional disorder, mixed type 10012252 Delusional disorder, persecutory type 10053195 Delusional disorder, somatic type 10012254 Delusional disorder, unspecified type 10012255 Delusional perception 10012258 | Delusion of parasitosis | 10012242 |
| Delusion of theft 10084030 Delusional disorder, erotomanic type 10012249 Delusional disorder, grandiose type 10012250 Delusional disorder, jealous type 10012251 Delusional disorder, mixed type 10012252 Delusional disorder, persecutory type 10053195 Delusional disorder, somatic type 10012254 Delusional disorder, unspecified type 10012255 Delusional perception 10012258 | Delusion of reference | 10012244 |
| Delusional disorder, erotomanic type Delusional disorder, grandiose type Delusional disorder, jealous type Delusional disorder, mixed type Delusional disorder, persecutory type Delusional disorder, somatic type Delusional disorder, unspecified type Delusional perception 10012259 10012259 10012259 10012258 | Delusion of replacement | 10012245 |
| Delusional disorder, grandiose type Delusional disorder, jealous type Delusional disorder, mixed type Delusional disorder, persecutory type Delusional disorder, somatic type Delusional disorder, unspecified type Delusional perception 10012250 10012251 10012252 10012252 10012254 | Delusion of theft | 10084030 |
| Delusional disorder, jealous type 10012251 Delusional disorder, mixed type 10012252 Delusional disorder, persecutory type 10053195 Delusional disorder, somatic type 10012254 Delusional disorder, unspecified type 10012255 Delusional perception 10012258 | Delusional disorder, erotomanic type | 10012249 |
| Delusional disorder, mixed type Delusional disorder, persecutory type Delusional disorder, somatic type Delusional disorder, unspecified type Delusional perception 10012252 10012254 | Delusional disorder, grandiose type | 10012250 |
| Delusional disorder, persecutory type 10053195 Delusional disorder, somatic type 10012254 Delusional disorder, unspecified type 10012255 Delusional perception 10012258 | Delusional disorder, jealous type | 10012251 |
| Delusional disorder, somatic type 10012254 Delusional disorder, unspecified type 10012255 Delusional perception 10012258 | Delusional disorder, mixed type | 10012252 |
| Delusional disorder, unspecified type 10012255 Delusional perception 10012258 | Delusional disorder, persecutory type | 10053195 |
| Delusional perception 10012258 | Delusional disorder, somatic type | 10012254 |
| | Delusional disorder, unspecified type | 10012255 |
| Dementia of the Alzheimer's type, with delusions 10012295 | Delusional perception | 10012258 |
| | Dementia of the Alzheimer's type, with delusions | 10012295 |

| SMQ Code: 20000117 Category: A Scope: Narrow 10063033 Depressive delusion 10012411 Epileptic psychosis 10059232 Erotomanic delusion 10015134 Flight of ideas 10016777 Hallucination 10019063 Hallucination, auditory 10019070 Hallucination, gustatory 10019071 Hallucination, olfactory 10019072 Hallucination, synaesthetic 10062824 Hallucination, visual 10019074 Hallucination, wisual 10019075 Hallucinations, mixed 10019075 Hypnagogic hallucination 10020927 Hypnopompic hallucination 10020928 Hysterical psychosis 10062645 Ideas of reference 10021121 Illusion 10021403 Jealous delusion 10023164 Loose associations 10024825 Mixed delusion 10076429 Neclogism 10028916 Neuroleptic-induced deficit syndrome 10075295 Paranoia 10033864 Paranoid personality disorder 10033869 < | | |
|---|---|---|
| Category: A Scope: Narrow 10063033 Depressive delusion 10063033 Derailment 10012411 Epileptic psychosis 10059232 Erotomanic delusion 10015134 Flight of ideas 10016777 Hallucination 10019063 Hallucination, auditory 10019070 Hallucination, gustatory 10019071 Hallucination, olfactory 10019072 Hallucination, synaesthetic 10062824 Hallucination, tactile 10019074 Hallucination, wisual 10019075 Hallucinations, mixed 10019079 Hypnagogic hallucination 10020927 Hypnopompic hallucination 10020927 Hypnopompic hallucination 10020928 Hysterical psychosis 1002645 Ideas of reference 1002112 Illusion 10021403 Jealous delusion 10023164 Loose associations 10024825 Mixed delusion 10076429 Neuroleptic-induced deficit syndrome 10075295 Paranoia 1 | SMQ: 'Psychosis and psychotic disorders' | |
| Scope: Narrow 10063033 Depressive delusion 10063033 Derailment 10012411 Epileptic psychosis 10059232 Erotomanic delusion 10015134 Flight of ideas 10016777 Hallucination 10019063 Hallucination, auditory 10019070 Hallucination, gustatory 10019071 Hallucination, olfactory 10019072 Hallucination, synaesthetic 10062824 Hallucination, tactile 10019074 Hallucination, visual 10019079 Hypnagogic hallucination 10020927 Hypnopompic hallucination 10020927 Hypnopompic hallucination 10020928 Hysterical psychosis 10021403 Ideas of reference 10021212 Illusion 10021403 Jealous delusion 10023164 Loose associations 10024825 Mixed delusion 10076429 Neuroleptic-induced deficit syndrome 10075295 Paranoia 10033864 Paranoid personality disorder 100 | | |
| Derailment 10012411 Epileptic psychosis 10059232 Erotomanic delusion 10015134 Flight of ideas 10016777 Hallucination 10019063 Hallucination, auditory 10019070 Hallucination, gustatory 10019071 Hallucination, olfactory 10019072 Hallucination, synaesthetic 10062824 Hallucination, tactile 10019074 Hallucination, visual 10019079 Hypnagogic hallucination 10020927 Hypnopompic hallucination 10020927 Hysterical psychosis 10062645 Ideas of reference 10021212 Illusion 10021403 Jealous delusion 10023164 Loose associations 10024825 Mixed delusion 10076429 Neologism 10075295 Paranoia 10033864 Paranoid personality disorder 10033869 | Scope: Narrow | |
| Epileptic psychosis 10059232 Erotomanic delusion 10015134 Flight of ideas 10016777 Hallucination 10019063 Hallucination, auditory 10019070 Hallucination, gustatory 10019071 Hallucination, olfactory 10019072 Hallucination, synaesthetic 10062824 Hallucination, tactile 10019074 Hallucination, visual 10019075 Hallucinations, mixed 10019079 Hypnagogic hallucination 10020927 Hypnopompic hallucination 10020928 Hysterical psychosis 10062645 Ideas of reference 10021212 Illusion 10021403 Jealous delusion 10023164 Loose associations 10024825 Mixed delusion 10076429 Neologism 10028916 Neuroleptic-induced deficit syndrome 10033864 Paranoid personality disorder 10033869 | Depressive delusion | 10063033 |
| Erotomanic delusion 10015134 Flight of ideas 10016777 Hallucination 10019063 Hallucination, auditory 10019070 Hallucination, gustatory 10019071 Hallucination, olfactory 10019072 Hallucination, synaesthetic 10062824 Hallucination, tactile 10019074 Hallucination, visual 10019075 Hallucinations, mixed 10019079 Hypnagogic hallucination 10020927 Hypnopompic hallucination 10020928 Hysterical psychosis 10062645 Ideas of reference 10021212 Illusion 10021403 Jealous delusion 10023164 Loose associations 10024825 Mixed delusion 10076429 Neologism 10028916 Neuroleptic-induced deficit syndrome 10073864 Paranoia 10033864 Paranoid personality disorder 10033869 | Derailment | 10012411 |
| Flight of ideas 10016777 Hallucination 10019063 Hallucination, auditory 10019070 Hallucination, gustatory 10019071 Hallucination, olfactory 10019072 Hallucination, synaesthetic 10062824 Hallucination, tactile 10019074 Hallucination, visual 10019075 Hallucinations, mixed 10019079 Hypnagogic hallucination 10020927 Hypnopompic hallucination 10020928 Hysterical psychosis 10062645 Ideas of reference 10021212 Illusion 10021403 Jealous delusion 10023164 Loose associations 10024825 Mixed delusion 10076429 Neologism 10028916 Neuroleptic-induced deficit syndrome 10073864 Paranoid personality disorder 10033864 | Epileptic psychosis | 10059232 |
| Hallucination 10019063 Hallucination, auditory 10019070 Hallucination, gustatory 10019071 Hallucination, olfactory 10019072 Hallucination, synaesthetic 10062824 Hallucination, tactile 10019074 Hallucination, visual 10019075 Hallucinations, mixed 10019079 Hypnagogic hallucination 10020927 Hypnopompic hallucination 10020928 Hysterical psychosis 10062645 Ideas of reference 10021212 Illusion 10021403 Jealous delusion 10023164 Loose associations 10024825 Mixed delusion 10076429 Neologism 10078916 Neuroleptic-induced deficit syndrome 10075295 Paranoia 10033864 Paranoid personality disorder 10033869 | Erotomanic delusion | 10015134 |
| Hallucination, auditory 10019070 Hallucination, gustatory 10019071 Hallucination, olfactory 10019072 Hallucination, synaesthetic 10062824 Hallucination, tactile 10019074 Hallucination, visual 10019075 Hallucinations, mixed 10019079 Hypnagogic hallucination 10020927 Hypnopompic hallucination 10020928 Hysterical psychosis 10062645 Ideas of reference 10021212 Illusion 10021403 Jealous delusion 10023164 Loose associations 10024825 Mixed delusion 10076429 Neologism 10078916 Neuroleptic-induced deficit syndrome 10075295 Paranoia 10033864 Paranoid personality disorder 10033869 | Flight of ideas | 10016777 |
| Hallucination, gustatory 10019071 Hallucination, olfactory 10019072 Hallucination, synaesthetic 10062824 Hallucination, tactile 10019074 Hallucination, visual 10019075 Hallucinations, mixed 10019079 Hypnagogic hallucination 10020927 Hypnopompic hallucination 10020928 Hysterical psychosis 10062645 Ideas of reference 10021212 Illusion 10021403 Jealous delusion 10023164 Loose associations 10024825 Mixed delusion 10076429 Neologism 10078295 Paranoia 10033864 Paranoid personality disorder 10033869 | Hallucination | 10019063 |
| Hallucination, olfactory 10019072 Hallucination, synaesthetic 10062824 Hallucination, tactile 10019074 Hallucination, visual 10019075 Hallucinations, mixed 10019079 Hypnagogic hallucination 10020927 Hypnopompic hallucination 10020928 Hysterical psychosis 10062645 Ideas of reference 10021212 Illusion 10021403 Jealous delusion 10023164 Loose associations 10024825 Mixed delusion 10076429 Neologism 10028916 Neuroleptic-induced deficit syndrome 10075295 Paranoia 10033864 Paranoid personality disorder 10033869 | Hallucination, auditory | 10019070 |
| Hallucination, synaesthetic 10062824 Hallucination, tactile 10019074 Hallucination, visual 10019075 Hallucinations, mixed 10019079 Hypnagogic hallucination 10020927 Hypnopompic hallucination 10020928 Hysterical psychosis 10062645 Ideas of reference 10021212 Illusion 10021403 Jealous delusion 10023164 Loose associations 10024825 Mixed delusion 10076429 Neologism 10028916 Neuroleptic-induced deficit syndrome 10075295 Paranoia 10033864 Paranoid personality disorder 10033869 | Hallucination, gustatory | 10019071 |
| Hallucination, tactile 10019074 Hallucination, visual 10019075 Hallucinations, mixed 10019079 Hypnagogic hallucination 10020927 Hypnopompic hallucination 10020928 Hysterical psychosis 10062645 Ideas of reference 10021212 Illusion 10021403 Jealous delusion 10023164 Loose associations 10024825 Mixed delusion 10076429 Neologism 10075295 Paranoia 10033864 Paranoid personality disorder 10033869 | Hallucination, olfactory | 10019072 |
| Hallucination, visual 10019075 Hallucinations, mixed 10019079 Hypnagogic hallucination 10020927 Hypnopompic hallucination 10020928 Hysterical psychosis 10062645 Ideas of reference 10021212 Illusion 10021403 Jealous delusion 10023164 Loose associations 10024825 Mixed delusion 10076429 Neologism 10075295 Paranoia 10033864 Paranoid personality disorder 10033869 | Hallucination, synaesthetic | 10062824 |
| Hallucinations, mixed 10019079 Hypnagogic hallucination 10020927 Hypnopompic hallucination 10020928 Hysterical psychosis 10062645 Ideas of reference 10021212 Illusion 10021403 Jealous delusion 10023164 Loose associations 10024825 Mixed delusion 10076429 Neologism 10028916 Neuroleptic-induced deficit syndrome 10075295 Paranoia 10033864 Paranoid personality disorder 10033869 | Hallucination, tactile | 10019074 |
| Hypnagogic hallucination 10020927 Hypnopompic hallucination 10020928 Hysterical psychosis 10062645 Ideas of reference 10021212 Illusion 10021403 Jealous delusion 10023164 Loose associations 10024825 Mixed delusion 10076429 Neologism 10028916 Neuroleptic-induced deficit syndrome 10075295 Paranoia 10033864 Paranoid personality disorder 10033869 | Hallucination, visual | 10019075 |
| Hypnopompic hallucination 10020928 Hysterical psychosis 10062645 Ideas of reference 10021212 Illusion 10021403 Jealous delusion 10023164 Loose associations 10024825 Mixed delusion 10076429 Neologism 10028916 Neuroleptic-induced deficit syndrome 10075295 Paranoia 10033864 Paranoid personality disorder 10033869 | Hallucinations, mixed | 10019079 |
| Hysterical psychosis 10062645 Ideas of reference 10021212 Illusion 10021403 Jealous delusion 10023164 Loose associations 10024825 Mixed delusion 10076429 Neologism 10028916 Neuroleptic-induced deficit syndrome 10075295 Paranoia 10033864 Paranoid personality disorder 10033869 | Hypnagogic hallucination | 10020927 |
| Ideas of reference 10021212 Illusion 10021403 Jealous delusion 10023164 Loose associations 10024825 Mixed delusion 10076429 Neologism 10028916 Neuroleptic-induced deficit syndrome 10075295 Paranoia 10033864 Paranoid personality disorder 10033869 | Hypnopompic hallucination | 10020928 |
| Illusion 10021403 Jealous delusion 10023164 Loose associations 10024825 Mixed delusion 10076429 Neologism 10028916 Neuroleptic-induced deficit syndrome 10075295 Paranoia 10033864 Paranoid personality disorder 10033869 | Hysterical psychosis | 10062645 |
| Jealous delusion 10023164 Loose associations 10024825 Mixed delusion 10076429 Neologism 10028916 Neuroleptic-induced deficit syndrome 10075295 Paranoia 10033864 Paranoid personality disorder 10033869 | Ideas of reference | 10021212 |
| Loose associations Mixed delusion 10076429 Neologism 10028916 Neuroleptic-induced deficit syndrome 10075295 Paranoia 10033864 Paranoid personality disorder 10033869 | Illusion | 10021403 |
| Mixed delusion 10076429 Neologism 10028916 Neuroleptic-induced deficit syndrome 10075295 Paranoia 10033864 Paranoid personality disorder 10033869 | Jealous delusion | 10023164 |
| Neologism10028916Neuroleptic-induced deficit syndrome10075295Paranoia10033864Paranoid personality disorder10033869 | Loose associations | 10024825 |
| Neuroleptic-induced deficit syndrome 10075295 Paranoia 10033864 Paranoid personality disorder 10033869 | Mixed delusion | 10076429 |
| Paranoia 10033864 Paranoid personality disorder 10033869 | Neologism | 10028916 |
| Paranoid personality disorder 10033869 | Neuroleptic-induced deficit syndrome | 10075295 |
| | Paranoia | 10033864 |
| Parkinson's disease psychosis 10074835 | Paranoid personality disorder | 10033869 |
| | Parkinson's disease psychosis | 10074835 |

| SMQ: 'Psychosis and psychotic disorders' SMQ Code: 20000117 Category: A Scope: Narrow | |
|---|---|
| Paroxysmal perceptual alteration | 10063117 |
| Persecutory delusion | 10034702 |
| Postictal psychosis | 10070669 |
| Post-injection delirium sedation syndrome | 10072851 |
| Posturing | 10036437 |
| Psychosis postoperative | 10065617 |
| Psychotic behaviour | 10037249 |
| Psychotic disorder | 10061920 |
| Psychotic disorder due to a general medical condition | 10061921 |
| Reactive psychosis | 10053632 |
| Rebound psychosis | 10074833 |
| Schizoaffective disorder | 10039621 |
| Schizoaffective disorder bipolar type | 10068889 |
| Schizoaffective disorder depressive type | 10068890 |
| Schizophrenia | 10039626 |
| Schizophreniform disorder | 10039647 |
| Schizotypal personality disorder | 10039651 |
| Senile psychosis | 10039987 |
| Shared psychotic disorder | 10040535 |
| Somatic delusion | 10041317 |
| Somatic hallucination | 10062684 |
| Substance-induced psychotic disorder | 10072388 |
| Tangentiality | 10043114 |
| Thought blocking | 10043495 |
| Thought broadcasting | 10052214 |
| Thought insertion | 10043496 |

| SMQ: 'Psychosis and psychotic disorders' SMQ Code: 20000117 Category: A Scope: Narrow | |
|---|---|
| Thought withdrawal | 10043497 |
| Transient psychosis | 10056326 |
| Waxy flexibility | 10047853 |

## 13.9.10. Mood Disorders

Medical concept of mood disorders. All preferred terms from HLGT 'Mood disorders and disturbances NEC', under SOC 'Psychiatric disorders'; HLGT Code 10027946.

| Preferred Term | PT Code |
|----------------------------------|----------|
| Affect lability | 10054196 |
| Affective ambivalence | 10077173 |
| Affective disorder | 10001443 |
| Alexithymia | 10077719 |
| Anger | 10002368 |
| Apathy | 10002942 |
| Blunted affect | 10005885 |
| Boredom | 10048909 |
| Constricted affect | 10010778 |
| Crying | 10011469 |
| Diencephalic syndrome of infancy | 10012774 |
| Discouragement | 10084257 |
| Dysphoria | 10013954 |
| Emotional disorder | 10014551 |
| Emotional distress | 10049119 |
| Emotional poverty | 10014557 |
| Euphoric mood | 10015535 |
| Flat affect | 10016759 |

| Preferred Term | PT Code |
|--------------------------------------------------|----------|
| Frustration tolerance decreased | 10077753 |
| Inappropriate affect | 10021588 |
| Irritability | 10022998 |
| Laziness | 10051602 |
| Lethargy | 10024264 |
| Listless | 10024642 |
| Moaning | 10027783 |
| Mood altered | 10027940 |
| Mood disorder due to a general medical condition | 10027944 |
| Mood swings | 10027951 |
| Morose | 10027977 |
| Neuroleptic-induced deficit syndrome | 10075295 |
| Premenstrual dysphoric disorder | 10051537 |
| Premenstrual syndrome | 10036618 |
| Screaming | 10039740 |
| Seasonal affective disorder | 10039775 |
| Steroid withdrawal syndrome | 10042028 |
| Substance-induced mood disorder | 10072387 |

# 13.9.11. Anxiety

Notes: Medical concept of anxiety disorders. All preferred terms from HLGT "Anxiety disorders and symptoms", under SOC "Psychiatric disorders"; HLGT Code 10002861.

| Preferred Terms | PT Code |
|-----------------------|----------|
| Acrophobia | 10000605 |
| Activation syndrome | 10066817 |
| Acute stress disorder | 10001084 |
| Aerophobia | 10080300 |
| Agitation | 10001497 |

| Agitation postoperative 10049989 Agoraphobia 10001502 Akathisia 10001540 Algophobia 10078056 Animal phobia 10002518 Anniversary reaction 10074066 Anticipatory anxiety 10002758 Anxiety 10002855 Anxiety disorder 10057666 Anxiety disorder due to a general medical condition 1005859 Arachnophobia 10051408 Astraphobia 10071070 Body dysmorphic disorder 10052793 Burnout syndrome 10052793 Burnout syndrome 1006369 Catastrophic reaction 10082329 Cibophobia 10082413 Claustrophobia 10010219 Compulsive cheek biting 10076510 Compulsive handwashing 10071263 Compulsive hoarding 10068007 Compulsive shopping 10067948 Cryophobia 10082662 Dermatillomania 10065701 Dysmorphophobia 10049096 Emetophobia | Preferred Terms | PT Code |
|---|---|---|
| Akathisia 10001540 Algophobia 10078056 Animal phobia 10002518 Anniversary reaction 10074066 Anticipatory anxiety 10002758 Anxiety 10002855 Anxiety disorder 10057666 Anxiety disorder due to a general medical condition 1002859 Arachnophobia 10051408 Astraphobia 10071070 Body dysmorphic disorder 10052793 Burnout syndrome 10065369 Catastrophic reaction 10082329 Cibophobia 10082413 Claustrophobia 10009244 Compulsions 10010219 Compulsive cheek biting 10076510 Compulsive handwashing 10071263 Compulsive hoarding 10068007 Compulsive shopping 10067948 Cryophobia 10082662 Dermatillomania 10065701 Dysmorphophobia 10049096 | Agitation postoperative | 10049989 |
| Algophobia 10078056 Animal phobia 10002518 Anniversary reaction 10074066 Anticipatory anxiety 10002855 Anxiety 10002855 Anxiety 10002855 Anxiety disorder 10057666 Anxiety disorder 10051408 Astraphobia 10051408 Astraphobia 10071070 Body dysmorphic disorder 10065369 Catastrophic reaction 10082329 Cibophobia 10082413 Claustrophobia 10009244 Compulsions 10010219 Compulsive cheek bitting 10076510 Compulsive handwashing 10068007 Compulsive hoarding 10066241 Compulsive shopping 10067948 Cryophobia 10082662 Dermatillomania 10065701 Dysmorphophobioa 10082662 | Agoraphobia | 10001502 |
| Animal phobia 10002518 Anniversary reaction 10074066 Anticipatory anxiety 10002855 Anxiety 10002855 Anxiety disorder 10057666 Anxiety disorder due to a general medical condition 10002859 Arachnophobia 10078372 Autophobia 10071070 Body dysmorphic disorder 10052793 Burnout syndrome 10065369 Catastrophic reaction 10082329 Cibophobia 10082329 Cibophobia 10082413 Claustrophobia 10009244 Compulsive check biting 10076510 Compulsive check biting 10076241 Compulsive lip biting 10066241 Compulsive shopping 10065701 Dysmorphophobia 10082662 Dermatillomania 10065701 Dysmorphophobia 10049996 | Akathisia | 10001540 |
| Anniversary reaction 10074066 Anticipatory anxiety 10002758 Anxiety 10002855 Anxiety 10002855 Anxiety disorder 10057666 Anxiety disorder due to a general medical condition 10002859 Arachnophobia 10078372 Autophobia 10071070 Body dysmorphic disorder 10052793 Burnout syndrome 10065369 Catastrophic reaction 10082329 Cibophobia 10009244 Compulsions 10010219 Compulsive cheek biting 10076510 Compulsive handwashing 10071263 Compulsive lip biting 10066241 Compulsive shopping 10065701 Dysmorphophobia 10082662 Dermatillomania 10065701 Dysmorphophobia 10049096 | Algophobia | 10078056 |
| Anxiety 10002758 Anxiety 10002855 Anxiety 10002855 Anxiety disorder 10057666 Anxiety disorder due to a general medical condition 10002859 Arachnophobia 10051408 Astraphobia 10078372 Autophobia 10071070 Body dysmorphic disorder 10052793 Burnout syndrome 10065369 Catastrophic reaction 10082329 Cibophobia 10082413 Claustrophobia 10009244 Compulsions 10010219 Compulsive cheek biting 10076510 Compulsive handwashing 10076510 Compulsive lip biting 10066241 Compulsive shopping 100667948 Cryophobia 10082662 Dermatillomania 10065701 Dysmorphophobia 10049096 | Animal phobia | 10002518 |
| Anxiety | Anniversary reaction | 10074066 |
| Anxiety disorder 10057666 Anxiety disorder due to a general medical condition 10002859 Arachnophobia 10078372 Autophobia 10071070 Body dysmorphic disorder 10052793 Burnout syndrome 10065369 Catastrophic reaction 10082329 Cibophobia 10082413 Claustrophobia 10009244 Compulsions 10010219 Compulsive cheek biting 10071263 Compulsive handwashing 10071263 Compulsive hoarding 10066241 Compulsive shopping 10067948 Cryophobia 10082662 Dermatillomania 10049096 | Anticipatory anxiety | 10002758 |
| Anxiety disorder due to a general medical condition 10002859 Arachnophobia 10051408 Astraphobia 10078372 Autophobia 10071070 Body dysmorphic disorder 10052793 Burnout syndrome 10065369 Catastrophic reaction 10082329 Cibophobia 10082413 Claustrophobia 10010219 Compulsions 10010219 Compulsive cheek biting 10076510 Compulsive handwashing 10071263 Compulsive hoarding 10068007 Compulsive shopping 10067948 Cryophobia 10082662 Dermatillomania 10065701 Dysmorphophobia 10049096 | Anxiety | 10002855 |
| Arachnophobia 10051408 Astraphobia 10078372 Autophobia 10071070 Body dysmorphic disorder 10052793 Burnout syndrome 10065369 Catastrophic reaction 10082329 Cibophobia 10082413 Claustrophobia 10009244 Compulsions 10010219 Compulsive cheek biting 10076510 Compulsive handwashing 10071263 Compulsive hoarding 10068007 Compulsive shopping 10067948 Cryophobia 10082662 Dermatillomania 10065701 Dysmorphophobia 10049096 | Anxiety disorder | 10057666 |
| Astraphobia 10078372 Autophobia 10071070 Body dysmorphic disorder 10052793 Burnout syndrome 10065369 Catastrophic reaction 10082329 Cibophobia 10082413 Claustrophobia 10009244 Compulsions 10010219 Compulsive cheek biting 10076510 Compulsive handwashing 10071263 Compulsive hoarding 10068007 Compulsive shopping 1006241 Compulsive shopping 10067948 Cryophobia 10082662 Dermatillomania 10065701 Dysmorphophobia 10049096 | Anxiety disorder due to a general medical condition | 10002859 |
| Autophobia 10071070 Body dysmorphic disorder 10052793 Burnout syndrome 10065369 Catastrophic reaction 10082329 Cibophobia 10082413 Claustrophobia 10009244 Compulsions 10010219 Compulsive cheek biting 10076510 Compulsive handwashing 10071263 Compulsive hoarding 10068007 Compulsive shopping 10067948 Cryophobia 10082662 Dermatillomania 10065701 Dysmorphophobia 10049096 | Arachnophobia | 10051408 |
| Body dysmorphic disorder 10052793 Burnout syndrome 10065369 Catastrophic reaction 10082329 Cibophobia 10082413 Claustrophobia 10009244 Compulsions 10010219 Compulsive cheek biting 10076510 Compulsive handwashing 10071263 Compulsive hoarding 10068007 Compulsive lip biting 10066241 Compulsive shopping 10082662 Dermatillomania 10065701 Dysmorphophobia 10049096 | Astraphobia | 10078372 |
| Burnout syndrome 10065369 Catastrophic reaction 10082329 Cibophobia 10082413 Claustrophobia 10009244 Compulsions 10010219 Compulsive cheek biting 10076510 Compulsive handwashing 10071263 Compulsive hoarding 10068007 Compulsive lip biting 10066241 Compulsive shopping 10067948 Cryophobia 10082662 Dermatillomania 10049096 | Autophobia | 10071070 |
| Catastrophic reaction 10082329 Cibophobia 10082413 Claustrophobia 10009244 Compulsions 10010219 Compulsive cheek biting 10076510 Compulsive handwashing 10071263 Compulsive hoarding 10068007 Compulsive lip biting 10066241 Compulsive shopping 10082662 Dermatillomania 10065701 Dysmorphophobia 10049096 | Body dysmorphic disorder | 10052793 |
| Cibophobia 10082413 Claustrophobia 10009244 Compulsions 10010219 Compulsive cheek biting 10076510 Compulsive handwashing 10071263 Compulsive hoarding 10068007 Compulsive lip biting 10066241 Compulsive shopping 10087948 Cryophobia 10082662 Dermatillomania 10065701 Dysmorphophobia 10049096 | Burnout syndrome | 10065369 |
| Claustrophobia 10009244 Compulsions 10010219 Compulsive cheek biting 10076510 Compulsive handwashing 10071263 Compulsive hoarding 10068007 Compulsive lip biting 10066241 Compulsive shopping 10067948 Cryophobia 10082662 Dermatillomania 10065701 Dysmorphophobia 10049096 | Catastrophic reaction | 10082329 |
| Compulsions 10010219 Compulsive cheek biting 10076510 Compulsive handwashing 10071263 Compulsive hoarding 10068007 Compulsive lip biting 10066241 Compulsive shopping 10067948 Cryophobia 10082662 Dermatillomania 10065701 Dysmorphophobia 10049096 | Cibophobia | 10082413 |
| Compulsive cheek biting 10076510 Compulsive handwashing 10071263 Compulsive hoarding 10068007 Compulsive lip biting 10066241 Compulsive shopping 10067948 Cryophobia 10082662 Dermatillomania 10065701 Dysmorphophobia 10049096 | Claustrophobia | 10009244 |
| Compulsive handwashing 10071263 Compulsive hoarding 10068007 Compulsive lip biting 10066241 Compulsive shopping 10067948 Cryophobia 10082662 Dermatillomania 10065701 Dysmorphophobia 10049096 | Compulsions | 10010219 |
| Compulsive hoarding 10068007 Compulsive lip biting 10066241 Compulsive shopping 10067948 Cryophobia 10082662 Dermatillomania 10065701 Dysmorphophobia 10049096 | Compulsive cheek biting | 10076510 |
| Compulsive lip biting 10066241 Compulsive shopping 10067948 Cryophobia 10082662 Dermatillomania 10065701 Dysmorphophobia 10049096 | Compulsive handwashing | 10071263 |
| Compulsive shopping 10067948 Cryophobia 10082662 Dermatillomania 10065701 Dysmorphophobia 10049096 | Compulsive hoarding | 10068007 |
| Cryophobia 10082662 Dermatillomania 10065701 Dysmorphophobia 10049096 | Compulsive lip biting | 10066241 |
| Dermatillomania 10065701 Dysmorphophobia 10049096 | Compulsive shopping | 10067948 |
| Dysmorphophobia 10049096 | Cryophobia | 10082662 |
| | Dermatillomania | 10065701 |
| Emetophobia 10070637 | Dysmorphophobia | 10049096 |
| | Emetophobia | 10070637 |

| Preferred Terms | PT Code |
|---------------------------------------|----------|
| Fear | 10016275 |
| Fear of animals | 10016276 |
| Fear of closed spaces | 10016277 |
| Fear of crowded places | 10050365 |
| Fear of death | 10066392 |
| Fear of disease | 10016278 |
| Fear of eating | 10050366 |
| Fear of falling | 10048744 |
| Fear of injection | 10073753 |
| Fear of open spaces | 10016279 |
| Fear of pregnancy | 10067035 |
| Fear of surgery | 10084519 |
| Fear of weight gain | 10016280 |
| Fear-related avoidance of activities | 10080136 |
| Generalised anxiety disorder | 10018075 |
| Glossophobia | 10080077 |
| Haemophobia | 10073458 |
| Haphephobia | 10067580 |
| Herpetophobia | 10081809 |
| Hydrophobia | 10053317 |
| Hyperarousal | 10080831 |
| Immunisation anxiety related reaction | 10075205 |
| Kinesiophobia | 10078430 |
| Limited symptom panic attack | 10024511 |
| Mysophobia | 10078769 |
| Nail picking | 10066779 |
| Nervousness | 10029216 |
| Neurosis | 10029333 |

| Preferred Terms | PT Code |
|---|---|
| Noctiphobia | 10057946 |
| Nocturnal fear | 10057948 |
| Nosocomephobia | 10083993 |
| Nosophobia | 10063546 |
| Obsessive need for symmetry | 10077179 |
| Obsessive rumination | 10056264 |
| Obsessive thoughts | 10029897 |
| Obsessive-compulsive disorder | 10029898 |
| Obsessive-compulsive symptom | 10077894 |
| Ochlophobia | 10050095 |
| Osmophobia | 10060765 |
| Paediatric autoimmune neuropsychiatric disorders associated with streptococcal infection | 10072147 |
| Panic attack | 10033664 |
| Panic disorder | 10033666 |
| Panic reaction | 10033670 |
| Paruresis | 10069024 |
| Performance fear | 10034432 |
| Phagophobia | 10050096 |
| Pharmacophobia | 10069423 |
| Phobia | 10034912 |
| Phobia of driving | 10056676 |
| Phobia of exams | 10034913 |
| Phobic avoidance | 10034918 |
| Phonophobia | 10054956 |
| Photaugiaphobia | 10064420 |
| Postpartum anxiety | 10082233 |
| Postpartum neurosis | 10036419 |


| | T |
|--------------------------------|----------|
| Preferred Terms | PT Code |
| Postpartum stress disorder | 10056394 |
| Post-traumatic stress disorder | 10036316 |
| Procedural anxiety | 10075204 |
| Pseudoangina | 10056610 |
| Selective mutism | 10039917 |
| Separation anxiety disorder | 10040045 |
| Sitophobia | 10080170 |
| Social anxiety disorder | 10041242 |
| Social fear | 10041247 |
| Stress | 10042209 |
| Tension | 10043268 |
| Terminal agitation | 10077416 |
| Thanatophobia | 10064723 |
| Thermophobia | 10075147 |
| Trichotemnomania | 10072752 |
| Trichotillomania | 10044629 |

# 13.9.12. Sleep Disorders

Medical concept of sleep disorders. All preferred terms from (1) HLGT 'Sleep Disorders and Disturbances', 'Psychiatric disorders' SOC plus (2) HLGT 'Sleep disturbances (incl subtypes)', 'Nervous system' SOC. Numerous duplicated preferred terms e.g. middle insomnia.

| HLGT Sleep Disorders and Disturbances, HLGT Code 10040991 | |
|-----------------------------------------------------------|----------|
| Preferred Term | PT Code |
| Abnormal dreams | 10000125 |
| Abnormal sleep-related event | 10061613 |
| Advanced sleep phase | 10001423 |
| Behavioural induced insufficient sleep syndrome | 10081938 |
| Behavioural insomnia of childhood | 10072072 |
| Breathing-related sleep disorder | 10006344 |
| Cataplexy | 10007737 |
| Circadian rhythm sleep disorder | 10009191 |
| Confusional arousal | 10067494 |
| Delayed sleep phase | 10012209 |
| Dyssomnia | 10061827 |
| Exploding head syndrome | 10080684 |
| Hypersomnia | 10020765 |
| Hypersomnia related to another mental condition | 10020767 |
| Hypersomnia-bulimia syndrome | 10053712 |
| Hypnagogic hallucination | 10020927 |
| Hypnopompic hallucination | 10020928 |
| Hyposomnia | 10067530 |
| Initial insomnia | 10022035 |
| Insomnia | 10022437 |
| Insomnia related to another mental condition | 10022443 |
| Irregular sleep phase | 10022995 |
| Irregular sleep wake rhythm disorder | 10080301 |

| HLGT Sleep Disorders and Disturbances, HLGT Code 10040991 | |
|-------------------------------------------------------------------|----------|
| Loss of dreaming | 10065085 |
| Middle insomnia | 10027590 |
| Narcolepsy | 10028713 |
| Nightmare | 10029412 |
| Non-24-hour sleep-wake disorder | 10078086 |
| Parasomnia | 10061910 |
| Paradoxical insomnia | 10083337 |
| Periodic limb movement disorder | 10064600 |
| Pickwickian syndrome | 10035004 |
| Poor quality sleep | 10062519 |
| Rapid eye movement sleep behaviour disorder | 10077299 |
| Rapid eye movements sleep abnormal | 10037841 |
| Shift work disorder | 10078088 |
| Sleep apnoea syndrome | 10040979 |
| Sleep attacks | 10040981 |
| Sleep disorder | 10040984 |
| Sleep disorder due to a general medical condition | 10063910 |
| Sleep disorder due to general medical condition, hypersomnia type | 10040985 |
| Sleep disorder due to general medical condition, insomnia type | 10040986 |
| Sleep disorder due to general medical condition, mixed type | 10040987 |
| Sleep disorder due to general medical condition, parasomnia type | 10040988 |
| Sleep inertia | 10067493 |
| Sleep paralysis | 10041002 |
| Sleep sex | 10067492 |
| Sleep talking | 10041009 |
| Sleep terror | 10041010 |
| Sleep-related eating disorder | 10067315 |
| Somnambulism | 10041347 |

| HLGT Sleep Disorders and Disturbances, HLGT Code 10040991 | |
|-------------------------------------------------------------|----------|
| Somnolence | 10041349 |
| Somnolence neonatal | 10041350 |
| Sopor | 10058709 |
| Stupor | 10042264 |
| Terminal insomnia | 10068932 |
| Upper airway resistance syndrome | 10063968 |
| HLGT Sleep disturbances (incl subtypes), HLGT code 10040998 | |
| Abnormal dreams | 10000125 |
| Abnormal sleep-related event | 10061613 |
| Advanced sleep phase | 10001423 |
| Behavioural induced insufficient sleep syndrome | 10081938 |
| Behavioural insomnia of childhood | 10072072 |
| Breathing-related sleep disorder | 10006344 |
| Cataplexy | 10007737 |
| Central-alveolar hypoventilation | 10007982 |
| Circadian rhythm sleep disorder | 10009191 |
| Confusional arousal | 10067494 |
| Delayed sleep phase | 10012209 |
| Dyssomnia | 10061827 |
| Fatal familial insomnia | 10072077 |
| Hypersomnia | 10020765 |
| Hyposomnia | 10067530 |
| Initial insomnia | 10022035 |
| Insomnia | 10022437 |
| Irregular sleep phase | 10022995 |
| Irregular sleep wake rhythm disorder | 10080301 |
| Loss of dreaming | 10065085 |
| Microsleep | 10076954 |

| HLGT Sleep Disorders and Disturbances, HLGT Code 10040991 | |
|-----------------------------------------------------------|----------|
| Middle insomnia | 10027590 |
| Narcolepsy | 10028713 |
| Non-24-hour sleep-wake disorder | 10078086 |
| Periodic limb movement disorder | 10064600 |
| Pickwickian syndrome | 10035004 |
| Poor quality sleep | 10062519 |
| Rapid eye movement sleep behaviour disorder | 10077299 |
| Rapid eye movements sleep abnormal | 10037841 |
| Shift work disorder | 10078088 |
| Sleep apnoea syndrome | 10040979 |
| Sleep deficit | 10080881 |
| Sleep inertia | 10067493 |
| Sleep paralysis | 10041002 |
| Sleep sex | 10067492 |
| Sleep talking | 10041009 |
| Sleep terror | 10041010 |
| Sleep-related eating disorder | 10067315 |
| Somnambulism | 10041347 |
| Sudden onset of sleep | 10050014 |
| Terminal insomnia | 10068932 |
| Upper airway resistance syndrome | 10063968 |

#### 13.9.14. Seizures

Medical concept of seizures. Only narrow terms from SMQ 'Convulsions' selected plus selected PTs of possible seizure events from HLT 'Disturbances in consciousness NEC' under SOC 'Nervous systems disorders' and HLT 'Confusion and disorientation' under SOC 'Psychiatric disorders'.

| SMQ: 'Convulsions' | |
|-----------------------------------------------------------------|----------|
| SMQ Code: 20000079<br>Category: A | |
| Scope: Narrow | |
| Preferred Term | PT Code |
| 1p36 deletion syndrome | 10082398 |
| 2-Hydroxyglutaric aciduria | 10078971 |
| Acquired epileptic aphasia | 10052075 |
| Acute encephalitis with refractory, repetitive partial seizures | 10076948 |
| Alcoholic seizure | 10056347 |
| Alpers disease | 10083857 |
| Aspartate-glutamate-transporter deficiency | 10079140 |
| Atonic seizures | 10003628 |
| Atypical benign partial epilepsy | 10056699 |
| Automatism epileptic | 10003831 |
| Autonomic seizure | 10049612 |
| Baltic myoclonic epilepsy | 10054895 |
| Benign familial neonatal convulsions | 10067866 |
| Benign rolandic epilepsy | 10070530 |
| Biotinidase deficiency | 10071434 |
| CEC syndrome | 10083749 |
| CDKL5 deficiency disorder | 10083005 |
| Change in seizure presentation | 10075606 |
| Clonic convulsion | 10053398 |
| Congenital bilateral perisylvian syndrome | 10082716 |
| Convulsion in childhood | 10052391 |
| Convulsions local | 10010920 |
| Convulsive threshold lowered | 10010927 |
| CSWS syndrome | 10078827 |
| Deja vu | 10012177 |

| SMQ: 'Convulsions'<br>SMQ Code: 20000079 | |
|-----------------------------------------------------------------|----------|
| Category: A | |
| Scope: Narrow | |
| Double cortex syndrome | 10073490 |
| Dreamy state | 10013634 |
| Drug withdrawal convulsions | 10013752 |
| Early infantile epileptic encephalopathy with burst-suppression | 10071545 |
| Eclampsia | 10014129 |
| Epilepsy | 10015037 |
| Epilepsy surgery | 10079824 |
| Epilepsy with myoclonic-atonic seizures | 10081179 |
| Epileptic aura | 10015049 |
| Epileptic psychosis | 10059232 |
| Faciobrachial dystonic seizure | 10084187 |
| Febrile convulsion | 10016284 |
| Febrile infection-related epilepsy syndrome | 10079438 |
| Focal dyscognitive seizures | 10079424 |
| Frontal lobe epilepsy | 10049424 |
| Gelastic seizure | 10082918 |
| Generalised onset non-motor seizure | 10083376 |
| Generalised tonic-clonic seizure | 10018100 |
| Glucose transporter type 1 deficiency syndrome | 10078727 |
| GM2 gangliosidosis | 10083933 |
| Grey matter heterotopia | 10082084 |
| Hemimegalencephaly | 10078100 |
| Hyperglycaemic seizure | 10071394 |
| Hypocalcaemic seizure | 10072456 |
| Hypoglycaemic seizure | 10048803 |
| Hyponatraemic seizure | 10073183 |

| SMQ: 'Convulsions'<br>SMQ Code: 20000079<br>Category: A<br>Scope: Narrow | |
|---|---|
| Idiopathic generalised epilepsy | 10071081 |
| Infantile spasms | 10021750 |
| Jeavons syndrome | 10084303 |
| Juvenile myoclonic epilepsy | 10071082 |
| Lafora's myoclonic epilepsy | 10054030 |
| Lennox-Gastaut syndrome | 10048816 |
| Migraine-triggered seizure | 10076676 |
| Molybdenum cofactor deficiency | 10069687 |
| Multiple subpial transection | 10079825 |
| Myoclonic epilepsy | 10054859 |
| Myoclonic epilepsy and ragged-red fibres | 10069825 |
| Neonatal epileptic seizure | 10082068 |
| Neonatal seizure | 10082067 |
| Partial seizures | 10061334 |
| Partial seizures with secondary generalisation | 10056209 |
| Petit mal epilepsy | 10034759 |
| Polymicrogyria | 10073489 |
| Post stroke epilepsy | 10076982 |
| Post stroke seizure | 10076981 |
| Postictal headache | 10052470 |
| Postictal paralysis | 10052469 |
| Postictal psychosis | 10070669 |
| Postictal state | 10048727 |
| Post-traumatic epilepsy | 10036312 |
| Schizencephaly | 10073487 |
| Seizure | 10039906 |

| SMQ: 'Convulsions' SMQ Code: 20000079 Category: A Scope: Narrow | |
|---|---|
| Seizure anoxic | 10039907 |
| Seizure cluster | 10071350 |
| Seizure like phenomena | 10071048 |
| Severe myoclonic epilepsy of infancy | 10073677 |
| Simple partial seizures | 10040703 |
| Status epilepticus | 10041962 |
| Sudden unexplained death in epilepsy | 10063894 |
| Temporal lobe epilepsy | 10043209 |
| Tonic clonic movements | 10051171 |
| Tonic convulsion | 10043994 |
| Tonic posturing | 10075125 |
| Topectomy | 10073488 |
| Transient epileptic amnesia | 10081728 |
| Tuberous sclerosis complex | 10080584 |
| Uncinate fits | 10045476 |
| Additional selected preferred terms from HLT Disturbances in consciousness NEC, HLT code 10013509 and HLT Confusion and disorientation, HLT code 10010301. | |
| Preferred Term | PT Code |
| Confusional state | 10010305 |
| Loss of consciousness | 10024855 |
| Syncope | 10042772 |
| Sopor | 10058709 |
| Stupor | 10042264 |
| Altered state of consciousness | 10050093 |
| Depressed level of consciousness | 10012373 |
| Consciousness fluctuating | 10050093 |

# 13.9.15. Weight Gain

Medical concept of weight gain. Selected PTs from HLT 'General nutritional disorders NEC', under SOC 'Metabolism and nutrition disorders', and HLT 'Physical examination procedures and organ system status', under SOC 'Investigations' and HLT 'General signs and symptoms NEC', under SOC 'General disorders and administration site conditions'.

| PTs (Select) from HLT General nutritional disorders NEC, HLT code 10018067 | |
|---|---|
| Preferred Term | PT Code |
| Abdominal fat apron | 10077983 |
| Overweight | 10033307 |
| Abnormal weight gain | 10000188 |
| Central obesity | 10065941 |
| Obesity | 10029883 |
| Abdominal fat apron | 10077983 |
| Overweight | 10033307 |
| Abnormal weight gain | 10000188 |
| Central obesity | 10065941 |
| Obesity | 10029883 |
| PTs (Select) from HLT Physical examination procedures and organ system status, HLT Code 10071941 | |
| Preferred Term | PT Code |
| Weight abnormal | 10056814 |
| Weight increased | 10047899 |
| Waist circumference increased | 10064863 |
| Body mass index abnormal | 10074506 |
| Body mass index increased | 10005897 |
| PTs (Select) from HLT General signs and symptoms NEC, HLT Code 10018072 | |
| Preferred Term | PT Code |
| Fat tissue increased | 10016251 |
| Sarcopenic obesity | 10083992 |

# 13.9.16. Rhabdomyolysis

Medical concept of rhabdomyolysis. Only narrow terms only for SMQ 'Rhabdomyolysis/myopathy' plus 2 additional preferred terms selected from HGLT 'muscle disorders' under SOC 'Musculoskeletal and connective tissue disorders'.

| SMQ: 'Rhabdomyolysis/myopathy' SMQ Code: 20000002 Category: A Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Muscle necrosis | 10028320 |
| Myoglobin blood increased | 10028625 |
| Myoglobin blood present | 10059888 |
| Myoglobin urine present | 10028631 |
| Myoglobinaemia | 10058735 |
| Myoglobinuria | 10028629 |
| Myopathy | 10028641 |
| Myopathy toxic | 10028648 |
| Necrotising myositis | 10074769 |
| Rhabdomyolysis | 10039020 |
| Thyrotoxic myopathy | 10081524 |
| PTs (Select) from HGLT muscle disorders, HLGT Code 10028302 | |
| Preferred Term | PT Code |
| Myalgia | 10028411 |
| Myositis | 10028653 |

#### 13.9.17. Pancreatitis

Medical concept of acute pancreatitis. Only narrow terms of SMQ 'Acute pancreatitis' selected. Algorithmic approach for this SMQ not used due to complexity in applying and poor specificity of remaining categories. Category A selected as PTs because more specific for concept (only narrow terms).

| SMQ: 'Acute pancreatitis' | |
|------------------------------------|----------|
| SMQ Code: 20000022 | |
| Category: A Scope: Narrow | |
| Preferred Term | PT Code |
| Cullen's sign | 10059029 |
| Grey Turner's sign | 10075426 |
| Haemorrhagic necrotic pancreatitis | 10076058 |
| Hereditary pancreatitis | 10056976 |
| Immune-mediated pancreatitis | 10083072 |
| Ischaemic pancreatitis | 10066127 |
| Oedematous pancreatitis | 10052400 |
| Pancreatic abscess | 10048984 |
| Pancreatic cyst drainage | 10082531 |
| Pancreatic haemorrhage | 10033625 |
| Pancreatic necrosis | 10058096 |
| Pancreatic phlegmon | 10056975 |
| Pancreatic pseudoaneurysm | 10081762 |
| Pancreatic pseudocyst | 10033635 |
| Pancreatic pseudocyst drainage | 10033636 |
| Pancreatic pseudocyst haemorrhage | 10083813 |
| Pancreatic pseudocyst rupture | 10083811 |
| Pancreatitis | 10033645 |
| Pancreatitis acute | 10033647 |
| Pancreatitis haemorrhagic | 10033650 |
| Pancreatitis necrotising | 10033654 |
| Pancreatitis relapsing | 10033657 |
| Pancreatorenal syndrome | 10056277 |
| Subacute pancreatitis | 10084554 |

# 13.9.18. Impact on Creatinine

Medical concept of worsening renal function/renal failure in the context of impact on creatinine. Only narrow terms from SMQ 'Acute renal failure' plus all PTs from HLT 'Renal failure and impairment', under SOC 'Renal and urinary disorders'. Numerous duplicated preferred terms e.g. renal failure

| SMQ: 'Acute renal failure'<br>SMQ Code: 20000003<br>Category: A<br>Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Acute kidney injury | 10069339 |
| Acute phosphate nephropathy | 10069688 |
| Anuria | 10002847 |
| Azotaemia | 10003885 |
| Continuous haemodiafiltration | 10066338 |
| Dialysis | 10061105 |
| Foetal renal impairment | 10078987 |
| Haemodialysis | 10018875 |
| Haemofiltration | 10053090 |
| Neonatal anuria | 10049778 |
| Nephropathy toxic | 10029155 |
| Oliguria | 10030302 |
| Peritoneal dialysis | 10034660 |
| Prerenal failure | 10072370 |
| Renal failure | 10038435 |
| Renal failure neonatal | 10038447 |
| Renal impairment | 10062237 |
| Renal impairment neonatal | 10049776 |
| Subacute kidney injury | 10081980 |

| Renal Failure and Impairment HLT, HLT Code 100384 | 43 |
|---------------------------------------------------|----------|
| Preferred Term | PT Code |
| Acute Kidney injury | 10069339 |
| Anuria | 10002847 |
| Atypical haemolytic uraemic syndrome | 10079840 |
| Cardiorenal syndrome | 10068230 |
| Chronic kidney disease | 10064848 |
| Crush syndrome | 10050702 |
| Diabetic end stage renal disease | 10012660 |
| End stage renal disease | 10077512 |
| Foetal renal impairment | 10078987 |
| Haemolytic uraemic syndrome | 10018932 |
| Hepatorenal failure | 10019845 |
| Hepatorenal syndrome | 10019846 |
| Nail-patella syndrome | 10063431 |
| Neonatal anuria | 10049778 |
| Oliguria | 10030302 |
| Pancreatorenal syndrome | 10056277 |
| Postoperative renal failure | 10056675 |
| Postrenal failure | 10059345 |
| Prerenal failure | 10072370 |
| Propofol infusion syndrome | 10063181 |
| Renal failure | 10038435 |
| Renal failure neonatal | 10038447 |
| Renal impairment | 10062237 |
| Renal impairment neonatal | 10049776 |
| Renal injury | 10061481 |
| Scleroderma renal crisis | 10062553 |
| Traumatic anuria | 10044501 |

# 13.9.19. Safety During Pregnancy

Use AE terms co-reported in pregnancy exposures to CAB.

# 13.10. Appendix 10: Identification of COVID-19 Adverse Events

COVID-19 adverse events are identified based on MedDRA coded values and/or AE referenced in the COVID-19 Coronavirus Infection assessment. The Lowest Level Terms (LLTs) and codes, Preferred Terms (PTs), High Level Terms (HLTs), High Level Group Terms (HLGTs), and System Organ Classes (SOCs), below are from MedDRA 23.0. In case there is a change to the version of MedDRA at time of reporting, the coded values based on the MedDRA version at the time of reporting will be used. The additional events may also be added based on the blinded review of AE data collected on study prior to the database freeze.

SOC: Infections and infestations

| LLT | | | | |
|---|---|---|---|---|
| code | LLT | PT | HLT | HLGT |
| | | | | Viral |
| 1008445 | | Asymptomati | Coronaviru | infectious |
| 9 | Asymptomatic COVID-19 | c COVID-19 | s infections | disorders |
| | | | | Viral |
| 1008446 | | Asymptomati | Coronaviru | infectious |
| 7 | Asymptomatic SARS-CoV-2 infection | c COVID-19 | s infections | disorders |
| | | | | Viral |
| 1005398 | | Coronavirus | Coronaviru | infectious |
| 3 | Corona virus infection | infection | s infections | disorders |
| | | | | Viral |
| 1005190 | | Coronavirus | Coronaviru | infectious |
| 5 | Coronavirus infection | infection | s infections | disorders |
| | | | | Viral |
| 1008438 | | | Coronaviru | infectious |
| 2 | Coronavirus disease 2019 | COVID-19 | s infections | disorders |
| | | | Virus | Microbiology |
| 1007025 | | | identificatio | and serology |
| 5 | | Coronavirus | n and | investigation |
| | Coronavirus test positive | test positive | serology | S |
| | | | | Therapeutic |
| | | | | procedures |
| 1008446 | | | | and |
| 0 | | COVID-19 | Antiinfectiv | supportive |
| | COVID-19 treatment | treatment | e therapies | care NEC |
| 1008463 | | | | Viral |
| 9 | | SARS-CoV-2 | Coronaviru | infectious |
| | SARS-CoV-2 sepsis | sepsis | s infections | disorders |
| | | | Virus | Microbiology |
| 1008427 | | | identificatio | and serology |
| 1 | | SARS-CoV-2 | n and | investigation |
| | SARS-CoV-2 test positive | test positive | serology | S |

| LLT | | DT | | 0.7 |
|---|---|---|---|---|
| code | LLT | PT | HLT | HLGT |
| 1008464 | | 04000 1/0 | | Viral |
| 0 | CARC Cal/ 2 vina amaia | SARS CoV-2 | Coronaviru | infectious |
| | SARS CoV-2 viraemia | viraemia | s infections | disorders |
| 1008426 | | | Caranaviru | Viral |
| 8 | COVID-19 | COVID-19 | Coronaviru s infections | infectious<br>disorders |
| 0 | COVID-19 | COVID-19 | SIMECTIONS | Viral |
| 1008440 | | | Coronaviru | infectious |
| 1000440 | COVID-19 respiratory infection | COVID-19 | s infections | disorders |
| I | COVID-19 respiratory infection | COVID-19 | 5 II II ECLIONS | Viral |
| 1008427 | SARS-CoV-2 acute respiratory | | Coronaviru | infectious |
| 0 | disease | COVID-19 | s infections | disorders |
| | diocaso | OOVID 10 | o imodiono | Viral |
| 1008427 | | | Coronaviru | infectious |
| 2 | SARS-CoV-2 infection | COVID-19 | s infections | disorders |
| | | | | Viral |
| 1008438 | | COVID-19 | Coronaviru | infectious |
| 1 | Coronavirus pneumonia | pneumonia | s infections | disorders |
| | | | | Viral |
| 1008438 | | COVID-19 | Coronaviru | infectious |
| 0 | COVID-19 pneumonia | pneumonia | s infections | disorders |
| | | | | Viral |
| 1008438 | | COVID-19 | Coronaviru | infectious |
| 3 | Novel COVID-19-infected pneumonia | pneumonia | s infections | disorders |
| | | | | Viral |
| 1008445 | | Suspected | Coronaviru | infectious |
| 1 | Suspected COVID-19 | COVID-19 | s infections | disorders |
| 4000445 | | | | Viral |
| 1008445 | 0 | Suspected | Coronaviru | infectious |
| 2 | Suspected SARS-CoV-2 infection | COVID-19 | s infections | disorders |
| 1000110 | | 0400 0-1/0 | Infectious | Ancillary |
| 1008446 | CARC Cal/ 2 comics | SARS-CoV-2 | disorders | infectious |
| 1 | SARS-CoV-2 carrier | carrier | carrier | topics |

# 13.11. Appendix 11: Abbreviations & Trade Marks

# 13.11.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| A&R | Analysis and Reporting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library (GSK Standards Library) |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| MMRM | Mixed Model Repeated Measures |
| PBMC | Peripheral Blood Mononuclear Cells |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PopPK | Population PK |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| SAC | Statistical Analysis Complete |

| Abbreviation | Description |
|--------------|---------------------------------|
| SDSP | Study Data Standardization Plan |
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |

# 13.11.2. Trademarks

| Trademarks of the GlaxoSmithKline Group of Companies |
|------------------------------------------------------|
| Cabotegravir |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| Rilpivirine |
| SAS |

## 13.12. Appendix 12: List of Data Displays

All data displays will use the term "subject" rather than "participant" in accordance with CDSIC and GSK Statistical Display Standards.

Where applicable, all summary displays will present data across both the Intervention and Extension phases unless explicitly stated otherwise in the display title.

At EOS, the RAPIDO Data Viewer will be produced to allow for the clinical team to review ADaM data directly related to adverse events, exposure, HIV-1 RNA, and labs. This will take the place of some, previously standard generic listings from these categories. Listings including results of pregnancy details will only be included if a pregnancy occurs.

#### 13.12.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|------------|
| Study Population | 1.1 to 1.27 | |
| Efficacy | 2.1 to 2.16 | 2.1 to 2.4 |
| Safety | 3.1 to 3.75 | 3.1 to 3.4 |
| Other | 4.1 to 4.4 | |
| Section | List | ings |
| ICH Listings | 1 to | 24 |
| Other Listings | 25 t | o 57 |

#### 13.12.2. Mock Example Shell Referencing

Nonstandard specifications will be referenced as indicated below (where a study specific mock shell is available) or the location of a similar display produced for a different study in the HARP reporting environment will be provided as reference. If required example mock-up displays provided in <u>Appendix 13</u>: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------|--------|--------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAF_Fn | SAF_Tn | SAF_Ln |
| Other | OTR_Tn | OTR_Fn | OTR_Ln |

#### 13.12.3. Deliverables

| Delivery | Description |
|---|---|
| IA1 | Interim Analysis Statistical Analysis Complete at IA (Month 4) when 50% of subjects have received their 3 <sup>rd</sup> injection. |
| IA2 | Interim Analysis Statistical Analysis Complete at IA (Month 4) when 100% of subjects have received their 3 <sup>rd</sup> injection. |


| Delivery | Description |
|----------|-------------------------------------------|
| HL | Headline at Month 12 |
| M12 | Statistical Analysis Complete at Month 12 |
| EOS | End of Study |
## 13.12.4. Study Population Tables

| Stud | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard /<br>Example Shell | Title | Programming Notes | Deliverable |
| Subje | ect Disposition | | | | |
| 1.1. | Safety | ES1 | Summary of Subject Disposition for the Subject Conclusion Record | ICH E3, FDAAA, EudraCT | HL, M12,<br>EOS |
| 1.2. | Safety | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | ICH E3 | M12, EOS |
| 1.3. | Safety | DISP_T1 | Summary of Subject Disposition at Each Study Phase | ICH E3 Intervention/Extension phase: status and reason for withdrawal based on date and reason collected in the study treatment discontinuation form. Long term Follow-up: completion/withdrawal based on data collected in the Study Conclusion form. For the Intervention Phase, columns should report OLI results, LA results, & Total results; All other phases only list total results Under withdrawals, add subcategory for Covid-19 | M12, EOS |

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard /<br>Example Shell | Title | Programming Notes | Deliverable |
| 1.4. | Safety | DISP_T2 | Summary of Reason for Withdrawal at Each Study Phase | FDAAA, EudraCT For Intervention Phase, columns should report OLI results, LA results, & Total results; All other phases only list total results | IA2, HL, M12,<br>EOS |
| | | | | See mockup for relevant Covid-19 Subcategories | |
| 1.5. | Safety | ES11 | Summary of Outcome of Adverse Events Which Led to Study Withdrawal/Treatment Discontinuation at Each Study Phase | EudraCT | M12, EOS |
| 1.6. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements | M12 |
| 1.7. | Enrolled | NS1 | Summary of Number of Subjects by Country and Site ID | EudraCT/Clinical Operations | IA1, HL, M12 |
| Proto | col Deviation | | | | |
| 1.8. | Enrolled | DV1 | Summary of Important Protocol Deviations | ICH E3 | M12, EOS |
| 1.9. | Enrolled | DV1 | Summary of Important COVID-19 Related Protocol Deviations | Update the label for the first row to<br>be "ANY IMPORTANT COVID-19<br>RELATED PROTOCOL<br>DEVIATIONS" | M12, EOS |
| 1.10. | Enrolled | DV1 | Summary of Important Non-COVID-19 Protocol Deviations | Update the label for the first row to be "ANY IMPORTANT NON-COVID-19 RELATED PROTOCOL DEVIATIONS" | M12, EOS |
| 1.11. | Enrolled | DV1 | Summary of COVID-19 Protocol Deviations by Site | Update the label for the first row to be "ANY COVID-19 RELATED PROTOCOL DEVIATIONS". Summary for each site and 'Total' across sites. | IA2, HL, M12,<br>EOS |

| Study | Population Ta | bles | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard /<br>Example Shell | Title | Programming Notes | Deliverable |
| 1.12. | Enrolled | DV1 | Summary of All Implementation Protocol Deviations by Site | Update the label for the first row to be "ANY IMPLEMENTATION RELATED PROTOCOL DEVIATIONS" Summary for each site and 'Total' across sites. | HL, M12,<br>EOS |
| Popu | lation Analysed | j | | | |
| 1.13. | Screened | SP1 | Summary of Study Populations | GSK Statistical Display Standard | M12, EOS |
| 1.14. | Enrolled | SP2 | Summary of Exclusions from the Safety Population | GSK Statistical Display Standard | M12 |
| Demo | graphic and B | aseline Characteristics | | | |
| 1.15. | Safety | DM1 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT Include Baseline CD4+ Cell Count Results and CDC HIV-1 Infection Classification. | IA1, HL, M12 |
| 1.16. | Enrolled | DM11 | Summary of Age Ranges | EudraCT | M12 |
| 1.17. | Safety | DM6 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT | M12 |
| Prior | and Concomita | ant Medications | | | |
| 1.18. | Safety | MH1 | Summary of Past Medical Conditions | ICH E3 | M12 |
| 1.19. | Safety | MH4 | Summary of Past Cardiac, Gastrointestinal, Metabolism and Nutrition, Psychiatric, Renal and Urinary, Nervous System Conditions, and Hepatobiliary Disorders | ICH E3 | M12 |
| 1.20. | Safety | MH1 | Summary of Current Medical Conditions | ICH E3 | M12 |
| 1.21. | Safety | MH4 | Summary of Current Cardiac, Gastrointestinal, Metabolism and Nutrition, Psychiatric, Renal and Urinary, Nervous System Conditions, and Hepatobiliary Disorders | ICH E3 | M12 |

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard /<br>Example Shell | Title | Programming Notes | Deliverable |
| 1.22. | Safety | СМ9 | Summary of Concomitant Medications by Ingredient Combinations | ICH E3 See GSK Statistical Display Standard Multi-ingredient medications will be labelled according to the sum of their ingredients, i.e., Generic Term. | M12, EOS |
| 1.23. | Safety | 207966/primary_15/T1.30 | Summary of Prior Antiretroviral Therapy Taken during Screening | Remove the footnote. Follow definitions in Section 13.3.1 to determine the prior ART medications. | M12 |
| 1.24. | Safety | RF1 | Summary of HIV Risk Factors | | M12 |
| 1.25. | Safety | 201585/primary_02/T1.31 | Time Since First Antiretroviral Therapy Until Intervention Phase Start | Add footnote "Note: Duration is calculated as the day prior to first dose of CAB+RPV – the first recorded date of prior ART usage +1." | M12 |
| 1.26. | Safety | DM1 | Summary of Categorical Baseline BMI | | M12 |
| 1.27. | Safety | DM1 | Summary of Baseline BMI Based on Day 1 Weight Values | Repeat the descriptive BMI statistics from Table 1.15 and the categorical statistics from Table 1.26 using a newly calculated Baseline BMI based on Day 1 weight values instead of CRF reported BMI values. | EOS |

# 13.12.5. Efficacy Tables

| Effica | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/<br>Example Shell | Title | Programming Notes | Deliverable |
| Snap | shot | | | | |
| 2.1. | Safety | EFF_T1 | Summary of Study Outcomes (50 c/mL cutoff) at Month 12 (Intervention Phase) –Snapshot Analysis | | HL, M12 |
| 2.2. | Safety | EFF_T2 | Summary of Study Outcomes (50 c/mL cutoff) at Month 12 (Intervention Phase) –Snapshot Analysis Considering Covid-19 Based Events | With expanded COVID-19 related/Non-related categories | HL, M12 |
| 2.3. | Safety | SNAPSHOT4 | Proportion of Subjects with Plasma HIV-1 RNA ≥ 50 c/mL<br>Over Time (Intervention Phase) –Snapshot Analysis | Use Exact (Clopper-Pearson) method for 95% confidence Intervals. Expand to all visits, drop 'n' row, replace x (%) column data with x/n (%), drop '(Intervention Phase)' and use Observed Case instead of Snapshot for EOS | M12, EOS |
| 2.4. | Safety | SNAPSHOT4 | Proportion of Subjects with Plasma HIV-1 RNA < 50 c/mL<br>Over Time (Intervention Phase) –Snapshot Analysis | Use Exact (Clopper-Pearson) method for 95% confidence Intervals. Expand to all visits, drop 'n' row, replace x (%) column data with x/n (%), drop '(Intervention Phase)' and use Observed Case instead of Snapshot for EOS | M12, EOS |
| 2.5. | Safety | SNAPSHOT4 | Proportion of Subjects with Plasma HIV-1 RNA ≥ 50 c/mL<br>Over Time by Subgroup (Intervention Phase) –Snapshot<br>Analysis | Include the following subgroups: country, implementation arm, sex, age group, race group, and CD4 group as mentioned in Section 5.4.2. | M12 |

| Effica | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.6. | Safety | SNAPSHOT4 | Proportion of Subjects with Plasma HIV-1 RNA < 50 c/mL<br>Over Time by Subgroup (Intervention Phase) –Snapshot<br>Analysis | Include the following subgroups: country, implementation arm, sex, age group, race group, and CD4 group as mentioned in Section 5.4.2. | M12 |
| CVF | | | | | |
| 2.7. | Safety | VF1 | Cumulative Proportion of Subjects Meeting Confirmed Virologic Failure Criteria Over Time (Intervention Phase) | | HL, M12 |
| 2.8. | Safety | VF2 | Proportion of Subjects Meeting Confirmed Virologic Failure Criteria Over Time | | M12, EOS |
| Geno | type & Pheno | type | | | |
| 2.9. | Safety | 201584/primary_17/T7.1 | Summary of the Prevalence of Treatment-Emergent Major<br>Resistance Mutations of INI, NRTI, NNRTI and PI Class at<br>time of CVF - Plasma Sample | Known resistance mutations per Section 13.5.5. Include 95% confidence Intervals using Exact (Clopper-Pearson) method. | HL, M12,<br>EOS |
| 2.10. | Safety | 201584/primary_17/T7.2 | Summary of Viral load, Genotypic and Phenotypic data for Subjects Who Met Confirmed Virologic Failure Criteria | | M12, EOS |
| 2.11. | Safety | 201584/primary_17/T7.4 | Summary of Viral load, Genotypic and Phenotypic data for Subjects Who Did Not Meet Confirmed Virologic Failure Criteria | Only include subjects with available genotypic or phenotypic data. | M12, EOS |
| CD4 | | | | | |
| 2.12. | Safety | LB1 | Summary of CD4+ Cell Count (cells/mm^3) by Visit | | M12, EOS |
| 2.13. | Safety | LB1 | Summary of Change from Baseline in CD4+ Cell Count (cells/mm^3) by Visit | | M12, EOS |

| Effica | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.14. | Safety | LB1 | Summary of CD4+/CD8+ Ratio Cell Count (cells/mm^3) at Baseline & Month 12 | | M12 |
| HIV A | ssociated Co | nditions | | | |
| 2.15. | Safety | CDC2 | Summary of Post-Baseline CDC Stage 3 HIV-1 Associated Conditions Including Recurrences | | M12, EOS |
| 2.16. | Safety | CDC2 | Summary of Post-Baseline CDC Stage 3 HIV-1 Associated Conditions Excluding Recurrences | | M12, EOS |

## 13.12.6. Efficacy Figures

| Efficacy: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard<br>/ Example<br>Shell | Title | Programming Notes | Deliverable |
| Snapsh | not | | | | |
| 2.1. | Safety | SNAPSHOT8 | Percent (95% CI) of Subjects with Plasma HIV-1 RNA ≥ 50 copies/mL Over Time (Intervention Phase) –Snapshot Analysis | Use Exact (Clopper-Pearson) method for 95% confidence Intervals. Drop '(Intervention Phase)', Observed cases to be used at EOS instead of Snapshot | M12, EOS |
| 2.2. | Safety | SNAPSHOT8 | Percent (95% CI) of Subjects with Plasma HIV-1 RNA < 50 copies/mL Over Time (Intervention Phase) –Snapshot Analysis | Use Exact (Clopper-Pearson) method for 95% confidence Intervals. Drop '(Intervention Phase)', Observed cases to be used at EOS instead of Snapshot | M12, EOS |

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| 2.3. | Safety | SNAPSHOT10 | Individual HIV-1 RNA Plasma Profiles by Visit for Subjects with HIV-1 RNA >= 50 copies/mL at Month 12 per Snapshot Algorithm | The 1st vertical line indicates start of study treatment at Intervention Phase. The second vertical reference line indicates last IP on-treatment study day. i.e. min (last IP injection dose+35 days, LTFU HAART start date, date of last oral CAB+RPV+1). This vertical line is only for subjects who withdraw from Intervention Phase/Extension phase. | M12 |
| 2.4. | Safety | SNAPSHOT10 | Individual HIV-1 RNA Plasma Profiles by Visit for Subjects with Confirmed Virologic Failure | Same as Figure 2.3. | M12, EOS |

# 13.12.7. Safety Tables

| Safe | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/ Example Shell | Title | Programming Notes | Deliverable |
| Expo | sure | | | , | |
| 3.1. | Safety | 207966/primary_15/T3.1 | Summary of Exposure to Study Treatment by Implementation Arm (Intervention Phase) | Includes Oral Bridging | IA2, M12 |
| 3.2. | Safety | 207966/primary_15/T3.1 | Summary of Exposure to Study Treatment by Implementation Arm | Includes Oral Bridging | M12, EOS |
| 3.3. | Safety | <u>SAF T1</u> | Summary of Adherence to CAB LA + RPV LA Dosing Schedule by Visit, Country, and Site (Intervention Phase) | See Section 13.5.2 for Covid Impact Remove Covid-19 impact results from IA1. | IA1, IA2,<br>HL, M12 |
| 3.4. | Safety | <u>SAF_T2</u> | Summary of Adherence to CAB LA + RPV LA Dosing Schedule by Visit and Subgroup (Intervention Phase) | See Section 13.5.2 for Covid Impact Include all subgroups listed in Section 5.4.2 except for Site & Country | HL, M12 |
| 3.5. | Safety | SAF_T1 | Summary of Adherence to CAB LA + RPV LA Dosing Schedule by Visit, Country, and Site | See Section 13.5.2 for Covid Impact | EOS |
| 3.6. | Safety | <u>SAF_T2</u> | Summary of Adherence to CAB LA + RPV LA Dosing Schedule by Visit and Subgroup | See Section 13.5.2 for Covid Impact Include all subgroups listed in Section 5.4.2 except for Site & Country | EOS |

| Safet | y: Tables | | | | |
|---|---|---|---|---|---|
| 3.7. | Safety | Study 201584 (primary_02): Table 3.114 | Summary of Categorized Needle Length and Gauge for CAB Injection | | M12, EOS |
| 3.8. | Safety | Study 201584 (primary_02): Table 3.115 | Summary of Categorized Needle Length and Gauge for RPV Injection | | M12, EOS |
| Adve | rse Events (A | AEs) | | | |
| 3.9. | Safety | AE99 | Adverse Event Overview by Study Phase and Overall | High level summary to include counts of overall AEs, Serious AEs, AEs leading to withdrawal, related AEs, AEs related to Covid-19, AEs related to Covid-19 leading to withdrawal, fatal AEs Overall breakdown to be condensed to Int + Ext phases. | HL, M12,<br>EOS |
| 3.10. | Safety | AE3 | Summary of Adverse Events by Overall Frequency | ICH E3 | M12, EOS |
| 3.11. | Safety | AE5B | Summary of Adverse Events by System Organ Class and Maximum Grade | ICH E3 | HL, M12,<br>EOS |
| 3.12. | Safety | AE5B | Summary of Adverse Events by System Organ Class and Maximum Grade — Excluding Study Drug Injection Site Reactions | | M12, EOS |
| 3.13. | Safety | AE5B | Summary of Adverse Events by System Organ Class and Maximum Grade (Oral Lead-in Period) | | M12 |
| 3.14. | LTFU | AE5B | Summary of Adverse Events by System Organ Class and Maximum Grade (Long Term Follow-up Period) | | M12, EOS |
| 3.15. | Safety | AE3 | Summary of Common (>=5%) Adverse Events by Overall Frequency | ICH E3 | M12, EOS |
| 3.16. | Safety | AE3 | Summary of Common (>=1%) Grade 2-5 Adverse Events by Overall Frequency | ICH E3 | M12, EOS |

| Safet | y: Tables | | | | |
|---|---|---|---|---|---|
| 3.17. | Safety | 201584/primary_7/T3.46 | Summary of Adverse Events by Visit and Maximum Severity – Overall and Common | | HL, M12,<br>EOS |
| 3.18. | Safety | AE3 | Summary Drug-Related Adverse Events by Overall Frequency | ICH E3 | M12, EOS |
| 3.19. | Safety | AE5B | Summary of Drug-Related Adverse Events by System Organ Class and Maximum Grade | ICH E3 | HL, M12,<br>EOS |
| 3.20. | Safety | AE5B | Summary of Drug-Related Adverse Events by System Organ Class and Maximum Grade (Oral Lead-in Period) | ICH E3 | M12 |
| 3.21. | LTFU | AE5B | Summary of Drug-Related Adverse Events by System Organ Class and Maximum Grade (Long Term Follow-up Period) | ICH E3 | M12, EOS |
| 3.22. | Safety | AE5B | Summary of Drug-Related Adverse Events by System Organ Class and Maximum Grade — Excluding Study Drug Injection Site Reactions | | M12, EOS |
| 3.23. | Safety | AE15 | Summary of Common (>=5%) Non-serious Adverse<br>Events by System Organ Class and Preferred Term<br>(Number of Subjects and Occurrences) | FDAAA, EudraCT | M12, EOS |
| 3.24. | Safety | AE3 | Summary of Common (>=1%) Drug-Related Grade 2-5 Adverse Events by Overall Frequency | ICH E3 | M12, EOS |
| 3.25. | Safety | AE3 | Summary of Non-Serious Drug-Related Adverse<br>Events by Overall Frequency | Plain Language Summary requirements. | M12, EOS |
| 3.26. | Safety | 201584/primary_7/T3.46 | Summary of Drug-Related Adverse Events by Visit and Maximum Severity – Overall and Common | | M12, EOS |
| Serio | us and Other | r Significant Adverse Events | | | |
| 3.27. | Safety | AE5B | Summary of Serious Adverse Events by System Organ Class and Maximum Grade | ICH E3 | HL, M12,<br>EOS |

| Safet | y: Tables | | | | |
|---|---|---|---|---|---|
| 3.28. | Safety | AE5B | Summary of Serious Adverse Events by System Organ Class and Maximum Grade (Oral Lead-in Period) | ICH E3 | M12 |
| 3.29. | LTFU | AE5B | Summary of Serious Adverse Events by System<br>Organ Class and Maximum Grade (Long Term Follow-up Period) | ICH E3 | M12, EOS |
| 3.30. | Safety | AE16 | Summary of Serious Adverse Events by System<br>Organ Class and Preferred Term (Number of Subjects<br>and Occurrences) | FDAAA, EudraCT | M12, EOS |
| 3.31. | Safety | 201584/primary_7/T3.46 | Summary of Serious Adverse Events by Visit and Maximum Severity – Overall and Common | | M12, EOS |
| 3.32. | Safety | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term | GSK Statistical Display Standard | HL, M12,<br>EOS |
| 3.33. | Safety | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term (Oral Lead-in Period) | GSK Statistical Display Standard | M12 |
| 3.34. | LTFU | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term (Long Term Follow-up Period) | GSK Statistical Display Standard | M12, EOS |
| 3.35. | Safety | 201584/primary_7/T3.46 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by Visit and Maximum Severity – Overall and Common | | M12, EOS |

| Safet | | | | | |
|---|---|---|---|---|---|
| Salet | y: Tables | | | | |
| 3.36. | Safety | AE1 | Summary of Serious Adverse Events Leading to<br>Permanent Discontinuation of Study Treatment or<br>Withdrawal from Study by System Organ Class and<br>Preferred Term | GSK Statistical Display Standard | M12, EOS |
| Labo | ratory: Chemi | istry | | | Laboratory: Chemistry |
| 3.40. | Safety | | | | |
| | Salety | LB1 | Summary of Chemistry Changes from Baseline | ICH E3 | M12, EOS |
| 3.41. | LTFU | LB1 | Summary of Chemistry Changes from Baseline Summary of Chemistry Changes from Baseline (Long Term Follow-up Population) | ICH E3 | M12, EOS<br>M12, EOS |
| 3.41. | <del>'</del> | | Summary of Chemistry Changes from Baseline (Long | | |
| 3.42. | LTFU | LB1 | Summary of Chemistry Changes from Baseline (Long Term Follow-up Population) Summary of Chemistry Results by Maximum Grade | ICH E3 | M12, EOS<br>HL, M12, |
| 3.42. | LTFU<br>Safety | LB1 | Summary of Chemistry Changes from Baseline (Long Term Follow-up Population) Summary of Chemistry Results by Maximum Grade | ICH E3 | M12, EOS<br>HL, M12, |
| 3.42.<br><b>Labo</b> | LTFU Safety ratory: Hemat | LB1<br>LB16 | Summary of Chemistry Changes from Baseline (Long Term Follow-up Population) Summary of Chemistry Results by Maximum Grade Increase Post-Baseline Relative to Baseline | ICH E3 ICH E3 Includes pre-specified parameters | M12, EOS<br>HL, M12,<br>EOS |

Laboratory: Hepatobiliary (Liver)

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| 3.46. | Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting | GSK Statistical Display Standard | M12, EOS |
| 3.47. | Safety | LIVER10 | Summary of Post Baseline Hepatobiliary Laboratory Abnormalities | GSK Statistical Display Standard<br>See hepatobiliary abnormality<br>criteria Section 13.7.1 | HL, M12,<br>EOS |
| 3.48. | Safety | LIVER11 | Summary of Liver Restart/Re-Challenges | GSK Statistical Display Standard | M12, EOS |
| Vital Si | gns | | | | |
| 3.49. | Safety | VS1 | Summary of Change from Baseline in Vital Signs | ICH E3<br>Include Baseline values, weight, and<br>BMI | M12, EOS |
| Cardio | vascular Risl | <b>Factors</b> | | | |
| 3.50. | Safety | FH1 | Summary of Family History of Cardiovascular Risk Factors | GSK Statistical Display Standard | M12 |
| 3.51. | Safety | SU1 | Summary of Substance Use | GSK Statistical Display Standard | M12 |
| COVID | -19 Adverse I | Events | | | l |
| 3.52. | Safety | PAN1 | Summary of COVID-19 Assessments for Subjects with COVID-19 Adverse Events | GSK Statistical Display Standard Includes events across all phases | IA2, M12,<br>EOS |
| 3.53. | Safety | PAN2 | Summary of COVID-19 Additional Assessments for Subjects with COVID-19 Adverse Events | GSK Statistical Display Standard<br>Includes events across all phases | M12, EOS |
| 3.54. | Safety | PAN3 | Summary of COVID-19 Symptoms for Subjects with COVID-19 Adverse Events | GSK Statistical Display Standard Includes events across all phases | M12, EOS |
| 3.55. | Safety | PAN10 | Incidence of Covid-19 Adverse Events Overall and by Subgroup | Subgroups include Sex,<br>Implementation Arm<br>Includes events across all phases | M12, EOS |

| Safety: | Safety: Tables | | | |
|---|---|---|---|---|
| Adverse Events of Special Interest | | | | |
| 3.56. | Safety | 201584/primary_27/T3.140 | Summary of Depression, Anxiety and Suicidal or Suicidal Ideation/Behaviour Adverse Events by System Organ Class, Maximum DAIDS Toxicity Grade, and History of Depression, Anxiety or Suicidal Ideation/Behaviour at Screening | M12, EOS |
| 3.57. | Safety | 201584/primary_07/T3.122 | Summary of Depression Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | M12, EOS |
| 3.58. | Safety | 201584/primary_07/T3.125 | Summary of Anxiety Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | M12, EOS |
| 3.59. | Safety | 201584/primary_07/T3.128 | Summary of Suicidal Ideation/Behaviour Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | M12, EOS |
| 3.60. | Safety | 201584/primary_07/T3.134 | Summary of Seizures Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | M12, EOS |
| 3.61. | Safety | 201584/primary_07/T3.137 | Summary of Hepatic Safety Profile: Assessment of Risk of Hepatoxicity Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | M12, EOS |
| 3.62. | Safety | 201584/primary_07/T3.140 | Summary of Hypersensitivity Reactions (HSR) Adverse<br>Events of Special Interest by System Organ Class and<br>Preferred Term (Number of Subjects and Occurrences) | M12, EOS |
| 3.63. | Safety | 201584/primary_07/T3.143 | Summary of Rash Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | M12, EOS |

| Safety: | Safety: Tables | | | |
|---|---|---|---|---|
| 3.64. | Safety | 201584/primary_07/T3.149 | Summary of Bipolar Disorder Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | M12, EO |
| 3.65. | Safety | 201584/primary_07/T3.152 | Summary of Psychosis Adverse Events of Special Interest by<br>System Organ Class and Preferred Term (Number of<br>Subjects and Occurrences) | M12, EO |
| 3.66. | Safety | 201584/primary_07/T3.155 | Summary of Mood Disorders Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | M12, EO |
| 3.67. | Safety | 201584/primary_07/T3.158 | Summary of Sleep Disorders Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | M12, EO |
| 3.68. | Safety | 201584/primary_07/T3.161 | Summary of Hyperglycaemia Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | M12, EO |
| 3.69. | Safety | 201584/primary_07/T3.161 | Summary of Weight Gain Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | M12, EO |
| 3.70. | Safety | 201584/primary_07/T3.164 | Summary of Rhabdomyolysis Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | M12, EO |
| 3.71. | Safety | 201584/primary_07/T3.167 | Summary of Pancreatitis Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | M12, EO |
| 3.72. | Safety | 201584/primary_07/T3.170 | Summary of Impact on Creatinine Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | M12, EO |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| 3.73. | Safety | 201584/primary_07/T3.173 | Summary of Safety in Pregnancy Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | M12, EOS |
| 3.74. | Safety | 207966/primary_15/T3.109 | Summary of Characteristics of Adverse Events of Special Interest | | M12, EOS |
| 3.75. | Safety | AE99 | Adverse Event Overview by Study Phase and Subgroup | Repeat Table 3.9 for all relevant subgroups including country, sex, age group, race group, and CD4 group as mentioned in Section 5.4.2. Do not include LTFU data. Include BMI >=30/<30 as a subgroup | M12 |





## 13.12.8. Safety Figures

| Safet | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard /<br>Example Shell | Title | Programming Notes | Deliverable |
| Adve | rse Events | | | | |
| 3.1. | Safety | 201584/primary_07/F3.14 | Plot of Incidence of Study Drug Injection Site Reaction Adverse Events by Implementation Arm and Visit (Overall and Common) – CAB and/or RPV | Sort by CAB+RPV, CAB, then RPV<br>ISR onset assigned to most recent<br>IM injection Visit | M12, EOS |

| Labo | Laboratory | | | | |
|---|---|---|---|---|---|
| 3.3. | Safety | LIVER14 | Scatter Plot of Maximum vs. Baseline for ALT | GSK Statistical Display Standard | M12, EOS |
| 3.4. | Safety | LIVER9 | Scatter Plot of Maximum Total Bilirubin vs Maximum ALT – eDISH Plot | GSK Statistical Display Standard | M12, EOS |

## 13.12.9. Other Tables

| Study \ | Study Visit Length | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard<br>/ Example<br>Shell | Title | Programming Notes | Deliverable |
| 4.1 | Safety | OTR_T1 | Summary of Study Visit Length (minutes) by Visit,<br>Country, and Site (Intervention Phase) | Include overall summary for each visit and country. | IA1, IA2, HL, M12 |
| 4.2 | Safety | OTR_T2 | Summary of Study Visit Length (minutes) by Visit and Subgroup (Intervention Phase) | Include all subgroups listed in Section 5.4.2 except for Site & Country | M12 |
| 4.3 | Safety | NS1 | Summary of Remote & Nursing Visits by Visit, Country, and Site | Include overall summary for each visit and country. Add footnote: "All remote visits were recorded in response to missed visits due to Covid-19." | IA2, M12, EOS |
| 4.4 | Safety | NS1 | Summary of Remote & Nursing Visits by Visit and Subgroup | Include all subgroups listed in Section 5.4.2 except for Site & Country Add footnote: "All remote visits were recorded in response to missed visits due to Covid-19." | M12, EOS |

## 13.12.10. ICH Listings

| ICH: | Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard /<br>Example Shell | Title | Programming Notes | Deliverable |
| Subj | ject Dispositio | n | | | |
| 1. | Enrolled | ES2 | Listing of Reasons for Study Withdrawal | ICH E3 Add column for Phase, Visit, and Implementation arm | M12, EOS |
| 2. | Enrolled | SD2 | Listing of Reasons for Study Treatment Discontinuation | ICH E3 Add column for Phase, Visit, and Implementation arm | HL, M12, EOS |
| Prot | ocol Deviation | S | | | |
| 3. | Enrolled | DV2 | Listing of Important Protocol Deviations | ICH E3 Add column for Phase, Visit, and Implementation arm Add a column on the right for "COVID-19 Related". The possible values in this column are Y and N, where Y indicates the deviation is COVID-19 related and N indicates the deviation is non-COVID-19 related. | IA1, IA2, M12,<br>EOS |
| 4. | Enrolled | DV2 | Listing of Protocol Deviations Related to COVID-19 | Add column for Phase, Visit, and Implementation arm | HL, M12, EOS |
| 5. | Enrolled | DV2 | Listing of Implementation Science Protocol Deviations | Add column for Phase, Visit, and Implementation arm | HL, M12, EOS |
| 6. | Safety | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | ICH E3 | M12 |
| Pop | ulations Analy | sed | | | |
| 7. | Enrolled | SP3 | Listing of Subjects Excluded from Safety Population | ICH E3 | M12 |

| ICH: | Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard /<br>Example Shell | Title | Programming Notes | Deliverable |
| Dem | ographic and | Baseline Characteristics | | | |
| 8. | Safety | DM2 | Listing of Demographic Characteristics | ICH E3 | M12 |
| 9. | Safety | DM9 | Listing of Race | ICH E3 | M12 |
| Effic | асу | | | | |
| 10. | Safety | SNAPSHOT11 | Listing of Qualitative and Quantitative Plasma HIV-1 RNA Data | | HL, M12 |
| 11. | Safety | SNAPSHOT12 | Listing of Study Outcome (50 copies/mL cutoff) at Month 12 – Snapshot Analysis | | HL, M12 |
| 12. | Safety | VF4 | Listing of Plasma HIV-1 RNA and CD4+ Cell Count for subjects with Confirmed Virologic Failure | | M12, EOS |
| Expo | osure and Tre | atment Compliance | | | |
| 13. | Safety | 207966/primary_15/L12 | Listing of Exposure Data | ICH E3<br>Remove Phase Day | M12 |
| Adve | erse Events | , | | | |
| 14. | Safety | AE8 | Listing of All Adverse Events | ICH E3 Add column for Phase, Visit, and Implementation arm; see gsk1265744/mid207966/primary_15/L19 | HL, M12 |
| 15. | Safety | AE8 | Listing of Grade 3-5 Adverse Events | Add column for Phase, Visit, and Implementation arm; see gsk1265744/mid207966/primary_15/L19 | M12 |
| 16. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | ICH E3 | M12 |
| 17. | Safety | 201584/primary_07/L22 | Listing of Changes in Intensity/Grades of Study Drug Injection Site Adverse Events | Remove phase treatment, add visit | M12, EOS |

| ICH: | Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard /<br>Example Shell | Title | Programming Notes | Deliverable |
| 18. | Safety | AE8 | Listing of COVID-19 Adverse Events | Add column for Phase, Visit, and Implementation arm; see gsk1265744/mid207966/primary_15/L19 Include Y/N column checked if the AE lead to discontinuation | HL, M12 |
| 19. | Safety | PAN12 | Listing of COVID-19 Assessments and Symptom Assessments | Add column for Phase and Visit | M12 |
| 20. | Safety | PAN5 | Country Level Listing of Start Dates of COVID-19 Pandemic Measures | | M12, EOS |
| Serie | ous and Other | Significant Adverse Eve | ents | | |
| 21. | Safety | AE8 | Listing of Fatal Serious Adverse Events | ICH E3 Add column for Phase, Visit, and Implementation arm | M12 |
| 22. | Safety | AE8 | Listing of Non-Fatal Serious Adverse Events | ICH E3 Add column for Phase, Visit, and Implementation arm | M12, EOS |
| 23. | Safety | AE8 | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | ICH E3 Add column for Phase, Visit, and Implementation arm | M12, EOS |
| Labo | oratory | | | | |
| 24. | Safety | LB14 | Listing of Laboratory Data with Character Results | ICH E3 Add Category, Phase/Period, Visit | M12 |

# 13.12.11. Non-ICH Listings

| Non-IC | H: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard GSK<br>Statistical Display<br>Standard / Example<br>Shell | Title | Programming Notes | Deliverable |
| Subjec | t Disposition | | | | |
| 25. | Screened | ES7 | Listing of Reasons for Screen Failure | Journal Guidelines | M12 |
| 26. | Screened | ES9 | Listing of Subjects Who Were Rescreened | | M12 |
| 27. | Enrolled | SD2 | Listing of Reasons for Study Treatment Discontinuation During the Oral Lead-in Period | Add column for Visit and Implementation arm | M12 |
| 28. | Safety | TA1 | Listing of Planned and Actual Treatments by Implementation Arm | GSK Statistical Display Standard | M12 |
| 29. | Safety | TA1 | Listing of Subjects with Missed Visits Due to Covid-19 by Implementation Arm | Add a column indicating whether a remote visit was performed (Y/N) | M12, EOS |
| Prior a | nd Concomita | nt Medications | | | |
| 30. | Safety | 207966/primary_15/Listing<br>36 | Listing of Prior ART Medications | Remove the column 'Phase during Which Concomitant' | M12 |
| 31. | Safety | 207966/primary_15/Listing<br>37 | Listing of Concomitant ART Medications | Add column for Phase, Visit, and Implementation arm Add a column specifying "SOC Oral Bridging?" which has values of "Yes" and "No". | HL, M12,<br>EOS |
| 32. | Safety | 207966/primary_15/Listing<br>38 | Listing of ART Medications Received during Long-term Follow-up Phase | Remove the column 'Phase during Which Concomitant' | M12, EOS |
| Medica | l History | | | | |
| 33. | Safety | 201584/primary_01/L43 | Listing of Medical History of Seizure | | M12 |

| Efficacy | / | | | | |
|---|---|---|---|---|---|
| 34. | Safety | CDC4 | Listing of CDC Classification of HIV-1 Infection at Baseline | | M12 |
| 35. | Safety | CDC5 | Listing of CDC Stage 3 HIV-1 Associated Conditions | Add column for Phase, Visit | M12, EOS |
| Exposu | re | | | | |
| 36. | Safety | EX3 | Listing of Actual Visit Dates and Day Since Last Dose | Add column for implementation arm | IA1, IA2,<br>M12, EOS |
| 37. | Safety | 207966/primary_15/L60 | Listing of Oral Bridging Exposure Data | Add visit to phase. Add column for implementation arm and to identify COVID relatedness. | HL, M12,<br>EOS |
| 38. | Safety | 207966/primary_15/L60 | Listing of Exposure Data for Subjects Who Received Oral Bridging | Add visit to phase. Add columns for implementation arm, Total Volume Injected / Duration of Oral Treatment | M12 |
| Hepato | biliary (Liver) | | | | |
| 39. | Safety | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting | GSK Statistical Display Standard<br>Add column for Phase, Visit | M12, EOS |
| 40. | Safety | LIVER15 | Liver Stopping Event Profile | GSK Statistical Display Standard<br>Add column for Phase, Visit | M12, EOS |
| 41. | Safety | LIVER13 | Listing of Subjects Meeting Hepatobiliary Laboratory<br>Criteria Post-Baseline | GSK Statistical Display Standard<br>Add column for Phase, Visit | HL, M12,<br>EOS |
| 42. | Safety | LB12 | Listing of ALT, AST, Bilirubin (including Total and Direct Bilirubin), INR, and ALP for Subjects Meeting Hepatobiliary Lab Abnormality Criteria | Add column for Phase, Visit | M12, EOS |

| Other | | | | | |
|---|---|---|---|---|---|
| 43. | Safety | EG3 | Listing of All ECG Values for Subjects with Recorded ECG Data | GSK Statistical Display Standard<br>Add column for Phase, Visit | M12 |
| 44. | Safety | PREG1 | Listing of Subjects Who Became Pregnant During the Study | GSK Statistical Display Standard<br>Add column for Phase, Visit | M12, EOS |
| 45. | Safety | 201584/primary_17/L54 | Listing of Replication Capacity in IN and PR/RT Region | Add column for Phase, Visit | M12, EOS |
| Vital Sig | gns | | | | |
| 46. | Safety | VS5 | Listing of Vital Sign Results | GSK Statistical Display Standard<br>Required for ClinPharm studies<br>only. | M12 |
| Pharma | cokinetic | | | | |
| 47. | Safety | PK07 | Listing of Plasma CAB Pharmacokinetic Concentration-<br>Time Data | | M12, EOS |
| 48. | Safety | PK07 | Listing of Plasma RPV Pharmacokinetic Concentration-<br>Time Data | | M12, EOS |
| Pregna | ncy (condition | nal on incidence of pregnan | су) | | |
| 49. | Safety | PREG_01 | Listing of Pregnancy Details and Outcomes | Results to be pulled from the<br>Pregnancy Notification Form | EOS |
| 50. | Safety | PREG_02 | Listing of Pregnancy Outcomes | Results to be pulled from the<br>Pregnancy Follow-up Form | EOS |
| 51. | Safety | 207966/primary_15/Listing<br>37 | Listing of Concomitant Medications for Pregnant Participants During and After Pregnancy | Results should reconcile with the Pregnancy Notification and Follow-up Forms Follow specifications for the current Listing 31 | EOS |
| 52. | Safety | SNAPSHOT11 | Listing of Qualitative and Quantitative Plasma HIV-1 RNA Data for Pregnant Participants | Follow specifications for the current Listing 10 | EOS |
| 53. | Safety | 207966/primary_15/L12 | Listing of Exposure Data for Pregnant Participants | Follow specifications for the current Listing 13 | EOS |

| 54. | Safety | AE8 | Listing of Adverse Events for Pregnant Participants During and After Pregnancy | Follow specifications for the current Listing 14 | EOS |
|---|---|---|---|---|---|
| 55. | Safety | LB5A | Listing of All Laboratory Data for Pregnant Participants During and After Pregnancy | | EOS |
| 56. | Safety | PK07 | Listing of Plasma CAB Pharmacokinetic Concentration-<br>Time Data for Pregnant Participants During and After<br>Pregnancy | Follow specifications for the current Listing 43 | EOS |
| 57. | Safety | PK07 | Listing of Plasma RPV Pharmacokinetic Concentration-<br>Time Data for Pregnant Participants During and After<br>Pregnancy | Follow specifications for the current Listing 44 | EOS |

## 13.13. Appendix 13: Example Mock Shells for Data Displays

Protocol: 213199 Page 1 of x

Population: Safety

# Table DISP\_T1 Summary of Subject Disposition at Each Study Phase

| Study Phase | | | F | AB Oral +<br>RPV Oral<br>(N=100) | CA | B LA + RPV<br>LA<br>(N=100) | | Total<br>(N=200) |
|---|---|---|---|---|---|---|---|---|
| Intervention Phase | ENTERED | | | / ° ) | | / ° \ | | (° ) |
| intervention Phase | COMPLETED | | | (xx.x%) | | (xx.x%) | | (xx.x%) |
| | | | | (xx.x%) | | (xx.x%) | XX | (xx.x%) |
| | WITHDRAWN | | | (xx.x%) | | (xx.x%) | XX | (xx.x%) |
| | COVID-19 | RELATED | XX | (xx.x%) | XX | (xx.x%) | XX | (xx.x%) |
| Completed Intervention Phase but Withdrew Prior to Extension Phase | ENTERED | | | | | | XX | (xx.x%) |
| | COMPLETED | | | | | | XX | (xx.x%) |
| | WITHDRAWN | | | | | | XX | (xx.x%) |
| | COVID-19 | RELATED | | | | | XX | (xx.x%) |
| Extension Phase | ENTERED COMPLETED WITHDRAWN COVID-19 | RELATED | | | | | XX<br>XX<br>XX | (xx.x%)<br>(xx.x%)<br>(xx.x%)<br>(xx.x%) |
| Long-term Follow-up Phase | ENTERED<br>COMPLETED<br>WITHDRAWN<br>COVID-19 | RELATED | | | | | XX<br>XX<br>XX | (xx.x%)<br>(xx.x%)<br>(xx.x%)<br>(xx.x%) |

213199

Intervention/Extension phase status and reason for withdrawal is based on date and reason collected in the study treatment discontinuation form.

A subject is considered to have entered the Extension phase if the subject received a Month 14 injection or had any assessments collected at any Extension phase nominal visit.

A subject is considered to have entered the Long-term Follow-up phase if they have received at least one CAB and/or RPV injection and have started Long-term Follow-up ART

Long-term Follow-up completion/withdrawal is based on data collected in the Study Conclusion form. PPD /arenv/arprod/gsk1265744/mid209493/primary\_01/drivers/t\_sp\_sd\_phase.sas 02FEB2021 11:58 Protocol: 213199 Page 1 of x

Population: Safety

Table DISP\_T2
Summary of Reasons for Withdrawal at Each Study Phase

| Phase | Primary Reason[1]/Subreason[2] for Withdrawal | CAB Oral + RPV<br>Oral<br>(N=100) | CAB LA + RPV<br>LA<br>(N=100) | Total<br>(N=200) |
|---|---|---|---|---|
| Intervention | ADVERSE EVENT | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Phase | | | | |
| | COVID-19 RELATED | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | LACK OF EFFICACY | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | PROTOCOL DEVIATION | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | COVID-19 RELATED | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | PROHIBITED MEDICATION USE | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | NON-COMPLIANCE WITH STUDY TREATMENT | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | SUBJECT REACHED PROTOCOL-DEFINED STOPPING | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | CRITERIA | | | |
| | STUDY TERMINATED BY SPONSOR | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | LOST TO FOLLOW-UP | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | INVESTIGATOR SITE CLOSED | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | PHYSICIAN DECISION | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | WITHDRAWAL BY SUBJECT | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | COVID-19 RELATED | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | FREQUENCY OF INJECTIONS | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Long-term Follow-up Phase | LOST TO FOLLOW-UP | | | xx (xx.x%) |
| | WITHDRAWAL BY SUBJECT | | | xx (xx.x%) |
| | SUBJECT RELOCATED | | | x (xx.x%) |

213199

BURDEN OF PROCEDURES x (xx.x%)

- [1] Subjects may have only one primary reason.
- [2] Percentages for subreasons may sum to more or less than 100%. Subjects may have more than one subreason underneath a single primary reason. Subjects are not required to indicate subreasons. Intervention/Extension phase: status and reason for withdrawal based on date and reason collected in the study treatment discontinuation form. Long term Follow-up: completion/withdrawal based on data collected in the Study Conclusion form.

Protocol: 213199 

Population: Safety

Table EFF\_T1
Summary of Study Outcomes (50 c/mL cutoff) at Month 12 (Intervention Phase)
- Snapshot Analysis

| Outcome | Q4W IM<br>(N=xx) |
|---------------------------------------------------------|------------------|
| HIV-1 RNA<50 c/mL | xx (xx%) |
| HIV-1 RNA>=50 c/mL | xx (xx%) |
| Data in window not below threshold | xx (xx%) |
| Discontinued for lack of efficacy | xx (xx%) |
| Discontinued for other reason while not below threshold | xx (xx%) |
| Change in ART [1] | xx (xx%) |
| No Virologic Data | xx (xx%) |
| Discontinued study due to AE or Death | xx (xx%) |
| Discontinued study for Other Reasons | xx (xx%) |
| On study but missing data in window | xx (xx%) |

<sup>[1]</sup> Excludes CAB + RPV Oral Bridging and COVID-19 related temporary oral bridging with SOC.

Protocol: mid213199 

Population: Safety

Table EFF\_T2
Summary of Study Outcomes (50 c/mL cutoff) at Month 12 (Intervention Phase)
- Snapshot Analysis

| | Q4W IM |
|---------------------------------------------------------|----------|
| Outcome | (N=xx) |
| HIV-1 RNA<50 c/mL | xx (xx%) |
| HIV-1 RNA>=50 c/mL | xx (xx%) |
| Data in window not below threshold | xx (xx%) |
| Non-COVID-19 related | xx (xx%) |
| Discontinued for lack of efficacy | xx (xx%) |
| Discontinued for other reason while not below threshold | xx (xx%) |
| COVID-19 related | xx (xx%) |
| Discontinued for lack of efficacy | xx (xx%) |
| Discontinued for other reason while not below threshold | xx (xx%) |
| Change in ART [1] | xx (xx%) |
| No Virologic Data | xx (xx%) |
| Non-COVID-19 related | xx (xx%) |
| Discontinued study due to AE or Death | xx (xx%) |
| Discontinued study for Other Reasons | xx (xx%) |
| On study but missing data in window | xx (xx%) |
| COVID-19 related | xx (xx%) |
| Discontinued study due to AE or Death | xx (xx%) |
| Discontinued study for Other Reasons | xx (xx%) |
| On study but missing data in window | xx (xx%) |

<sup>[1]</sup> Excludes CAB + RPV Oral Bridging and COVID-19 related temporary oral bridging with SOC.

Protocol: mid213199 

Population: Safety

### Table SAF T1

Summary of Adherence to CAB LA + RPV LA Dosing Schedule by Visit, Country, Site, and COVID Impacted/Non-Impacted (Intervention Phase)

Country: xxxxx {Programmer's Note: repeat for each of 5 countries overall, each individual site, and total}

Site ID: xxxx

COVID-19: xxx {non-impacted + impacted/non-impacted/impacted}

| Timeliness of Injections Relative to Date of<br>Projected Dosing Visits | Month 2 | Month 4 | Month 6 | Month 8 | Month 10 | Month 12 | Total |
|---|---|---|---|---|---|---|---|
| No. of Expected Injection Visits | XXXX | xxxx | xxxx | xxxx | xxxx | xxxx | xxxx |
| <-14 days | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| -14 days to - 8 days | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| -7 days to - 1 days | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| 0 | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| 1 days to 7 days | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| 8 days to 14 days | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| > 14 days | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| Missed Injection without OB (non-COVID-19 | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| related) | | | | | | | |
| Missed Injection without OB (COVID-1 related) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| Missed Injection with OB (non-COVID-19 related) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| Missed Injection with OB (COVID-19 related) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| Late Out of Window Injections (days outside +7 day window) | | | | | | | |
| n | XXX | XXX | XXX | XXX | XXX | XXX | xxx |
| Mean | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | xxx.x |
| SD | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Median | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| Q1 | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Q3 | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Min | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

| Timeliness of Injections Relative to Date of | Month 2 | Month 4 | Month 6 | Month 8 | Month 10 | Month 12 | Total |
|---|---|---|---|---|---|---|---|
| Projected Dosing Visits | | | | | | | |
| Max | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

213199

Protocol: mid213199 

Population: Safety

Table SAF T2

Summary of Adherence to CAB LA + RPV LA Dosing Schedule by Visit, Subgroup, and COVID Impacted/Non-Impacted (Intervention Phase)

Subgroup: xxxx {Programmer's Note: repeat for each subgroup}

COVID-19: xxx { Programmer's Note: repeat for non-impacted + impacted/non-impacted/impacted}

| Timeliness of Injections Relative to Date of Projected Dosing Visits | Month 2 | Month 4 | Month 6 | Month 8 | Month 10 | Month 12 | Total |
|---|---|---|---|---|---|---|---|
| Trojected Dearing Vibros | | | | | | | |
| No. of Expected Injection Visits | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX |
| <-14 days | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| -14 days to - 8 days | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| -7 days to - 1 days | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| 0 | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| 1 days to 7 days | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| 8 days to 14 days | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| > 14 days | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| Missed Injection without OB (non-COVID-19 | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| related) | | | | | | | |
| Missed Injection without OB (COVID-1 related) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| Missed Injection with OB (non-COVID-19 related) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| Missed Injection with OB (COVID-19 related) | xx (%) | xx (응) | xx (%) | xx (%) | xx (%) | xx (%) | xx (%) |
| Late Out of Window Injections (days outside +7 day window) | | | | | | | |
| n | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Mean | XXX.X | XXX.X | XXX.X | XXX.X | xxx.x | XXX.X | XXX.X |
| SD | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx |
| Median | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| Q1 | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Q3 | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Min | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

| Timeliness of Injections Relative to Date of | Month 2 | Month 4 | Month 6 | Month 8 | Month 10 | Month 12 | Total |
|---|---|---|---|---|---|---|---|
| Projected Dosing Visits | | | | | | | |
| Max | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Protocol: mid213199 

Population: Safety

# Table OTR\_T1 Summary of Study Visit Length (minutes) by Visit, Country, and Site

| Country | N | | | Month 1 | Month 2 | Month 6 | Month 8 | Total |
|---|---|---|---|---|---|---|---|---|
| Site | | | | | | | | |
| Overall | | Lead Time | n | XXX | XXX | XXX | XXX | XXX |
| Overall | | | | | | | | |
| | | | Mean | XX.X | XX.XX | XX.X | XX.X | XX.X |
| | | | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | Min. | XX | XX | XX | XX | XX |
| | | | Max. | XX | XX | XX | XX | XX |
| | | Process | n | XXX | XXX | XXX | XXX | XXX |
| | | Time | | | | | | |
| | | | Mean | XX.X | XX.XX | XX.X | XX.X | XX.X |
| | | | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | Min. | XX | XX | XX | XX | XX |
| | | | Max. | XX | XX | XX | XX | XX |
| | | Total | n | XXX | XXX | XXX | XXX | XXX |
| | | Time | | | | | | |
| | | | Mean | XX.X | XX.XX | XX.X | XX.X | XX.X |
| | | | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | Etc. | XX.X | XX.X | XX.X | XX.X | XX.X |

Lead Time = Actual Start Time of Appointment - Arrival Time.

213199

Process Time = Actual End Time of Appointment - Actual Start Time of Appointment. [Programmers Note: repeat for each, country site, and total]

Protocol: mid213199


Population: Safety

Table OTR T2

## Summary of Study Visit Length (minutes) by Visit and Subgroup

| Subgroup<br>Strata | N | | | | Month 2 | | Month 8 | Total |
|---|---|---|---|---|---|---|---|---|
| | | Total Mimo | | | | | | |
| Sex | | Lead Time | n | XXX | XXX | XXX | XXX | XXX |
| Male | | | | | | | | |
| | | | Mean | XX.X | XX.XX | XX.X | XX.X | XX.X |
| | | | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | Q3 | XX.X | xx.x | XX.X | xx.x | XX.X |
| | | | Min. | XX | XX | XX | XX | XX |
| | | | Max. | XX | XX | XX | XX | XX |
| | | Process | n | XXX | XXX | XXX | XXX | XXX |
| | | Time | | | | | | |
| | | | Mean | XX.X | XX.XX | XX.X | XX.X | XX.X |
| | | | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | Q1 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | Q3 | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | Min. | XX | XX | XX | XX | XX |
| | | | Max. | XX | XX | XX | XX | XX |
| | | Total | n | xxx | XXX | XXX | xxx | xxx |
| | | Time | | | | | | |
| | | | Mean | XX.X | XX.XX | XX.X | XX.X | XX.X |
| | | | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | | Etc. | XX.X | XX.X | XX.X | XX.X | XX.X |

Lead Time = Actual Start Time of Appointment - Arrival Time.

Process Time = Actual End Time of Appointment - Actual Start Time of Appointment.

[Programmers Note: repeat for each Subgroup and Strata]

Preg\_01

| Protocol: 213199 | | | | | eg_01 | | | | Page 1 of x |
|---|---|---|---|---|---|---|---|---|---|
| Population: Safety | У | | | | | | | | |
| | | | | Listing 49 | | | | (Data as o | f: 30MAY2011) |
| | | | Listing | of Pregnancy | Details | | | | |
| Site Id.: ppn | | | | | | | | | |
| FFU | | | | | | N | Previous | | |
| | | | | | | | ancies | | |
| | | | | Contraceptio | | Fregii | ancies | | |
| | | | | n?/Contracep | | | | | |
| Unique Subject | | Date of | | tion | | | | | |
| Id./ | | Last | Estimated | Type/Concept | | | | | |
| Subject | Mother's | Menstrual | Date of | ion Type | Relevant Lab | | | | |
| Id./Implementatio | | Period/ | Delivery/ | (Normal, | Tests and | | | Additional F | agrara that |
| n Arm | Birth | 1 | _ | IVF)[1] | Procedures | Dro-torm | F::11-+orm | May Impact P | |
| II ALIII | BILCH | Study Day | Study Day | IVF)[I] | FIOCEGUIES | Fie-ceim | ruii-ceim | May Impact F | regnancy |
| | | 0010 | 0010 | Y/Birth | Amniocentesi | Spontaneo | NT 1 | | |
| PPD (CAR IA + | xxxx | 2012- <b>рр</b> р<br>т23:59/ | 2012- <b>PPD</b><br>T23:59/ | Control/Norm | s performed | us | Births | | |
| /CAB LA +<br>RPV LA ARM-e | | 1 | 1 | al | s periormed | Abortion | | | |
| RPV LA ARM-e | | 1 | 1 | aı | | (n): x | (n): x | | |
| | | | | | | | Stillbirt | | |
| | | | | | | | hs (n): x | | |
| | | | | | | (n): x | ns (n): x | | |
| | | | | | | Other | Born | | |
| | | | | | | (n): x | w/Defects | | |
| | | | | | | (n): x | (n): x | | |
| nnn | xxxx | 2012- <b>PPD</b> | 2012- <b>PPD</b> | N/ /Normal | | Spontaneo | | | |
| PPD /CAB LA + | XXXX | т23:59/ | т23:59/ | N/ /NOIMAI | | us | Births | | |
| RPV LA ARM-e | | 123:39/ | 1 | | | Abortion | | | |
| KLA TH WEM-6 | | _ | 1 | | | (n): x | (11): X | | |
| | | | | | | | Stillbirt | | |
| | | | | | | | hs (n): x | | |
| | | | | | | (n): x | 113 (11) . X | | |
| | | | | | | Other | Born | | |
| | | | | | | (n): x | w/Defects | | |
| | | | | | | (11). | (n): x | | |
| | | | | | | | () | | |
| [1] Normal concept | tion inclu | des the use | of fertility | drugs IVF = | in witro fert | ilization | | - | |
| | | | | arays. IVF - | In vicio lei | JIIIZACION. | | | |
| Directory/program | m.sas UlJ | ANZUU2 12:01 | | | | | | | |

Preg 02

| | | | | 1108 | _02 | | | |
|---|---|---|---|---|---|---|---|---|
| Protocol: 213199 | | | | | | | | Page 1 of x |
| Population: Safety | У | | | | | | | |
| | | | | Listing 50 | | | | (Data as of: 30MAY2011) |
| | | | Listino | g of Pregnancy O | utcomes | | | |
| Site Id.: ppp | | | | | | | | |
| | | | | Date of | | | | |
| Unique Subject | | | | Birth, miscarria | | | | |
| Id./ | | Foetal/Neonata | Origin of | ge, termination | Infant | | Pregnancy | |
| Subject | | l Status | Birth | / Study Day / | Sex/Length | Apgar Score | Dur- | |
| <pre>Id./Implementatio</pre> | Pregnancy | (Normal, Brith | Defect | Gestational | (cm)/Weight | (0-10) 1st | ation | |
| n Arm | Status [1] | Defect, Other) | Known? | Weeks | (g) | / 2nd | (days) [2] | Additional Pregnancy Details |
| PPD | Delivery: | Birth Defect | Yes : | 2012- <b>PPD</b> | M / 50 / | 8/8 | xx | |
| /CAB LA + | Normal | | xxxx | T23:59/ | 2500 | | | |
| RPV LA ARM-e | | | | 1 / 38 | | | | |
| PPD | PPD | NA | NA | 2012- <b>PPD</b> | NA | 0 | xx | SAE delivery complication |
| CAB LA + | | | | T23:59/ | | | | |
| RPV LA ARM-e | | | | 1 / 36 | | | | |

<sup>[1]</sup> Status options include Delivery: method specified, Stillbirth, Foetal death, Spontaneous abortion, Elective abortion, Other: specified.

<sup>[2]</sup> Pregnancy duration calculated as Date of Birth/Miscarriage/Termination - Date of Last Menstrual Period + 1.

/Directory/program.sas 01JAN2002 12:01

## Signature Page for 213199 TMF- 15213711 v 1.0

| Reason for signing: Approved | Name: PPD<br>Role: A<br>Date of signature: 12-Dec-2022 13:40:23 GMT+0000 |
|---|---|
| Reason for signing: Approved | Name: PPD Role: A Date of signature: 12-Dec-2022 13:44:41 GMT+0000 |
| Reason for signing: Approved | Name: PPD<br>Role: A<br>Date of signature: 12-Dec-2022 15:30:08 GMT+0000 |

Signature Page for TMF-15213711 v1.0